#### **Statistical Analysis Plan**

**Study ID: 205646** 

Official Title of Study: Reporting and Analysis Plan Addendum 2 for 205646, a Phase 3, Multi-Center,
Randomized, Double-Blind, Placebo-Controlled, 104-Week Study to Evaluate the
Efficacy and Safety of Belimumab Administered in Combination with Rituximab to
Adult Subjects with Systemic Lupus Erythematosus (SLE)

Date of Document: 22-JUL-2021

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan Addendum 2 |
| Title | : | Reporting and Analysis Plan Addendum 2 for 205646, a Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 104-Week Study to Evaluate the Efficacy and Safety of Belimumab Administered in Combination with Rituximab to Adult Subjects with Systemic Lupus Erythematosus (SLE) |
| Compound Number | : | GSK1550188 |
| <b>Effective Date</b> | : | Refer to Document Date |

#### **Description:**

- This second RAP addendum is supplemental to the RAP (Dated: 05/AUG/2020), and the first RAP addendum (Dated: 08/OCT/2020).
- It is based on protocol amendment 04 (Dated: 30/APR/2020) of study 205646.
- The main purpose of this addendum is to list an abridged set of outputs that will be produced for the final study report. These changes are being made following the first database lock and primary analyses at the end of Year 1 of the study.

#### Author(s)

| Author | Approval Method | |
|---|---|---|
| PPD | | eTMF |
| Principal Statistician | Principal Statistician (Immunology Biostatistics) | |

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **RAP Team Confirmations:**

| Reviewer | Approval Method |
|---------------------------------------------------|----------------------|
| Statistics Leader (Immunology Biostatistics) | E-mail filed in eTMF |
| Programming Leader (Immunology Programming) | E-mail filed in eTMF |
| Medical Monitor (Immunology Clinical Development) | E-mail filed in eTMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Approval Method |
|----------------------------------------------|-----------------|
| Statistics Leader (Immunology Biostatistics) | eTMF |
| Programming Leader (Immunology Programming) | eTMF |


205646

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| BREVI | ATIONS | | 4 |
| INTRO | ODUCTIO | )N | 5 |
| CHAN | IGES/CLA | ARIFICATIONS TO THE RAP | 5 |
| 2.1. | | | |
| | | | 5 |
| | 2.1.1. | | |
| | 2.1.2. | | |
| | 2.1.3. | | |
| | 2.1.4. | | |
| | 2.1.5. | | |
| | 2.1.6. | | |
| | 2.1.7. | Safety Tables | 14 |
| | 2.1.8. | Safety Figures | 19 |
| | 2.1.9. | | |
| | 2.1.10. | Health Outcomes Tables | 21 |
| | 2.1.11. | | |
| | 2.1.12. | Health Outcomes Listings | 22 |
| | 2.1.13. | | |
| | 2.1.14. | | |
| | 2.1.15. | | |
| 2.3. | | | |
| | 2.3.2. | Clarifications for the Year 2 reporting | 26 |
| | INTRO | INTRODUCTION CHANGES/CL/ 2.1. Modification analyse 2.1.1. 2.1.2. 2.1.3. 2.1.4. 2.1.5. 2.1.6. 2.1.7. 2.1.8. 2.1.9. 2.1.10. 2.1.11. 2.1.12. 2.1.13. 2.1.14. 2.1.15. 2.1.14. 2.1.15. 2.1.16. 2.1.17. 2.1.18. 2.2. New 'Intercent | analyses 2.1.1. Study Population Tables 2.1.2. Study Population Figures 2.1.3. Study Population Listings 2.1.4. Efficacy Tables 2.1.5. Efficacy Figures 2.1.6. Efficacy Listings 2.1.7. Safety Tables 2.1.8. Safety Figures 2.1.9. Safety Listings 2.1.10. Health Outcomes Tables 2.1.11. Health Outcomes Figures 2.1.12. Health Outcomes Listings 2.1.13. Biomarkers Tables 2.1.14. Biomarkers Figures 2.1.15. Biomarkers Listings 2.1.16. Pharmacokinetic Tables 2.1.17. Pharmacokinetic Tables 2.1.18. Pharmacokinetic Figures 2.1.18. Pharmacokinetic Listings 2.2. New 'Intent-to-Treat Year 2' Population 2.3. Biomarker and Pharmacokinetic (PK) 2.3.1. Specifications in the original RAP |

# **ABBREVIATIONS**

| Abbreviation | Description |
|---|---|
| ACR | American College of Rheumatology |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| anti-dsDNA | Anti-double-stranded DNA |
| ATC | Anatomical, Therapeutic, Clinical |
| BLyS | B-Lymphocyte Stimulator |
| COVID-19 | Coronavirus Disease 2019 |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| FACIT-Fatigue | Functional Assessment of Chronic Illness Therapy - Fatigue Scale |
| GSK | GlaxoSmithKline |
| IBA | Independent Blinded Assessor |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| IV | Intravenous |
| LLDAS | Lupus Low Disease Activity State |
| LSLV | Last Subject Last Visit |
| MCID | Minimal Clinically Important Difference |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MITT | Modified Intent-To-Treat |
| PGA | Physician Global Assessment |
| PI | Principal Investigator |
| PISR | Post-Injection Systemic Reactions |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| PtGA | Patient Global Assessment |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SLE | Systemic Lupus Erythematosus |
| SLEDAI-2K | Systemic Lupus Erythematosus Disease Activity Index 2000 |
| SLICC | Systemic Lupus International Collaborating Clinics |
| SOC | System Organ Class |
| TF | Treatment Failure |
| WPAI | Work Productivity and Activity Impairment Questionnaire |

#### 1. INTRODUCTION

This RAP addendum is supplemental to the RAP (Dated: 05/AUG/2020), and the first RAP addendum (Dated: 08/OCT/2020). It is based on protocol amendment 04 (Dated: 30/APR/2020) of study 205646.

The main purpose of this addendum is to list an abridged set of outputs that will be produced for the final study report. These changes are being made following the first database lock and primary analyses at the end of Year 1 of the study.

#### 2. CHANGES/CLARIFICATIONS TO THE RAP

# 2.1. Modifications to the planned list of outputs for the end of study analyses

As specified in the original RAP (Section 3.2), there are two database locks for this study, corresponding to the primary analyses and the end of study analyses.

- The primary analyses would include data up to the 52 week visit for the primary endpoint.
- The final analyses would be conducted following the last subject completion of year 2 (including all 8 week-follow-up visits).

The original RAP (Section 3.2) had the following text: "This RAP details the planned analysis for both database locks, with the expectation of an observed treatment benefit at Week 52. If the Week 52 reporting does not identify a treatment benefit, an abridged set of analysis may be conducted at the end of the study, which will be detailed in a RAP amendment or RAP addendum."

Following the results of the primary analyses, an abridged set of outputs will be produced and these are detailed below.

# 2.1.1. Study Population Tables

| Study Popula | Study Population Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Subject Dispo | osition | | | |
| 21.01. | 21.01 | Screened | Study Populations (Year 1&2) | |
| 21.02. | 21.02 | ITT | Subject Status (Year 1&2) | |
| 21.03. | 21.04 | ITT | Subject Status and Reason for Study Withdrawal (Year 1&2) | |
| 21.04. | 21.05 | ITT | Time to Withdrawal from the Study (Year 1&2) | |
| 21.05. | 21.06 | ITT | Treatment Status and Reasons for Discontinuing Belimumab SC Study Treatment (Year 1&2) | |
| 21.06. | 21.07 | ITT | Time to Belimumab SC Study Treatment Discontinuation [1] (Year 1&2) | |
| Protocol Dev | ations | | | |
| 21.07. | 21.09 | ITT Year 2 | Important Protocol Deviations after Week 52 (Year 2) | Use new 'ITT Year 2' Population defined in<br>Section 2.2. |
| Concomitant | Medications | | | |
| 21.08. | 21.11 | ITT Year 2 | Concomitant Medications by ATC Level 1 and ATC Level 4 Term (Year 2) | Use new 'ITT Year 2' Population defined in<br>Section 2.2. |
| 21.09. | 21.13 | ITT | First Medication Usage Resulting in Treatment Failure Designation (Year 1&2) | |
| Extent of Exp | osure | | | |
| 21.10. | 21.14 | ITT | Exposure to Belimumab SC (Study Treatment and Re-start [1]) (Year 1&2) | |

| Study Popula | Study Population Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 21.11. | 21.15 | ITT Year 2 | Exposure to Belimumab SC [1] (Arms A&B: Re-start; Arm C: Study Treatment) (Year 2) | <ul> <li>Belimumab doses that occur up to and including the Week 52 visit date are included as Year 1 doses. Belimumab doses that occur after the Week 52 visit date are included as Year 2 doses. This was incorrect in the original RAP Section 6.5.</li> <li>Use new 'ITT Year 2' Population defined in Section 2.2.</li> </ul> |
| Coronavirus I | Disease 2019 | (COVID-19) Par | ndemic | |
| 21.12. | NEW | ITT | COVID-19 Pandemic Visit Impacts (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |
| 21.13. | NEW | ITT | Reason for Study Withdrawal by Relationship to COVID-19 Pandemic (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |
| 21.14. | NEW | ITT | Reasons for Discontinuing Belimumab SC Study Treatment by Relationship to COVID-19 Pandemic (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |
| 21.15. | NEW | ITT | Important Protocol Deviations by Relationship to COVID-19 Pandemic (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |

# 2.1.2. Study Population Figures

| Study Popula | Study Population Figures | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Subject Dispo | sition | | | |
| 21.01. | 21.01 | ITT | Time to Withdrawal from Study (Year 1&2) | |
| 21.02. | 21.02 | ITT | Time to Belimumab SC Study Treatment Discontinuation (Year 1&2) | |
| COVID-19 Par | COVID-19 Pandemic | | | |
| 21.03. | NEW | ITT | Visits Impacted by COVID-19 Pandemic (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |

# 2.1.3. Study Population Listings

| Study Popula | Study Population Listings | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Subject Dispo | sition | | | |
| 21.01. | 21.01 | Randomized | Subject Disposition (Year 1&2) | |
| 21.02. | 21.02 | Randomized | Reasons for Study Withdrawal (Year 1&2) | |
| 21.03. | 21.03 | Randomized | Reasons for Belimumab SC Study Treatment Discontinuation (Year 1&2) | |
| Protocol Devi | ations | | | |
| 21.04. | 21.04 | Randomized | Important or COVID-19 Protocol Deviations (Year 1&2) | |
| Concomitant | Concomitant Medications | | | |
| 21.05. | 21.06 | Randomized | Concomitant Medications (Year 2) | |

| Study Popula | Study Population Listings | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 21.06. | 21.07 | Randomized | Medications that Result in Treatment Failure Designation (Year 2) | |
| Extent of Exp | osure | | | |
| 21.07. | 21.08 | Randomized | Study Treatment Administration (Year 1&2) | |
| COVID-19 Par | ndemic | | | |
| 21.08. | 21.09 | Randomized | Country Level Listing of Dates of Waves of COVID-19 Pandemic Measures | |
| 21.09. | NEW | Randomized | All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic (Year 1&2) | New output (recommended in GSK COVID-<br>19 guidance document) |

# 2.1.4. Efficacy Tables

| Efficacy Table | Efficacy Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Clinical Remi | ssion | | | |
| 22.01. | 22.01 | MITT | Clinical Remission (IBA) at Week 64 (Hybrid) | |
| 22.02. | 22.02 | MITT | Logistic Regression Analysis of Clinical Remission (IBA) at Week 64 (Hybrid) | |
| 22.03. | 22.03 | MITT | Disposition of Clinical Remission (IBA) at Week 64 (Hybrid) | |
| 22.04. | NEW | MITT | Disposition of Clinical Remission (IBA) by First Reason for Non-Response at Week 64 (Hybrid) | New output (omission in original RAP) |

| Efficacy Table | Efficacy Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 22.05. | 22.04 | MITT | Clinical Remission (IBA) and its Components at Week 64 (Hybrid) | The planned component for 'Corticosteroid >0 to <=5mg/day' has been modified to match the actual component of the endpoint, i.e. "Corticosteroids at a prednisone equivalent dose of 0 mg/day" The planned component for 'Corticosteroid to make to make the planned to |
| 22.06. | NEW | MITT | Clinical Remission (IBA) and its Components by Baseline C3/C4<br>Level & Anti-dsDNA at Week 64 (Hybrid) | <ul> <li>New output (key subgroup of interest)</li> <li>The planned component for 'Corticosteroid &gt;0 to &lt;=5mg/day' has been modified to match the actual component of the endpoint, i.e. "Corticosteroids at a prednisone equivalent dose of 0 mg/day"</li> </ul> |
| 22.07. | 22.08 | MITT | Clinical Remission (IBA) by Visit (Hybrid) (Year 2) | |
| 22.08. | 22.09 | MITT | Clinical Remission (PI) by Visit (Hybrid) (Year 2) | |
| 22.09. | 22.25 | MITT | Duration of Clinical Remission (PI) (Hybrid) (Year 1&2) | |
| 22.10. | 22.20 | MITT | Clinical Remission (PI) Sustained for at least 24 Weeks by Visit (Hybrid) (Year 2) | |
| 22.11. | 22.33 | MITT | Time to Clinical Remission (PI) Sustained for at least 24 weeks and maintained through to Week 104 [1] (Hybrid) | |
| Disease Cont | rol | | | |
| 22.12. | 22.10 | MITT | Disease Control (IBA) at Week 104 (Hybrid) | |
| 22.13. | 22.11 | MITT | Logistic Regression Analysis of Disease Control (IBA) at Week 104 (Hybrid) | |
| 22.14. | 22.12 | MITT | Disposition of Disease Control (IBA) at Week 104 (Hybrid) | |
| 22.15. | NEW | MITT | Disposition of Disease Control (IBA) by First Reason for Non-Response at Week 104 (Hybrid) | New output (omission in original RAP) |

| Efficacy Tables | | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 22.16. | 22.13 | MITT | Disease Control (IBA) and its Components at Week 104 (Hybrid) | |
| 22.17. | NEW | MITT | Disease Control (IBA) and its Components by Baseline C3/C4 Level & Anti-dsDNA at Week 104 (Hybrid) | New output (key subgroup of interest) |
| 22.18. | 22.17 | MITT | Disease Control (IBA) by Visit (Hybrid) (Year 1&2) | |
| 22.19. | 22.18 | MITT | Disease Control (PI) by Visit (Hybrid) (Year 1&2) | |
| 22.20. | NEW | MITT | Duration of Disease Control (PI) (Hybrid) (Year 1&2) | New output (omission in orginal RAP) |
| 22.21. | 22.24 | MITT | Time to Disease Control (PI) Sustained for at least 24 weeks and maintained through to Week 104 [1] (Hybrid) | |
| Complete Rei | mission | | | |
| 22.22. | 22.21 | MITT | Complete Remission (PI) by Visit (Hybrid) (Year 2) | |
| 22.23. | 22.19 | MITT | Complete Remission (PI) Sustained for at Least 24 Weeks by Visit (Hybrid) (Year 2) | |
| Flares | | | | |
| 22.24. | 22.22 | MITT | Time to First Severe Flare (Treatment Policy, TF=Severe Flare) (Year 1&2) (Modified SLE Flare Index) | |
| 22.25. | NEW | MITT | Time to First Severe Flare (Treatment Policy) (Year 1&2) (Modified SLE Flare Index) | New output (of interest following post SAC request for Year 1) Treatment Failures are not included as severe flares |
| 22.26. | 22.23 | MITT | Time to First Flare (Treatment Policy, TF=Flare) (Year 1&2) (Modified SLE Flare Index) | |
| Systemic Lup | ous Erythemat | osus Disease | Activity Index 2000 (SLEDAI-2K) | |
| 22.27. | 22.26 | MITT | SLEDAI-2K (PI) - Change from Baseline by Visit (Hypothetical) (Year 1&2) | |

| Efficacy Table | es | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 22.28. | 22.27 | MITT | SLEDAI-2K (PI) - Organ System Improvement by Organ System and Visit Among Subjects with Organ System Involvement at Baseline [1] (Treatment Policy) (Year 1&2) | |
| 22.29. | 22.28 | MITT | SLEDAI-2K (PI) - Organ System Worsening by Organ System and Visit Among Subjects with No Organ System Involvement at Baseline [1] (Observed) (Year 1&2) | |
| Physician Glo | bal Assessm | ent (PGA) | | |
| 22.30. | 22.29 | MITT | Physician Global Assessment (PGA) - Change from Baseline by Visit (Hypothetical) (Year 1&2) | |
| Systemic Lup | us Internation | nal Collaboratii | ng Clinics (SLICC) | |
| 22.31. | 22.30 | MITT | SLICC/ACR Damage Index Worsening (Change>0) Compared with Baseline at Week 104 (Treatment Policy, WOCF) | |
| Lupus Low D | isease Activit | y State (LLDAS | 5) | |
| 22.32. | 22.31 | MITT | Lupus Low Disease Activity State (LLDAS) (PI) by Visit (Treatment Policy) (Year 1&2) | |
| 22.33. | 22.32 | MITT | Lupus Low Disease Activity State (LLDAS) (PI) and its Components at Weeks 52, 64 and 104 (Treatment Policy) (Year 1&2) | |
| Modified Dise | ease Control | | | |
| 22.34. | 22.39 | MITT | SLEDAI-2K Score <=2 (IBA), Without Current Immunosuppressants, Without Current Belimumab dosing (Arms A & B) and Corticosteroids dose <=5mg/day at Week 104 (COVID-19 Modified, Treatment Policy) | |
| Proteinuria | | | | |
| 22.35. | NEW | ITT | Proteinuria Shifts from Baseline by Visit (Observed) (Year 1&2) | New output (of interest following post SAC request for Year 1) |

# 2.1.5. Efficacy Figures

| Efficacy Figures | | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Efficacy Figur | Efficacy Figures | | | |
| 22.01. | 22.01 | MITT | Clinical Remission (IBA) at Week 64 (Hybrid) | |
| 22.02. | 22.03 | MITT | Clinical Remission (PI) by Visit (Hybrid) (Year 2) | |
| 22.03. | 22.04 | MITT | Disease Control (IBA) at Week 104 (Hybrid) | |
| 22.04. | 22.06 | MITT | Time to First Severe Flare (Treatment Policy, TF=Severe Flare) (Year 1&2) (Modified SLE Flare Index) | |
| 22.05. | 22.07 | MITT | Time to First Flare (Treatment Policy, TF=Flare) (Year 1&2) (Modified SLE Flare Index) | |
| 22.06. | 22.10 | MITT | SLEDAI-2K (PI) - Change from Baseline by Visit (Observed) (Year 1&2) | |
| 22.07. | 22.11 | MITT | Physician Global Assessment (PGA) - Change from Baseline by Visit (Observed) (Year 1&2) | |
| 22.08. | NEW | ITT | Proteinuria Shifts from High at Baseline to Normal by Visit (Observed) (Year 1&2) | New output (of interest following post SAC request for Year 1) |

# 2.1.6. Efficacy Listings

| Efficacy Listin | Efficacy Listings | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Efficacy Listin | Efficacy Listings | | | |
| 22.01. | 22.01 | ITT | Disease Control, Clinical Remission, and Complete Remission by Visit (Year 1&2) | |

# 2.1.7. Safety Tables

| Safety Tables | | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Adverse Ever | nts | | | |
| 23.01. | 23.01 | ITT Year 2 | Adverse Events Summary - On Study (Year 2) | Use new 'ITT Year 2' Population defined in<br>Section 2.2. |
| 23.02. | 23.02 | ITT | Adverse Events Summary - On Study (Year 1&2) | |
| 23.03. | 23.03 | ITT Year 2 | Adverse Events by SOC and PT - On Study (Year 2) | Use new 'ITT Year 2' Population defined in<br>Section 2.2. |
| 23.04. | 23.04 | ITT | Adverse Events by SOC and PT - On Study (Year 1&2) | |
| 23.05. | 23.05 | ITT | Adverse Events by PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.06. | 23.06 | ITT | Study Treatment Related Adverse Events by SOC and PT – Belimumab Only [1] – On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.07. | 23.07 | ITT | Study Treatment Related Adverse Events by SOC and PT – Rituximab Only [1] – On Study (Year 1&2) | Now presents data for Year 1&2 |

| Safety Tables | Safety Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 23.08. | 23.08 | ITT | Study Treatment Related Adverse Events by SOC and PT – Both Belimumab & Rituximab [1] – On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.09. | NEW | ITT | Study Treatment Related Non-Serious Adverse Events by PT – Belimumab Only [1] – On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| 23.10. | NEW | ITT | Study Treatment Related Non-Serious Adverse Events by PT – Rituximab Only [1] – On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| 23.11. | NEW | ITT | Study Treatment Related Non-Serious Adverse Events by PT – Both Belimumab & Rituximab [1] – On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| 23.12. | 23.09 | ITT | Adverse Events by SOC, PT and Maximum Severity – On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.13. | 23.11 | ITT | Adverse Events by SOC and PT and Race - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.14. | 23.13 | ITT | Adverse Events by SOC and PT and Baseline C3/C4 Levels and Anti-dsDNA – On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.15. | 23.22 | ITT | Adverse Events Leading to Permanent Discontinuation of Study<br>Treatment by SOC and PT – Belimumab – On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.16. | 23.23 | ITT | Common [1] Non-Serious Adverse Events by SOC and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| Deaths and S | erious Advers | se Events | | |
| 23.17. | 23.18 | ITT | Death by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.18. | 23.19 | ITT Year 2 | Serious Adverse Events by SOC and PT - On Study (Year 2) | Use new 'ITT Year 2' Population defined in<br>Section 2.2. |
| 23.19. | 23.20 | ITT | Serious Adverse Events by SOC and PT - On Study (Year 1&2) | |
| 23.20. | 23.24 | ITT | Study Treatment Related Serious Adverse Events by SOC and PT - Belimumab Only [1] - On Study (Year 1&2) | Now presents data for Year 1&2 |

| Safety Tables | Safety Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 23.21. | 23.25 | ITT | Study Treatment Related Serious Adverse Events by SOC and PT - Rituximab Only [1] - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.22. | 23.26 | ITT | Study Treatment Related Serious Adverse Events by SOC and PT – Both Belimumab and Rituximab [1] - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.23. | NEW | ITT | Study Treatment Related Serious Fatal and Non-Fatal Adverse Events by PT – Belimumab Only [1] - On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| 23.24. | NEW | ITT | Study Treatment Related Serious Fatal and Non-Fatal Adverse Events by PT - Rituximab Only [1] - On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| 23.25. | NEW | ITT | Study Treatment Related Serious Fatal and Non-Fatal Adverse Events by PT – Both Belimumab and Rituximab [1] - On Study (Year 1&2) | New output (required for Plain Language<br>Summary) |
| Survival Stau | S | | | |
| 23.26. | 23.29 | ITT | Survival Status at Week 104 | |
| Adverse Ever | nts of Special | Interest (AESI) | | |
| 23.27. | 23.30 | ITT Year 2 | Adverse Events of Special Interest by Category - On Study (Year 2) | Use new 'ITT Year 2' Population defined in Section 2.2. |
| 23.28. | NEW | ITT | Adverse Events of Special Interest by Category - On Study (Year 1&2) | New output (omission in original RAP) |
| 23.29. | 23.31 | ITT | Malignant Neoplasm Adverse Events of Special Interest by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.30. | 23.32 | ITT | Post Belimumab SC Injection Systemic Reactions Adverse Events of Special Interest by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.31. | 23.33 | ITT | Serious Post Belimumab SC Injection Systemic Reactions Adverse<br>Events of Special Interest by Category and PT - On Study (Year<br>1&2) | Now presents data for Year 1&2 |

| Safety Tables | Safety Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 23.32. | 23.34 | ITT | Infection Adverse Events of Special Interest by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.33. | 23.35 | ITT | Infection Adverse Events of Special Interest Leading to Belimumab SC Study Treatment Discontinuation by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.34. | 23.36 | ITT | Depression/Suicide/Self-injury Adverse Events of Special Interest by Category and PT - On Study (Year 1&2) | Now presents data for Year 1&2 |
| 23.35. | 23.41 | ITT | Adverse Events of Special Interest including Exposure-Adjusted Incidence Rates by Category – On Study (Year 1&2) | Now presents data for Year 1&2 |
| COVID-19 Par | ndemic Adver | se Events | | |
| 23.36. | 23.42 | ITT | Exposure Adjusted Incidence Rates of Adverse Events Over Time in Relation to COVID-19 Pandemic – On Study (Year 1&2) | Now presents data for Year 1&2 |
| Columbia-Sui | icide Severity | Rating Scale ( | C-SSRS) | |
| 23.37. | 23.45 | ITT | C-SSRS Suicidal Ideation or Behavior during On Study Period (Year 1&2) | Now presents data for Year 1&2 |
| 23.38. | 23.46 | ITT | Treatment-Emergent C-SSRS Suicidal Ideation or Behavior On Study Relative to Pre-treatment (Year 1&2) | Now presents data for Year 1&2 |
| Laboratory R | esults | | | |
| 23.39. | 23.50 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Hematology (Year 1&2) | Now presents data for Year 1&2 |
| 23.40. | 23.51 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Hematology (Year 1&2) | Now presents data for Year 1&2 |
| 23.41. | 23.54 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Liver Function (Year 1&2) | Now presents data for Year 1&2 |

| Safety Tables | Safety Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 23.42. | 23.55 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Liver Function (Year 1&2) | Now presents data for Year 1&2 |
| 23.43. | 23.58 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Electrolytes (Year 1&2) | Now presents data for Year 1&2 |
| 23.44. | 23.59 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Electrolytes (Year 1&2) | Now presents data for Year 1&2 |
| 23.45. | 23.62 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Other Chemistries (Year 1&2) | Now presents data for Year 1&2 |
| 23.46. | 23.63 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Other Chemistries (Year 1&2) | Now presents data for Year 1&2 |
| 23.47. | 23.65 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Urinalysis (Year 1&2) | Now presents data for Year 1&2 |
| 23.48. | 23.66 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Urinalysis (Year 1&2) | Now presents data for Year 1&2 |
| 23.49. | 23.69 | ITT | Worst Post-Baseline Laboratory Toxicity Grade: Immunoglobulins (Year 1&2) | Now presents data for Year 1&2 |
| 23.50. | 23.70 | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Immunoglobulins (Year 1&2) | Now presents data for Year 1&2 |
| 23.51. | 23.71 | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Immunoglobulins (Year 1&2) | Now presents data for Year 1&2 |
| Immunogenicity | | | | |
| 23.52. | 23.76 | ITT | Immunogenic Response to Belimumab SC by Visit (Year 1&2) | Now presents data for Year 1&2 |
| Vital Signs | | | | |
| 23.53. | 23.78 | ITT | Vital Signs Change from Baseline by Visit (Observed) (Year 1&2) | Now presents data for Year 1&2 |

| Safety Tables | | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Serious Adve | rse Events (a | dditional outpu | ts) | |
| 23.54. | NEW | ITT Year 2 | Serious Adverse Events by SOC and PT - On Study (Year 2) | <ul> <li>New output (formatting appropriate for CSR)</li> <li>Use new 'ITT Year 2' Population defined in Section 2.2.</li> </ul> |
| 23.55. | NEW | ITT | Serious Adverse Events by SOC and PT - On Study (Year 1&2) | New output (formatting appropriate for CSR) |

# 2.1.8. Safety Figures

There are no Safety Figures to produce.

# 2.1.9. Safety Listings

| Safety Listings | | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Adverse Even | nts | | | |
| 23.01. | 23.02 | ITT | Adverse Events (Year 2) | |
| 23.02. | 23.03 | ITT | Adverse Events Related to Belimumab SC (Year 2) | |
| 23.03. | 23.05 | ITT | Adverse Events Resulting in Belimumab SC Study Treatment Discontinuation (Year 2) | |
| 23.04. | 23.07 | ITT | Year 1 Adverse Events reported after LSLV (Year 1) | |
| 23.05. | 23.08 | ITT | Serious Adverse Events (Year 2) | |

| Safety Listing | Safety Listings | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 23.06. | 23.11 | ITT | Reasons for Considering as a Serious Adverse Event (Year 2) | |
| 23.07. | 23.13 | ITT | MedDRA coding changes (Year 2) | |
| Laboratory R | Laboratory Results | | | |
| 23.08. | 23.14 | ITT | Laboratory Results: Hematology (Year 2) | |
| 23.09. | 23.15 | ITT | Laboratory Results: Liver Function (Year 2) | |
| 23.10. | 23.16 | ITT | Laboratory Results: Electrolytes (Year 2) | |
| 23.11. | 23.17 | ITT | Laboratory Results: Other Chemistries (Year 2) | |
| 23.12. | 23.18 | ITT | Laboratory Results: Urinalysis (Year 2) | |
| 23.13. | 23.19 | ITT | Laboratory Results: Immunoglobulins (Year 2) | |
| Immunogenio | ity | | | |
| 23.14. | 23.26 | ITT | Immunogenicity Results for Belimumab SC (Year 2) | |
| COVID-19 Pandemic | | | | |
| 23.15. | 23.27 | ITT | COVID-19 Assessments and Symptom Assessments for Subjects with COVID-19 Adverse Events (Year 1&2) | |

## 2.1.10. Health Outcomes Tables

| Health Outco | Health Outcomes Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Health Outco | me Tables | | | |
| 24.01. | 24.01 | MITT | Patient Global Assessment of Disease Activity Change from Baseline by Visit (Hypothetical) (Year 1&2) | |
| 24.02. | 24.02 | MITT | Lupus Quality of Life Domain Scores Change from Baseline by Visit (Hypothetical) (Year 1&2) | |
| 24.03. | 24.03 | MITT | FACIT-Fatigue Scale Score Change from Baseline by Visit (Hypothetical) (Year 1&2) | |
| 24.04. | 24.04 | MITT | Improvement in FACIT-Fatigue Scale Score exceeding the MCID (>=4 point increase) by Visit (Hypothetical) (Year 1&2) | |
| 24.05. | 24.05 | MITT | WPAI: Overall Work Productivity Impairment Change from Baseline by Visit (Hypothetical) (Year 1&2) | |
| 24.06. | 24.06 | MITT | WPAI: Percent Activity Impairment Score Change from Baseline by Visit (Hypothetical) (Year 1&2) | |

# 2.1.11. Health Outcomes Figures

| Health Outcom | Health Outcomes Figures | | |
|---|---|---|---|
| New output number | · Population Litie Major modifications since original RAP | | |
| Health Outcom | Health Outcome Figures | | |
| 24.01. | 24.02 | MITT | Lupus Quality of Life Domain Scores Change from Baseline by Visit (Observed) (Year 1&2) |

| Health Outcom | Health Outcomes Figures | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 24.02. | 24.03 | MITT | FACIT-Fatigue Scale Score Change from Baseline by Visit (Observed) (Year 1&2) | |
| 24.03. | 24.04 | MITT | Improvement in FACIT-Fatigue Scale Score Exceeding the MCID (>=4 points increase) by Visit (Observed) (Year 1&2) | |

# 2.1.12. Health Outcomes Listings

| Health Outcor | Health Outcomes Listings | | |
|---|---|---|---|
| New output number | Major modifications since original RAP | | |
| Health Outcom | Health Outcomes Listings | | |
| 24.01. | 24.04 | ITT | Health Care Resource Utilization (Year 1&2) |

## 2.1.13. Biomarkers Tables

| Biomarkers T | Biomarkers Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Immunoglobu | Immunoglobulins | | | |
| | | Immunoglobulin Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | | |

| Biomarkers T | Biomarkers Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 25.02. | 25.03 | ITT | Immunoglobulin Levels Shifts from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| Autoantibodi | es | | | |
| 25.03. | 25.06 | ITT | Autoantibody Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| 25.04. | 25.07 | ITT | Autoantibody Levels Change from Baseline by Visit among Subjects Positive at Baseline who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| 25.05. | 25.08 | ITT | Autoantibody Levels Shifts from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| Complement | | | | |
| 25.06. | 25.11 | ITT | Complement Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| 25.07. | 25.12 | ITT | Complement Levels Change from Baseline by Visit among Subjects with Low Complement at Baseline who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| 25.08. | 25.13 | ITT | Complement Levels Shifts from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |
| B Cells, T Cel | B Cells, T Cells and B-Lymphocyte Stimulator | | | |
| 25.09. | 25.15 | ITT | B Cells, T Cells and B-Lymphocyte Stimulator Change from<br>Baseline by Visit among Subjects who Completed Week 52 On<br>Treatment (Observed) (Year 1&2) | |

# 2.1.14. Biomarkers Figures

| Biomarkers F | Biomarkers Figures | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| Biomarker Fig | gures | | | |
| 25.01. | NEW | ITT | Immunoglobulin Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | New output (omission in original RAP) |
| 25.02. | NEW | ITT | Autoantibody Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | New output (omission in original RAP) |
| 25.03. | NEW | ITT | Complement Levels Change from Baseline by Visit among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | New output (omission in original RAP) |
| 25.04. | NEW | ITT | B Cells, T Cells and B-Lymphocyte Stimulator Change from<br>Baseline by Visit among Subjects who Completed Week 52 On<br>Treatment (Observed) (Year 1&2) | New output (omission in original RAP) |

# 2.1.15. Biomarkers Listings

| Biomarkers L | Biomarkers Listings | | |
|---|---|---|---|
| New output number | · Population Litie Major monitications since original RAP | | |
| Biomarker Lis | Biomarker Listings | | |
| 25.01. | 25.01 | ITT | Biomarker Results (Year 1&2) |
| 25.02. | 25.02 | ITT | B Cells, T Cells and B-Lymphocyte Stimulator Results (Year 1&2) |

#### 2.1.16. Pharmacokinetic Tables

| PK Tables | PK Tables | | | |
|---|---|---|---|---|
| New output number | Old output number | Population | Title | Major modifications since original RAP |
| 26.01. | 26.01 | PK | Belimumab Concentrations (ug/mL) among Subjects who Completed Week 52 On Treatment (Observed) (Year 1&2) | |

# 2.1.17. Pharmacokinetic Figures

There are no PK Figures to produce.

# 2.1.18. Pharmacokinetic Listings

| PK Listings | PK Listings | | |
|---|---|---|---|
| New output number Old output number Population Title Major modifications since original RAP | | Major modifications since original RAP | |
| 26.01. | 26.01 | PK | Serum Belimumab PK Concentrations (Observed) (Year 1&2) |

#### 2.2. New 'Intent-to-Treat Year 2' Population

An additional population has been defined for use in any Study Population and Adverse Event table that presents data only for Year 2.

The 'Intent-to-Treat Year 2' population is defined as "All ITT population participants who are ongoing in Year 2. This includes subjects who confirm that they are continuing in the study for Year 2 and/or have an exposure date or early withdrawal visit after the Week 52 visit date."

#### 2.3. Biomarker and Pharmacokinetic (PK)

#### 2.3.1. Specifications in the original RAP

The original RAP gave minimal information about the data that should be used in the Biomarker and PK analyses for the Year 2 reporting.

For Biomarkers, the original RAP Section 10.1 stated that "The Year 1&2 analyses will be performed on the observed data for subjects who completed Week 52 on treatment (Ongoing and on treatment at Week 52 analysis as defined in Section 7.1.5). No imputation will be performed for missing data (data post re-start Belimumab will not be considered)."

For PK, the original RAP Section 11 gave no details.

Section 2.3.2 clarifies the approach that will be used for Year 2 reporting of both Biomarker and PK data. The intended approach for Biomarkers (described above) is utilised, explained further and broadened so that the method is also consistent for PK analyses.

#### 2.3.2. Clarifications for the Year 2 reporting

The original definition of subjects who completed Week 52 on treatment (referenced in the original RAP Section 7.1.5) was based on the MITT population as it was intended to be used for Efficacy data. However, for Biomarker and PK analyses, this needs to be modified to be based on all subjects from the ITT population. Therefore, it has been copied directly but with the ITT population as the original population as follows:

All ITT population Arm A and Arm B participants who are ongoing after 52 weeks of the planned double-blind treatment period who received all of both IV doses of rituximab or rituximab-placebo, and did not have more than 28 consecutive days from baseline to Week 51 without a belimumab dose; includes ITT population Arm C subjects who remained on open-label belimumab through Week 52 and did not have more than 28 consecutive days baseline to Week 51 without a belimumab dose.

For Arms A&B, the Year 1&2 analyses will be performed on the observed data collected in Year 1 and prior to any re-start Belimumab in Year 2, for subjects who completed Week 52 on treatment.


205646

For Arm C, the Year 1&2 analyses will be performed on the observed data up to IP discontinuation, for subjects who completed Week 52 on treatment.

No imputation will be carried out for missing data.

Note that the PK outputs will be presented for the PK population.

# Signature Page for $\,205646\ TMF\text{-}13873132\ v1.0$

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 22-Jul-2021 12:38:41 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 22-Jul-2021 14:16:22 GMT+0000 |

Signature Page for TMF-13873132 v1.0

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan Addendum |
| Title | : | Reporting and Analysis Plan Addendum for 205646, a Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 104-Week Study to Evaluate the Efficacy and Safety of Belimumab Administered in Combination with Rituximab to Adult Subjects with Systemic Lupus Erythematosus (SLE) |
| <b>Compound Number</b> | : | GSK1550188 |
| Effective Date | • | 08-OCT-2020 |

#### **Description:**

- This RAP addendum is supplemental to the RAP (Dated: 05/AUG/2020), and based on protocol amendment 04 (Dated: 30/APR/2020) of study 205646.
- The purpose of this RAP addendum is to document minor additions/clarifications made after RAP approval but before Database Release.

#### Author(s)

| Author | Date | Approval<br>Method |
|---|---|---|
| PPD | 08-OCT-2020 | eTMF |
| Statistics Leader (Rheumatology Biostatistics) | | |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

#### The GlaxoSmithKline group of companies

#### **RAP Team Confirmations:**

| Reviewer | Date | Approval Method |
|---|---|---|
| Medical Monitor (Immuno-Inflammation Clinical Development) | 08-OCT-2020 | Email filed in eTMF |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | | Date | Approval Method |
|---|---|---|---|
| PPD<br>PPD | | 08-OCT-2020 | eTMF |
| PPD | (Rheumatology Biostatistics) | | - |
| PPD | | | |
| PPD | (Rheumatology Programming) | 08-OCT-2020 | <sub>o</sub> TME |
| Delegate for PPI | | 08-OC1-2020 | eTMF |
| PPD (Rheur | matology Programming) | | |


205646

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| AB | BREVI | ATIONS | 4 |
| 1. | INTRO | ODUCTION | 5 |
| 2. | CHAN | IGES/CLARIFICATIONS TO THE RAP | 5 |
| | 2.1. | Additional Cochran-Mantel-Haenszel (CMH) analysis (RAP Section 7) | 5 |
| | 2.2. | Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K Missing Item Scores (RAP Section 15.6.3, Section 15.6.4, Section 15.6.5, Section 15.6.6 and Section 15.6.9) | |
| | 2.3. | Tipping Point Analysis (RAP Section 7.1.6) | |
| | 2.4. | Analysis method to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the Primary Endpoint (RAP Section 7.1.7.1) | |
| | 2.5. | Clarification on Missing Data for SLEDAI-2K in additional COVID-19 Analyses (RAP Section 7.1.7.4) | |
| | 2.6. | Duration of Disease Control (RAP Section 15.6.4) | |
| | 2.7. | Lupus Low Disease Activity State (LLDAS) Missing Data (RAP Section 7.4 and Section 15.6.9) | |
| | 2.8. | LLDAS – clarification of endpoint definition (RAP Section 15.6.9) | |

## **ABBREVIATIONS**

| Abbreviation | Description |
|--------------|----------------------------------------------------------|
| CI | Confidence Interval |
| CMH | Cochran-Mantel-Haenszel |
| COVID-19 | Coronavirus Disease 2019 |
| CRF | Case Report Form |
| FDA | Food and Drug Administration |
| IBA | Independent Blinded Assessor |
| LLDAS | Lupus Low Disease Activity State |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NR | Non-Responder |
| PI | Principal Investigator |
| R | Responder |
| RAP | Reporting and Analysis Plan |
| SLEDAI-2K | Systemic Lupus Erythematosus Disease Activity Index 2000 |

# **Trademarks**

| Trademarks owned by GlaxoSmithKline group of companies | Trademarks not owned by GlaxoSmithKline group of companies |
|---|---|
| None | None |

#### 1. INTRODUCTION

This RAP addendum is supplemental to the RAP (Dated: 05/AUG/2020), and based on protocol amendment 04 (Dated: 30/APR/2020) of study 205646.

The purpose of this RAP addendum is to document minor additions/clarifications made after RAP approval but prior to Database Release.

#### 2. CHANGES/CLARIFICATIONS TO THE RAP

# 2.1. Additional Cochran-Mantel-Haenszel (CMH) analysis (RAP Section 7)

The RAP specifies that CMH analysis will be conducted for

- Disease Control at Week 52: RAP Section 7.1.5.1
- Clinical Remission at Week 64: RAP Section 7.2.5.1
- Disease Control at Week 104: RAP Section 7.3.5.1

Following re-review of the FDA Request 29 June 2020 – comment 5:

To facilitate an evaluation of benefit-risk, report point estimates and 95% CI for the difference in proportions for these endpoints

It was decided that most other binary endpoints would also conduct the CMH analysis. The exceptions are the following outputs:

- Disease control at Week 52 by subgroup
- Sensitivity analyses that were unadjusted for covariates (disease control and clinical remission)
- COVID-19 additional analyses using multiple imputation methods (disease control and clinical remission)

# 2.2. Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K Missing Item Scores (RAP Section 15.6.3, Section 15.6.4, Section 15.6.5, Section 15.6.6 and Section 15.6.9)

The RAP Section 15.6.3 states the following:

"SLEDAI-2K missing scores for laboratory parameters i.e.

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Will be imputed from the previous assessment if the previous assessment is no more than 35 days prior."

For clarification, the following rules apply for SLEDAI-2K missing item scores:

- It is only the 8 lab items that can be imputed. If any of the other 16 items are missing, they will be left missing.
- An imputed assessment cannot be used to impute another assessment.
- The imputation of these missing lab items is carried out independently for the Principal Investigator (PI) and Independent Blinded Assessor (IBA), i.e. the PI assessment of the lab items will never be carried forward to a missing IBA assessment and vice versa.

The following sections of the RAP should not re-define what happens with missing SLEDAI-2K item scores, they should all use the principles stated above:

- RAP Section 15.6.4: Disease Control
- RAP Section 15.6.5: Clinical Remission
- RAP Section 15.6.6: Complete Remission
- RAP Section 15.6.9: Lupus Low Disease Activity State (LLDAS)

## 2.3. Tipping Point Analysis (RAP Section 7.1.6)

The RAP Section 7.1.6 describes the tipping point analyses only in terms of "missing data caused by study withdrawal". This description is clarified here to also include any missing/partial non-informative SLEDAI-2K data, regardless of study withdrawal.

To explicitly clarify this in terms of the two strategies, the bold text has been added to the following existing RAP text:

"The first tipping point analysis will use the Hybrid strategy (as described in RAP Section 7.1.4 as per the primary estimand). If a subject's study withdrawal (or missing data) is subsequent to treatment failure the subject will still be considered as a non-responder, i.e. the non-responder assumption will only be varied for withdrawn subjects (or subjects with missing/partial non-informative SLEDAI-2K data) that were not treatment failures

The second tipping point analysis will use the treatment policy strategy (RAP Section 7.1.4). In this approach, treatment failure data is ignored, i.e. the non-responder

assumption is varied for all withdrawn subjects (or subjects with missing/partial non-informative SLEDAI-2K data) regardless of treatment failures."

# 2.4. Analysis method to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the Primary Endpoint (RAP Section 7.1.7.1)

The RAP Section 7.1.7.1 states the following text as the first step in the method for the imputation of missing data due to COVID-19:

A bayesian repeated measures logistic regression model will be fitted to the observed data, using a Markov Chain Monte Carlo (MCMC) approach, adjusting for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day). Non-informative priors will be used.

However, the planned approach is not a repeated measures approach, it is an imputation approach that will proceed sequentially through affected visits, so the text 'repeated measures' should be removed.

# 2.5. Clarification on Missing Data for SLEDAI-2K in additional COVID-19 Analyses (RAP Section 7.1.7.4)

Table 3 in the RAP (Section 7.1.7.4) displays a graphical representation of specific scenarios for individual subjects, in terms of their completion status or any Intercurrent Events, and the timing of them in relation to the COVID-19 environment onset date.

In the existing table, there was one row for subjects who complete at Week 52 after the COVID environment onset date. To cover the scenario of missing (or partial non-informative) SLEDAI-2K data, that row has been split into two rows, as shown in Table 1 below:
Table 1
 Graphical Representation of the Additional Analyses

| | environment<br>set date | Description | Primary<br>Analysis<br>Hybrid | COVID<br>Attributed | COVID<br>Environment | Pre-<br>COVID |
|---|---|---|---|---|---|---|
| X_ | 0 Comp. | Subject Completes Week 52 on or after COVID-19 environment onset date and has a completed (or partial but informative) S2K Score | R/NR | R/NR | Imputed | Excluded |
| X_ | 0 Comp. | Subject Completes Week 52 on or<br>after COVID-19 environment onset<br>date and has a missing or partial<br>non-informative S2K Score that<br>cannot be determined to definitely be<br>either R or NR | NR | Imputed | Imputed | Excluded |

Comp. = Completed; R/NR = Responder/Non-Responder based on SLEDAI-2K criteria; NR = Non-Responder

### 2.6. Duration of Disease Control (RAP Section 15.6.4)

The formula for the duration of disease control specified in RAP Section 15.6.4 should be as follows:

Duration of disease control = longest period where

Last visit of disease control – First visit of disease control + 1

Also, it is not appropriate to derive disease control at Baseline, therefore the first visit of disease control considered in this calculation will always be the first post-baseline visit where the subject meets the disease control criteria.

# 2.7. Lupus Low Disease Activity State (LLDAS) Missing Data (RAP Section 7.4 and Section 15.6.9)

The RAP does not explicitly state what happens when the subject has missing data for a component of their LLDAS assessment. Adding these clarifying sentences would be clearer:

"Within each criteria, a subject with an incomplete assessment (due to missing data) will be considered as missing, i.e. observed data will be presented for the individual criteria.

A subject is only considered an overall responder for LLDAS if they are a responder for all 6 criteria, i.e. missing data within one or more criteria would make them an overall non-responder."

# 2.8. LLDAS – clarification of endpoint definition (RAP Section 15.6.9)

Clarifications have been made to the LLDAS endpoint definition table in RAP Section 15.6.9. for the criteria of "well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents, excluding investigational drugs".

Firstly, the RAP Section 15.6.9 and protocol Section 7.7.14 refer to "Cyclosporine", however the MedDRA dictionary name is "Ciclosporin".

Secondly the existing text in RAP Section 15.6.9 (shown below) has been clarified to include the additional text shown in bold. This additional text makes it clearer that the Anti-TNF therapy and other biologics listed are just examples and it also provides additional examples of other biologics based on the Year 1 blinded data:

"Not to be taken within 28 days prior to the assessment:

- Intravenous Cyclophosphamide
- Other investigation agent


205646

- Anti-TNF therapy (e.g. adalimumab, etanercept, infliximab)
- Other biologics (e.g. abatacept, anakinra, commercial rituximab, tocilizumab)
- IVIG
- Plasmapheresis"

The following sentence has also been added to clarify the use of commercial Belimumab: "Subjects can take commercial Belimumab IV or SC and this doesn't prevent them from being a responder on this criteria for the LLDAS.".

### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 205646, a Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 104-Week Study to Evaluate the Efficacy and Safety of Belimumab Administered in Combination with Rituximab to Adult Subjects with Systemic Lupus Erythematosus (SLE) |
|---|---|---|
| <b>Compound Number</b> | : | GSK1550188 |
| Effective Date | : | 5-AUG-2020 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205646.
- This RAP is intended to describe the planned efficacy, safety, pharmacokinetics and biomarker analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author:**

| Author | | Approval Method |
|-----------------|---------------------------------|-----------------|
| PPD | | TME |
| Statistics Lead | er (Rheumatology Biostatistics) | eTMF |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Confirmationss:**

| Reviewer | Approval Method |
|------------------------------------------------------------|-----------------|
| Medical Monitor (Immuno-inflammation Clinical Development) | eTMF |
| Statistics Leader (Immuno-inflammation Biostatistics) | eTMF |
| Programming Leader (Rheumatology Biostatistics) | eTMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | | Approval Method |
|-----------------|------------------------------|-----------------|
| PPD | | TT) (T) |
| PPD | (Rheumatology Biostatistics) | eTMF |
| PPD | | |
| PPD | (Rheumatology Programming) | eTMF |
| Delegate for PP | D | CTIVII |
| PPD (Rheu | matology Programming) | |

### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 9 |
| 2. | SUMI | MARY OF KEY PROTOCOL INFORMATION | 9 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 9 |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | 14 |
| 3. | | NED ANALYSES | |
| | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | 16 |
| 4. | ANAL | YSIS POPULATIONS | |
| | 4.1. | | |
| | 4.2. | Per Protocol Population | 20 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | /ENTIONS | 22 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Study Day | |
| | 5.3. | Baseline Definitions | |
| | 5.4. | Multicentre Studies | |
| | 5.5. | Examination of Covariates, Strata and Subgroups | |
| | | 5.5.1. Covariates and Strata | |
| | <b>5</b> 0 | 5.5.2. Examination of Subgroups | |
| | 5.6. | Multiple Comparisons and Multiplicity | |
| | 5.7. | Cut-off Date for Primary Analyses (Year 1) | 26 |
| | 5.8. | Database for End of Study Analyses (Year 2 and Years 1&2 Combined) | 27 |
| | 5.9. | Study Withdrawal | |
| | 5.10. | Treatment Failures | |
| | 5.11. | On Study. | |
| | 5.12. | On Treatment | |
| | - | Race Hierarchy (minority rule) | |
| | 5.14. | | |
| | | Conventions | 29 |
| 6. | STUD | OY POPULATION ANALYSES | 30 |
| • | 6.1. | Overview of Planned Study Population Analyses | 30 |
| | 6.2. | Disposition of Subjects | |
| | 6.3. | Demographic and Baseline Characteristics | 31 |
| | 6.4. | Concomitant Medications | |
| | 6.5. | Extent of Exposure to Study Treatment | |
| | 6.6. | Time to Study Treatment Discontinuation | |
| 7. | EFFIC | CACY ANALYSES | 40 |
| | 7 1 | | |

| | 7.1.1. | | / Variables | |
|---|---|---|---|---|
| | 7.1.2. | | Measure | |
| | 7.1.3. | | n of Interest | |
| | 7.1.4. | | or Intercurrent (Post-Randomization) Events | |
| | 7.1.5. | | Analyses / Methods | |
| | | 7.1.5.1. | Statistical Methodology Specification | 45 |
| | 7.1.6. | | oint Analysis | 47 |
| | 7.1.7. | Additiona | Analyses to Assess the Impact of the | |
| | | | rus Disease 2019 (COVID-19) Pandemic on the | |
| | | Primary E | indpoint | 49 |
| | | 7.1.7.1. | COVID Attributed – Observed Data until | |
| | | | Intercurrent Events That Could be Attributable | |
| | | | to the COVID-19 Pandemic | 49 |
| | | 7.1.7.2. | COVID Environment – Observed Data Until the | |
| | | | COVID-19 Pandemic | 50 |
| | | 7.1.7.3. | Pre-COVID – MITT Population Prior to the | |
| | | | COVID-19 Pandemic | 51 |
| | | 7.1.7.4. | Graphical Representation of the Additional | |
| | | | Analyses | 52 |
| 7.2. | First Ma | jor Second | ary Efficacy Analyses | 55 |
| | 7.2.1. | Endpoint | / Variables | 55 |
| | 7.2.2. | Summary | Measure | 56 |
| | 7.2.3. | Populatio | n of Interest | 56 |
| | 7.2.4. | Strategy f | or Intercurrent (Post-Randomization) Events | 56 |
| | 7.2.5. | | Analyses / Methods | |
| | | 7.2.5.1. | | |
| | 7.2.6. | Additiona | Analyses to Assess the Impact of the | |
| | | Coronavir | rus Disease 2019 (COVID-19) Pandemic on the | |
| | | First Majo | or Secondary Endpoint | 58 |
| | | 7.2.6.1. | COVID Attributed – Observed data until | |
| | | | Intercurrent Events that could be attributable to | |
| | | | the COVID-19 pandemic | 58 |
| | | 7.2.6.2. | COVID Environment – Observed data until the | |
| | | | COVID-19 pandemic | 58 |
| | | 7.2.6.3. | Pre-COVID – MITT Population prior to the | |
| | | | COVID-19 pandemic | 58 |
| 7.3. | Second | Major Seco | ondary Efficacy Analyses | |
| | 7.3.1. | | / Variables | |
| | 7.3.2. | Summary | Measure | 58 |
| | 7.3.3. | | n of Interest | |
| | 7.3.4. | Strategy f | or Intercurrent (Post-Randomization) Events | 59 |
| | 7.3.5. | | Analyses / Methods | |
| | | 7.3.5.1. | Statistical Methodology Specification | 59 |
| | 7.3.6. | Additiona | Analyses to Assess the Impact of the | |
| | | Coronavir | rus Disease 2019 (COVID-19) Pandemic on the | |
| | | | lajor Secondary Endpoint | 60 |
| | | 7.3.6.1. | COVID Attributed – Observed Data Until | |
| | | | Intercurrent Events That Could be Attributable | |
| | | | to the COVID-19 Pandemic | 60 |
| | | 7.3.6.2. | COVID Modified – SLEDAI 2K-Score ≤2 (IBA), | |
| | | | Without Current Immunosuppressants Without | |

| | | Current Belimumab (arms A&B), and | |
|---|---|---|---|
| | | prednisone equivalent dose of ≤5mg/day at | |
| | | Week 104 | 60 |
| 7.4. | | ow Disease Activity State (LLDAS) | 62 |
| | 7.4.1. | Endpoint / Variables | 62 |
| | 7.4.2. | Summary Measure | 62 |
| | 7.4.3. | Population of Interest | |
| | 7.4.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.4.5. | Subgroup, Supportive and Sensitivity Analyses | |
| | 7.4.6. | Statistical Methodology Specification | |
| 7.5. | | econdary Efficacy Analyses - Proportion Endpoints (Hybrid) | |
| | 7.5.1. | Summary Measure | |
| | 7.5.2. | Population of Interest | |
| | 7.5.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.5.4. | Subgroup, Supportive and Sensitivity Analyses | |
| | 7.5.5. | Statistical Methodology Specification | 64 |
| 7.6. | Other S | econdary Efficacy Analyses - Proportion Endpoints | |
| | • | ed Case) | |
| | 7.6.1. | Summary Measure | |
| | 7.6.2. | Population of Interest | |
| | 7.6.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.6.4. | Subgroup, Supportive and Sensitivity Analyses | |
| | 7.6.5. | Statistical Methodology Specification | |
| 7.7. | | econdary Efficacy Analyses - Time to Event Endpoints | |
| | 7.7.1. | Summary Measures | |
| | 7.7.2. | Population of Interest | |
| | 7.7.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.7.4. | Subgroup, Supportive and Sensitivity Analyses | 66 |
| | 7.7.5. | Statistical Methodology Specification for Time to Event | |
| | | Endpoints | |
| 7.8. | Other S | econdary Efficacy Analyses - Duration Endpoints | 69 |
| | 7.8.1. | Population of Interest | 69 |
| | 7.8.2. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.8.3. | Endpoint / Variables | |
| | 7.8.4. | Subgroup, Supportive and Sensitivity Analyses | |
| | 7.8.5. | Statistical Methodology Specification for Duration | |
| | | Endpoints | |
| 7.9. | | econdary Efficacy Analyses Continuous Endpoints | |
| | 7.9.1. | Endpoint / Variables | |
| | 7.9.2. | Summary Measure | |
| | 7.9.3. | Population of Interest | |
| | 7.9.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.9.5. | Subgroup, Supportive and Sensitivity Analyses | 70 |
| | 7.9.6. | Statistical Methodology Specification for Continuous | |
| | | Endpoints | 71 |
| 7.10. | | econdary Efficacy Analyses: SLEDAI-2K Score ≤2 (IBA), | |
| | | Current Immunosuppressant and Corticosteroids | |
| | | day | 72 |
| | 7.10.1. | Endpoint / Variables | |
| | 7.10.2. | Summary Measure | |
| | 7.10.3 | Population of Interest | 73 |

| | | 7.10.4.<br>7.10.5. | , | |
|---|---|---|---|---|
| | | | 7.10.5.1. Statistical Methodology Specification | |
| | 7.11. | Addition | nal Efficacy Analyses | |
| | 7.12. | Addition | nal Analyses to Assess the Impact of the Coronavirus | |
| | | | 2019 (COVID-19) Pandemic on the Secondary Efficacy | |
| | | | nts | 76 |
| | | apo | | |
| 8. | SAFE | TY ANAL | YSES | 77 |
| • | 8.1. | | Events | |
| | <b>.</b> | 8.1.1. | Reporting Phases | |
| | | <b>0</b> 11111 | 8.1.1.1. Pre Treatment | |
| | | | 8.1.1.2. On Treatment (Year 1 only) | |
| | | | 8.1.1.3. On Study | 77 |
| | | | 8.1.1.4. Post Withdrawal/Completion | |
| | | 8.1.2. | Adverse Events Analyses | |
| | | 8.1.3. | Deaths, Serious Adverse Events, and Survival Status | |
| | | 8.1.4. | Adverse Events of Special Interest Analyses | |
| | | 8.1.5. | Post-Injection Systemic Reactions | |
| | | 8.1.6. | Additional Adverse Event Summaries to Assess the | 04 |
| | | 0.1.0. | Impact of the Coronavirus Disease 2019 (COVID-19) | |
| | | | Pandemic | 05 |
| | 8.2. | Columb | ia-Suicide Severity Rating Scale (C-SSRS) | |
| | 0.2. | 8.2.1. | C-SSRS Suicidal Ideation or Behaviour on Study [T13.52, | 00 |
| | | 0.2.1. | T23.45] | 07 |
| | | 8.2.2. | C-SSRS Suicidal Ideation or Behavior Relative to Pre- | 07 |
| | | 0.2.2. | | 07 |
| | | 0.00 | Treatment [T13.53, T23.46]. | 67 |
| | | 8.2.3. | C-SSRS Shift Changes in Categories from Pre-Treatment | 00 |
| | | 0.0.4 | to On-Study [T13.54, T23.47] | 00 |
| | | 8.2.4. | C-SSRS Shift Changes in Categories from Year 1 to Year | 00 |
| | 0.0 | Oliminal | 2 [T23.48] | |
| | 8.3. | | Laboratory Analyses | |
| | | 8.3.1. | | |
| | | 8.3.2. | Laboratory Toxicity ≥ 2 Grade Shift Post-Baseline | |
| | | 8.3.3. | Laboratory Reference Range Shifts from Baseline by Visit | |
| | | 8.3.4. | Immunoglobulin Reference Range Shifts from Baseline by | |
| | | 0.0.5 | Visit | |
| | | 8.3.5. | Worst Laboratory Toxicity Grade Post-Baseline | |
| | | 8.3.6. | Immunoglobulin Below LLN by Visit | |
| | | 8.3.7. | Immunoglobulin Relative to LLN by Visit | |
| | | 8.3.8. | Immunogenicity | |
| | | 8.3.9. | Further Research Samples | |
| | 8.4. | | afety Analyses | |
| | | 8.4.1. | Vital Signs | |
| | | 8.4.2. | Neurological Assessment | 92 |
| _ | | | | |
| 9. | | | COMES ANALYSES | |
| | 9.1. | | al Methodology Specification for Continuous Endpoints | 93 |
| | | 9.1.1. | Additional Analyses to Assess the Impact of the | |
| | | | Coronavirus Disease 2019 (COVID-19) Pandemic | |
| | | | (Continuous Endpoints upto Week 52 and Week 64) | 95 |

| | 9.2. | Statistica 9.2.1. | I Methodology Specification for Proportion Endpoints Additional Analyses to Assess the Impact of the | 96 |
|---|---|---|---|---|
| | | | Coronavirus Disease 2019 (COVID-19) Pandemic | 97 |
| | 9.3. | Health Ca | are Resource Utilization | |
| 10. | PHAR | MACODYI | NAMIC AND BIOMARKER ANALYSES | 98 |
| | 10.1. | Biomarke | er Change and Percent Change from Baseline Analyses | 99 |
| | 10.2. | | mmunoglobulins, Autoantibodies, and Complement by | |
| | | | | 101 |
| 11. | PHAR | MACOKIN | IETIC ANALYSES | 103 |
| | 11.1. | Primary F | Pharmacokinetic Analyses | 103 |
| | | 11.1.1. | Endpoint / Variables | 103 |
| | | | 11.1.1.1 Drug Concentration Measures | 103 |
| | | 11.1.2. | Population of Interest | |
| | | 11.1.3. | Statistical Analyses / Methods | 103 |
| | | | • | |
| 12. | POPU | LATION P | HARMACOKINETIC (POPPK) ANALYSES | 104 |
| | 12.1. | Statistica | I Analyses / Methods | 104 |
| 13. | PHAR | MACOKIN | IETIC / PHARMACODYNAMIC ANALYSES | 104 |
| 14. | REFE | RENCES | | 105 |
| 15. | | | | |
| | 15.1. | | 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | | | Exclusions from Per Protocol Population | |
| | 15.2. | | 2: Protocol Defined Schedule of Activities | |
| | 15.3. | Appendix | 3: Assessment Windows | 123 |
| | | | Definitions of Assessment Windows for Analyses | 123 |
| | 15.4. | | 4: Study Phases and Treatment Emergent Adverse | |
| | | | Study Phases for Concomitant Medication | |
| | | | Treatment Emergent Flag for Adverse Events | |
| | 15.5. | | 5: Data Display Standards & Handling Conventions | |
| | | 15.5.1. | Reporting Process | |
| | | 15.5.2. | Reporting Standards | |
| | 15.6. | | 6: Derived and Transformed Data | |
| | | 15.6.1. | General | |
| | | 15.6.2. | Study Population | |
| | | 15.6.3. | SLEDAI-2K Total and Organ System Domain | |
| | | 15.6.4. | Disease Control | |
| | | 15.6.5. | Clinical Remission | |
| | | 15.6.6. | Complete Remission | |
| | | 15.6.7. | SFI FLARE INDEX | |
| | | 15.6.8. | Physicians Global Assessment (PGA) Scoring | |
| | | 15.6.9. | Lupus Low Disease Activity State (LLDAS) | |
| | | 15.6.10. | Lupus QOL Scale | 142 |
| | | 15.6.11. | Work Productivity and Activity Impairment (WPAI) | 142 |


| | | 15.6.12. | (FACIT)(FACIT) | 111 |
|---|---|---|---|---|
| | | 15 6 12 | Disease Control Without Current Immunosuppressant and | 144 |
| | | 15.0.15. | · | 115 |
| | | 15 6 14 | with Current Corticosteroids ≤ 5mg/day | |
| | | | Prednisone Equivalent Conversion | |
| | | 15.0.15. | Treatment Failure Rules During Study Conduct | |
| | | | 15.6.15.2. SLE Medication Categories | |
| | | | 15.6.15.3. General Conventions | |
| | | | 15.6.15.4. Steroids | |
| | | | 15.6.15.5. Anti-malarials | |
| | | | 15.6.15.6. Other Immunosuppressant Agents | |
| | | | 15.6.15.7. Nonsteroidal Anti-inflammatory Drugs | 155 |
| | | | (NSAIDs), Aspirin, and Acetominophen | 154 |
| | | | 15.6.15.8. Prohibited Medications | |
| | | | 15.6.15.9. Belimumab in Year 2 | |
| | | 15 6 16 | Coronavirus Disease 2019 (COVID-19) Environment | 100 |
| | | 10.0.10. | Onset Date | 156 |
| | 15.7. | Appendix | 7: Reporting Standards for Missing Data | |
| | 10.11. | 15.7.1. | Premature Withdrawals | |
| | | 15.7.2. | Missing Data | |
| | | | 15.7.2.1. Missing and Partial Dates | |
| | 15.8. | Appendix | 8: Laboratory Parameters and Toxicity Grades | |
| | | | Adverse Event and Laboratory Value Severity Grade | |
| | | | Tables | 162 |
| | 15.9. | Appendix | (9: Biomarkers | |
| | 15.10. | | c 10: Abbreviations & Trade Marks | |
| | | | Abbreviations | |
| | | 15.10.2. | Trademarks | 172 |
| | 15.11. | <b>Appendix</b> | (11: List of Data Displays | 173 |
| | | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| 16 | ΔΤΤΛΟ | HMENTS | } | 174 |
| 10. | | | ent 1: AESI Preferred Term Definitions | |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol versions:

| Protocol Revision Chronology: | | |
|---|---|---|
| Amendment 4 (Global) | 30 APR 2020 | COVID-19 amendments |
| Amendment 3 (Global) | 15-AUG-2019 | Treatment for subjects with neutropenia corrected |
| Amendment 2 (Global) | 17-NOV-2018 | Sample size increased following potential unblinding issue identified. |
| Amendment1 / ARG | 02-JUL-2018 | Argentina Specific amendment |
| Amendment1 / DEU-2 | 27-NOV-2017 | Germany Specific amendment |
| Amendment1 / DEU -1 | 23-OCT-2017 | Germany Specific amendment |
| Amendment1 / KOR- 1 | 22-JUN 2017 | Korea Specific amendment |
| Amendment 1 (Global) | 17-APR-2017 | Comments and feedback from EMA and FDA |
| Original | 16-JAN-2017 | Original |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

This the 2<sup>nd</sup> version of the Reporting and Analysis Plan, and is in keeping with additional detail to that provided in the Protocol (30 APR 2020), and the critical components document of 27FEB2018. Additional clarification has been added to text copied from the protocol when referring to the SLEDAI-2K, to clarify when referring to the independent blinded assessor assessment (IBA) and when referring to the principal investigator assessment (PI). The derivation of the endpoints (including the primary) has been clarified to be in accordance with ICH E9 R1 terminology. Additional analysis to assess the impact of the COVID-19 pandemic has been added.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the efficacy of belimumab<br>and a single cycle of rituximab<br>administered in a combination<br>regimen to adult participants with SLE | <ul> <li>Proportion of participants with a state of disease control<br/>defined as a Systemic Lupus Erythematosus Disease<br/>Activity Index (SLEDAI)- 2K (IBA) score ≤2, achieved<br/>without immunosuppressants and with corticosteroids at a<br/>prednisone equivalent dose of ≤5 mg/day at Week 52</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Secondary Objectives: Efficacy (Major) | Secondary Endpoints: Efficacy (Major) |
| Secondary: Efficacy (Major) | <ul> <li>Proportion of participants with a state of clinical remission<br/>defined as a Clinical SLEDAI-2K score (IBA) =0 (Section<br/>15.6.3), achieved without immunosuppressants and with<br/>corticosteroids at a prednisone equivalent dose of 0<br/>mg/day at Week 64.</li> </ul> |
| | <ul> <li>Proportion of participants with a state of disease control<br/>defined as a SLEDAI-2K score (IBA) ≤2, achieved without<br/>immunosuppressants and with corticosteroids at a<br/>prednisone equivalent dose of ≤5 mg/day at Week 104</li> </ul> |
| Secondary Objectives: Efficacy (Other) | Secondary Endpoints: Efficacy (Other) |
| Secondary: Efficacy (Other) | <ul> <li>Proportion of participants with a state of disease control,<br/>defined as a SLEDAI-2K score (IBA) ≤2, achieved without<br/>immunosuppressants and with corticosteroids at a<br/>prednisone equivalent dose of ≤5 mg/day, by visit</li> </ul> |
| | <ul> <li>Proportion of participants with a state of clinical remission, defined as a Clinical SLEDAI-2K score (IBA) =0 (Section 15.6.3), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit.</li> </ul> |
| | <ul> <li>Proportion of participants with a state of complete<br/>remission, defined as SLEDAI-2K score (PI) =0, achieved<br/>without immunosuppressants and with corticosteroids at a<br/>prednisone equivalent dose of 0 mg/day, sustained for at<br/>least 24 weeks.</li> </ul> |
| | <ul> <li>Proportion of participants with a state of clinical<br/>remission, defined as Clinical SLEDAI-2K score (PI) =0<br/>(Section 15.6.3), achieved without immunosuppressants<br/>and with corticosteroids at a prednisone equivalent dose<br/>of 0 mg/day, sustained for at least 24 weeks.</li> </ul> |
| | <ul> <li>Proportion of participants with a state of complete<br/>remission, defined as a SLEDAI-2K score (PI) =0,<br/>achieved without immunosuppressants and with<br/>corticosteroids at a prednisone equivalent dose of 0<br/>mg/day, by visit</li> </ul> |
| | Time to first severe flare (as measured by the modified SLE Flare Index) |
| | Time to first flare (as measured by the modified SLE Flare Index) |
| | <ul> <li>Time to disease control sustained to Week 104, defined<br/>as SLEDAI-2K score (PI) ≤2, achieved without<br/>immunosuppressants and with corticosteroids at a<br/>prednisone equivalent dose of ≤5 mg/day.</li> </ul> |

| Objectives | En | dpoints |
|---|---|---|
| | • | Time to clinical remission sustained to Week 104, defined as Clinical SLEDAI-2K score (PI) =0 (Section 15.6.3), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. |
| | • | Duration of disease control, defined as SLEDAI-2K score (PI) $\leq$ 2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of $\leq$ 5 mg/day |
| | • | Duration of clinical remission, defined as Clinical SLEDAI-2K score (PI) =0 (Section 15.6.3), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. |
| | • | Change from baseline in SLEDAI-2K score (PI) by visit |
| | • | Proportion of participants with SLEDAI-2K (PI) organ improvement by visit |
| | • | Proportion of participants with SLEDAI-2K (PI) organ worsening by visit |
| | • | Change from baseline in Physician Global Assessment (PGA) by visit |
| | • | Proportion of participants with any SLICC Damage Index worsening (change >0) compared with baseline at Week 52 and Week 104 |
| | • | Proportion of participants that meet the Lupus Low Disease Activity State (LLDAS) response criteria by visit. The LLDAS incorporates multiple measures of disease activity, specifically: (1) SLEDAI-2K $\leq$ 4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anaemia or gastrointestinal activity; (2) no new features of lupus disease activity compared with the previous assessment; (3) PGA (scale 0-3) $\leq$ 1; (4) current prednisolone (or equivalent) dose $\leq$ 7.5 mg daily; and (5) well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents, excluding investigational drugs. |
| | • | Proportion of participants with a state of disease control, defined as a SLEDAI-2K score (PI) $\leq$ 2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of $\leq$ 5 mg/day, by visit; using the principal investigators assessment of SLEDAI-2K |
| | • | Proportion of participants with a state of clinical remission, defined as a Clinical SLEDAI-2K score (PI) =0 (Section 15.6.3), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose |

| Objectives | Endpoints |
|---|---|
| | of 0 mg/day, by visit; using the principal investigators assessment of SLEDAI-2K. |
| Secondary (Safety) Objectives | Secondary (Safety) Endpoints |
| Secondary: Safety To assess the safety and tolerability of belimumab and a single cycle of rituximab administered in a combination regimen to adult participants with SLE Secondary: Safety To assess the safety and tolerability of belimumab administered in a combination regimen to adult | Incidence of adverse events (AEs) including serious AEs (SAEs) and AEs of special interest (AESIs) |
| Secondary: Patient Reported Outcomes (PROs) Objectives | Secondary: Patient Reported Outcomes (PROs) Endpoints |
| Secondary: Patient Reported Outcomes (PROs) | Change from baseline in Patient Global Assessment (PtGA) by visit |
| To assess the impact of belimumab<br>and a single cycle of rituximab<br>administered in a combination | Change from baseline in LupusQoL domain summary scores (8 domains) by visit |
| regimen to adult participants with SLE | Change from baseline in FACIT-Fatigue score by visit |
| on PROs | <ul> <li>Proportion of participants with improvement in FACIT-<br/>Fatigue score exceeding the Minimal Clinically Important<br/>Difference (MCID, ≥4) by visit</li> </ul> |
| Exploratory: Pharmacokinetics and Biomarkers Objectives | Exploratory: Pharmacokinetics and Biomarkers Endpoints |
| Exploratory: Pharmacokinetics and | Belimumab and rituximab concentrations by visit |
| Biomarkers To assess pharmacokinetics of and | Change from baseline in autoantibodies by visit |
| biomarker response to belimumab and a single cycle of rituximab | Change from baseline in peripheral blood leukocytes including B cell subsets by visit |
| administered in a combination regimen to adult participants with SLE | Change in BLyS levels from baseline by visit |
| Exploratory: Patient Reported Work<br>Productivity Objectives | Exploratory: Patient Reported Work Productivity Endpoints |
| Exploratory: Patient Reported Work Productivity To explore the impact of belimumab | <ul> <li>Change from baseline in Work Productivity and Activity<br/>Impairment (WPAI): Lupus percent overall work<br/>productivity impairment by visit</li> </ul> |
| and a single cycle of rituximab administered in a combination regimen to adult participants with SLE on patient experience and productivity | Change from baseline in WPAI: Lupus percent activity impairment score by visit |

These are the protocol defined endpoints (Protocol Section 4), protocol Section 10.4.1 Efficacy analysis then clarifies further that:

For participants who withdraw prematurely from study treatment and for whom subsequent collection of data is not possible, it will be assumed for the primary analysis that they are treatment failures. A dropout/treatment failure = non-responder (DO/TF=NR) analysis will be used .

Hence when adopting the ICH Estimands and Sensitivity Analysis in Clinical Trials E9 R1 addendum terminology, an endpoint has been defined which combines this information.

### 2.3. Study Design



| Overview of St | rudy Design and Key Features |
|---|---|
| Schedule of Activities | <ul> <li>by intravenous (IV) infusions in a double-blind manner at Weeks 4 and 6 for Arms A and B.</li> <li>In Arms A and B, a pre-medication regimen will be given before each rituximab or rituximab-placebo infusion, including methylprednisolone 100 mg IV or equivalent, an oral antihistamine, and an acetaminophen or equivalent.</li> <li>Arm C (reference) is an open-label arm with belimumab subcutaneous (SC) 200 mg/week and standard therapy for 104 weeks.</li> <li>See Section 15.2 Appendix 2: Schedule of Activities</li> </ul> |
| Treatment<br>Assignment | <ul> <li>At least 280 participants will be randomized in a 1:2:1 ratio to 1 of 3 arms: belimumab plus rituximab-placebo (Arm A, control, target N=70), belimumab plus rituximab (Arm B, combination, target N=140), or belimumab plus standard therapy (Arm C, reference, target N=70).</li> <li>Arms A and B are double-blind; participants will receive belimumab 200 mg/week for 52 weeks.</li> <li>Arm C (reference) is an open-label arm with belimumab subcutaneous (SC) 200 mg/week and standard therapy for 104 weeks. Currently available standard therapy includes continuation of immunosuppressant agents throughout the course of the study (See Protocol Section 7.7.1.4 for detailed information regarding immunosuppressant medications dosing).</li> <li>At randomization, participants will be stratified by their screening SLEDAI-2K score (≤9 vs. ≥ 10), by immunosuppressant use at screening (immunosuppressant use vs. no use), and by screening corticosteroid dose (prednisone equivalent ≤10 mg/day vs. &gt;10 mg/day)</li> </ul> |
| Interim<br>Analysis | No formal interim analyses planned for this study |

## 2.4. Statistical Hypotheses / Statistical Analyses

The primary objective of the study is to demonstrate superiority (improvement in response rate) of co-administration of belimumab plus rituximab (Arm B: Combination) over belimumab monotherapy (Arm A: Control), when comparing the primary efficacy endpoint at Week 52 in subjects with SLE.

Analysis of the primary objective will use data from the whole population and therefore includes subjects from treatment Arms A, B, and C, even though the primary objective is only comparing treatment Arms A and B. Hence an exploratory assessment of the relative performance of Arm A (Control) and Arm B (Combination) vs. standard SLE therapy (Arm C: Reference) will also be conducted using the same analysis.

The primary efficacy endpoint is defined as: the proportion of participants with a state of disease control defined as a SLEDAI-2K score (IBA)  $\leq$ 2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of  $\leq$ 5mg/day at Week 52.

**Null Hypothesis (H<sub>0</sub>):** There is no difference between Arm B

(combination) and Arm A (control) in terms of the

primary endpoint at Week 52.

Alternative Hypothesis (H<sub>1</sub>): There is a difference between Arm B (combination)

and Arm A (control) in terms of the primary

endpoint at Week 52.

A step-down sequential testing procedure will be used to control the overall type 1 error rate for comparing Arm B (combination) vs Arm A (control). With this procedure, the primary endpoint and the two major secondary endpoints will be evaluated for statistical significance based on a pre-specified sequence for interpretation (i.e., disease control at Week 52, followed by clinical remission at Week 64 and then disease control at Week 104, see Figure 1). Specifically, endpoints will be tested in the sequence above (2-sided alpha=0.05) provided that statistical significance is achieved by all prior tests. If at any point in the sequence statistical significance is not met, then subsequent endpoints in the sequence cannot be deemed statistically significant. Analyses of other efficacy endpoints will not be subject to any multiple comparison procedure.

### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

There are no formal planned interim analyses.

An independent data monitoring committee (IDMC) will review unblinded safety data on an ongoing basis until all participants have completed the 104 week study (after which monitoring may be assumed by an internal GSK committee). The IDMC will include physicians with relevant clinical expertise and a statistician, none of whom is affiliated with the sponsor. The 1st IDMC data review meeting occurred in Sept 2018 (6months after the 1<sup>st</sup> subject was randomised) and continued in approximately 6 monthly intervals. Ad hoc meetings of the IDMC can also be requested as needed to review urgent safety information or AEs. Events to be monitored during the safety review will include at a minimum all SAEs (including deaths, serious psychiatric events, and serious infections). Grade 3 and Grade 4 laboratory abnormalities, opportunistic infections (serious and nonserious), malignancies, and hypersensitivity/anaphylactic reactions during the doubleblind treatment phase (Year 1) and double-blind observational phase (Year 2) for Arms A & B and open-label treatment phase (Years 1 and 2) for Arm C. In addition, the IDMC will receive information within 72 hours of all SAEs that are life threatening or result in death. Other SAEs, all opportunistic infections, irrespective of relationship to study treatment, and protocol specified events (i.e., IgG <250 mg/dL) will be provided to the IDMC bi-weekly for review.

## 3.2. Final Analyses

There will be two database locks for this study, corresponding to the primary analyses and the end of study analyses. The primary analyses will include data up to the 52 week visits for the primary endpoint.

The primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the Week 52 visit (or Early Withdrawal visit for those subjects who withdraw from the study during Year 1).
- 2. All required database cleaning activities have been completed and final database release (DBR) has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met, including:
  - Review of Protocol Deviations through Week 52
  - Adjudication of AESI through Week 52
  - Review of treatment failures through Week 52
- 4. Randomisation codes have been distributed according to RandAll NG procedures.
- 5. Database freeze (DBF) has been declared by Data Management.

A final analysis will be conducted following the last subject completion of year 2 (including all 8 week-follow-up visits) when all required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management as described in Steps 2, 3 and 5 above

This RAP details the planned analysis for both database locks, with the expectation of an observed treatment benefit at Week 52. If the Week 52 reporting does not identify a treatment benefit, an abridged set of analysis may be conducted at the end of the study, which will be detailed in a RAP amendment or RAP addendum.

## 4. ANALYSIS POPULATIONS

During the early conduct of the study some participants in ARM C (n=29) were inappropriately identified on a laboratory report which could have unblinded the independent blinded assessors. Blinding of Arms A and B was not compromised. For this reason the sample size was increased, and a Modified Intent To Treat (MITT) population has been created to exclude the potentially unblinded (to the independent blinded assessor) Arm C subjects.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened<br>(Enrolled) | All screened candidates who sign the ICF | Screen failures and<br>Study Population |
| Randomized | <ul> <li>All participants who were randomly assigned to treatment in the study.</li> <li>Any participant who receives a treatment randomization number will be considered to have been randomized.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Intent-To-Treat<br>(ITT) | <ul> <li>All randomized participants who received at least one dose of study treatment (Belimumab or Rituximab/placebo).</li> <li>This population will be based on the treatment the subject was randomized to.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Pharmacodynamic and Biomarker</li></ul> |
| Modified Intent-<br>To-Treat (MITT) | <ul> <li>All randomized participants who received at least one dose of study treatment (Belimumab or Rituximab/placebo).</li> <li>Arm C subjects randomized prior to 07 September 2018, whose independent blinded assessor had potential to be unblinded, are excluded from this population.</li> <li>This population will be based on the treatment the subject was randomized to.</li> </ul> | <ul><li>Efficacy</li><li>Health Outcomes</li></ul> |
| Per Protocol<br>(PP) | <ul> <li>All participants in the MITT population who comply with the protocol.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.2 (Per Protocol Population) and Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population.</li> <li>The PP set will not be analysed if this population comprises more than 85% of the MITT population.</li> </ul> | • Efficacy |

These additional populations will also be considered in order to consider missing data

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Ongoing on<br>study treatment<br>at Week 52 | All MITT population Arm A and Arm B participants who are ongoing after 52 weeks of the planned double-blind treatment period who received all of both IV doses of rituximab or rituximab-placebo, and did not have more than 28 consecutive days from baseline to Week 51 without a belimumab dose; includes MITT population Arm C subjects who remained on open-label belimumab through Week 52 and did not have more than 28 consecutive days baseline to Week 51 without a belimumab dose. | Sensitivity analysis of the primary efficacy endpoint |
| Ongoing on<br>study treatment<br>at Week 64 | All MITT population Arm A and Arm B participants who are ongoing after 64 weeks who received all of both IV doses of rituximab or rituximab-placebo, and did not have more than 28 consecutive days from baseline to Week 51 without a belimumab dose; includes MITT population Arm C subjects who remained on open-label belimumab through Week 64 and did not have more than 28 consecutive days from baseline to Week 63 without a belimumab dose. | Sensitivity analysis of the 1st Major secondary efficacy endpoint |
| Completers on study treatment | All MITT population Arm A and Arm B participants who complete Week 104 who received all of both IV doses of rituximab or rituximab-placebo, and did not have more than 28 consecutive days from baseline to Week 51 without a belimumab dose; includes MITT population Arm C subjects who remained on open-label belimumab through Week 104 and did not have more than 28 consecutive days from baseline to Week 103 without a belimumab dose. | Sensitivity analysis of the 2 <sup>nd</sup> Major secondary efficacy endpoint |
| As Treated | <ul> <li>All randomized participants who received at least one dose of study treatment (Belimumab or Rituximab/placebo).</li> <li>Subjects in Arms A or B who receive one or more infusions of rituximab will be included in Arm B for the As Treated analysis. Subject in Arm B who receive two doses of rituximab-placebo (and no rituximab) will be included in Arm A.</li> </ul> | If more than 5% of subjects received the incorrect RTX treatment, then the Primary efficacy endpoint will be repeated for this population |
| | | Safety endpoints<br>if more than 5%<br>received the<br>wrong RTX |

| | | treatment, then<br>this population<br>will replace the<br>ITT for safety |
|---|---|---|
| Pharmacokinetic (PK) | All participants in the ITT population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ]. values will be considered as non-missing values). | • PK |

The following additional populations will be defined as pre-COVID-19 populations. The COVID-19 environment onset date is defined in Section 15.6.16.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| MITT Week 52<br>prior to COVID-<br>19 | <ul> <li>All randomized participants who received at least one dose of study treatment and had their first dose of study medication early enough that they should have completed their Week 52 visit prior to the COVID-19 environment onset date, i.e. their first dose of study treatment was prior to the onset date minus 52 weeks</li> <li>Arm C subjects randomized prior to 07 September 2018, whose independent blinded assessor had potential to be unblinded, are excluded from this population</li> <li>This population will be based on the treatment the subject was randomized to.</li> </ul> | • Efficacy |
| MITT Week 64<br>prior to COVID-<br>19 | <ul> <li>All randomized participants who received at least one dose of study treatment and had their first dose of study medication early enough that they should have completed their Week 64 visit prior to the COVID-19 environment onset date, i.e. their first dose of study treatment was prior to the onset date minus 64 weeks</li> <li>Arm C subjects randomized prior to 07 September 2018, whose independent blinded assessor had potential to be unblinded, are excluded from this population</li> <li>This population will be based on the treatment the subject was randomized to.</li> </ul> | • Efficacy |

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed for both the double-blind phase (Year 1) and observational phase (Year 2) separately [T11.13, T21.09, L11.07, L21.04]. The tables will display the number and percentage of subjects who experience any important protocol deviation and for each deviation type.

All protocol deviations that relate to COVID-19 will be summarized and listed for both the double-blind phase (Year 1) and observational phase (Year 2) separately [T11.14, T21.10, L11.07, L21.04]. The tables will display the number and percentage of subjects who experience any protocol deviation related to COVID-19.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP). [Version 6].

- Year 1 data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.
- Year 2 data will be reviewed by the blinded study team prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.

All deviations will be discussed and adjudicated as important or not important according to the PDMP.

This preliminary assessment of the deviation resulting in the subject being excluded from the per protocol population, but will be subject to a final review as detailed in Section 4.2.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF [T11.12, L11.06].

# 4.2. Per Protocol Population

Periodic review of the per protocol population will be conducted during the course of the study, with a final assessment made prior to unblinding the data for the Year 1 reporting.

The per protocol population will be primarily based on an assessment of the important protocol deviations. However non-important deviations or other study conduct issues may be identified during the study that warrant a subject's exclusion from the per protocol population. This will be documented in the protocol deviation adjudication


205646

meeting minutes prior to database freeze. Only protocol deviations or study conduct issues that have the potential to impact the efficacy evaluation will lead to exclusion from the per protocol population.

The per protocol population will be derived based on the Year 1 data. If Year 2 reporting (or combined Year 1&2) per protocol analysis is required it will be based on the per protocol population defined for Year 1.

Subjects excluded from the Per Protocol (PP) population will be summarized [T11.15].

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code Description | | Description | Order in TLF |
| Α | Belimumab plus Placebo | BEL SC plus PBO IV | 1 |
| В | Belimumab plus Rituximab | BEL SC plus RTX IV | 2 |
| С | Belimumab Open-Label | BEL SC plus STD Therapy | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. BEL SC plus RTX IV vs BEL SC plus PBO IV
- 2. BEL SC plus RTX IV vs BEL SC plus STD Therapy
- 3. BEL SC plus PBO IV vs BEL SC plus STD Therapy

Table 1 Treatment Descriptors, Colors, Line Style and Symbols for Reporting in Double-Blind Phase

| Treatment<br>Descriptor | Color | SAS Color | Line Style | Symbol |
|---|---|---|---|---|
| BEL SC plus PBO<br>IV | Blue | CX0000FF | Dashed | Triangle (filled) |
| BEL SC plus RTX<br>IV | Green | CX2A8307 | Long dashes | Circle (filled) |
| BEL SC plus<br>Standard Therapy | Brown | CXA05000 | Solid | Square (open) |

## 5.2. Study Day

Study day is the number of days from Belimumab study treatment start date to the study day of interest and is calculated as:

| Criteria: | Study day is: |
|------------------------------------|---------------------------------------|
| Study date < treatment start date | Study date - treatment start date |
| Study date >= treatment start date | Study date - treatment start date + 1 |

Note: Study day cannot be zero. If either date is missing the study day is missing. Further detail is provided in Section 15.6.1

### 5.3. Baseline Definitions

For all the endpoints for both the Week 52 and Week 104 analysis (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments Considered as<br>Baseline | | Baseline Used in Data Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Efficacy | | | |
| SLEDAI-2K Principal Investigator (PI) | Х | Х | Day 1 |
| SLEDAI-2K Independent Blinded<br>Assessor (IBA) | | X | Day 1 |
| SLICC Damage Index | | Х | Day 1 |
| Physician Global Assessment (PGA) | | Х | Day 1 |
| Safety and Biomarker | | | |
| Laboratory assessments (including liver chemistry, serum immunoglobulin, Anti-dsDNA/ANA, and complement C3/C4) | X | X | Day 1 |
| Biomarkers (including Antiphospholipid antibodies, PBMC, B-Cells, BLys Protein, RNA for interferon, and immunogenicity) | | X | Day 1 |
| C-SSRS | Χ | Х | Day 1 |
| PROs | | | |
| Patient Global Assessment (PtGA) | | X | Day 1 |
| FACIT-Fatigue score | | X | Day 1 |
| LupusQoL | | X | Day 1 |
| WPAI: Lupus | | X | Day 1 |

Baseline dose of corticosteroids is the 7-day average based on the 7 days **prior** to, but not including, treatment start date.

Concomitant medications are considered to be present at baseline if the start date is prior to Day 1 and the end date is on or after Day 1. Medications or events with a start date on Day 1 are considered as being on treatment (Section 15.4.1).

Adverse events (AEs) are considered pre-treatment if the start date is prior to Day 1. AEs with a start date on or after Day 1 are considered as being treatment-emergent.

Baseline flares are flares that occur on or prior to the treatment start date. Therefore, flares that occur on Day 1 are not counted as post-baseline flares.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

### 5.4. Multicentre Studies

In this multicentre global study, enrolment will be presented by country and investigative site. Countries will be grouped into geographic regions for summary presentation [T11.01] as shown in Section 5.5.2.

### 5.5. Examination of Covariates, Strata and Subgroups

#### 5.5.1. Covariates and Strata

The list of strata is based on the randomization stratification and will be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest have not been identified for planned analyses, but may be considered for post-hoc analyses.

| Category | Details |
|-------------|------------------------------------------------|
| Strata (As | SLEDAI-2K: ≤9 vs. ≥10 |
| Randomized) | Immunosuppressant: Use vs. Non-use |
| | Corticosteroid dose: ≤10 mg/day vs. >10 mg/day |

The following covariates will be included in the analysis as detailed in Section 7 Efficacy Analyses

| Covariate | Details |
|---|---|
| SLEDAI-2K: ≤9 vs. ≥10 | Derived from the principal investigators' assessment at baseline (reference level: ≥10) |
| Immunosuppressant: Use vs. Non-use | Derived from reported concomitant medications at baseline (reference level: Non-use) |
| Corticosteroid dose: ≤10 mg/day vs. >10 mg/day | Derived from reported concomitant medications at baseline (reference level: >10mg/day) |
| Covariates | No additional covariates |

### 5.5.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered for post-hoc analyses.

- If the percentage of subjects responding is small within a subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the subgroup.

| Subgroup | Categories |
|---|---|
| Age Group | <65 vs. >=65 |
| | If there are less than 10 subjects >=65, this sub group will be |
| | summarised but not analysed |
| Race | Black vs. Non-Black |
| Gender | Female vs Male |
| Country Region | USA/Canada: USA and Canada, |
| | Europe: France, Germany, Netherlands, Spain |
| | Rest of World: All other countries |
| Baseline SLEDAI | ≤9 vs. ≥10 |
| Baseline Immunosuppressant | Use vs. Non-use |
| Use | |
| Baseline corticosteroid dose | ≤10 mg/day vs. >10 mg/day (Prednisone equivalent) |
| Baseline complement level | At least one low C3/C4 vs. No low C3/C4 |
| Baseline anti-dsDNA | ≥30 IU/mL vs. <30 IU/mL |
| Baseline C3/C4 levels & anti- | At least one low C3/C4 & anti-dsDNA ≥30 IU/mL vs. Not (At least |
| dsDNA | one low C3/C4 & anti-dsDNA ≥ 30 IU/mL) |
| Baseline BLyS (free) Protein | >= 75 <sup>th</sup> Percentile vs. < 75 <sup>th</sup> Percentile |
| Baseline RNA Interferon | Low vs. High |
| Signature | |

## 5.6. Multiple Comparisons and Multiplicity

The primary comparison of interest is the comparison between Arm B (combination) vs Arm A (control) for the primary endpoint (SLEDAI-2K $\leq$ 2 (IBA)) in the MITT population. This analysis will be adjusted for baseline SLEDAI-2K ( $\leq$ 9 vs.  $\geq$ 10), baseline immunosuppressant (Use vs. Non-use) and baseline corticosteroid dose ( $\leq$ 10 mg/day vs.  $\geq$ 10 mg/day).

For the analysis of the primary and the major secondary efficacy endpoints, a step-down sequential testing procedure will be used to control the overall type 1 error rate for comparing Arm B (combination) vs Arm A (control). With this procedure, the primary endpoint aand the two major secondary endpoints will be evaluated for statistical significance based on a pre-specified sequence for interpretation (i.e. the endpoints based on SLEDAI-2K score (IBA)  $\leq$  2 at Week 52, followed by Clinical SLEDAI-2K score (IBA) =0 at Week 64 and then SLEDAI-2K score (IBA)  $\leq$  2 at Week 104, see Figure 1). Specifically, endpoints will be tested in the sequence above (2-sided alpha=0.05)

provided that statistical significance is achieved by all prior tests. If at any point in the sequence statistical significance is not met, then subsequent endpoints in the sequence cannot be deemed statistically significant. The primary endpoint will be tested at the primary analysis using the first locked database; the first and second major secondary endpoints will be tested using the end of study locked database.

An overview of the multiplicity control is provided in Figure 1.

Figure 1 Overview of Multiplicity Control



Analyses of other efficacy endpoints will not be subject to any multiplicity adjustment.

## 5.7. Cut-off Date for Primary Analyses (Year 1)

For study participants continuing in the study past the Week 52 visit, the cut-off date in the Year 1 analysis dataset will be the date of the Week 52 visit.

For participants who discontinue from the study prior to the Week 52 visit, the exit/withdrawal visit will be assigned to an assessment window as defined in Section 15.3. Exit/withdrawal visit assigned to week 52 or earlier will be included in the week 52 report; exit/withdrawal visits assigned to an assessment window from Week 60 or later, will be reported in the Week 104 analysis.

Participants who withdraw at or prior to the Week 52 visit will have their follow-up visit included in the Year 1 reporting if the follow-up visit is prior to or on the day of the last subject's Week 52 visit. Follow-up visits that occur after the last subjects' Week 52

assessment will be reported in the Year 2 reporting. Hence subjects who withdraw at or prior to Week 52 will have a cut-off date that is the earliest of their week follow-up date and the last subject's Week 52 date.

Displays for the primary analysis reporting effort will include all data collected up to and including the Year 1 cut-off date for each participant. This includes adverse events and concomitant medications with a start date less than or equal to the cut-off date.

# 5.8. Database for End of Study Analyses (Year 2 and Years 1&2 Combined)

The final database will be an accumulation of all data from both Year 1 and Year 2 including the 8-week Follow-up visit.

### 5.9. Study Withdrawal

Study withdrawal (referred to in the protocol as dropout), is the combination of subjects who withdraw, are lost to follow-up (LTFU), or die during the study

Study withdrawal is defined as any subject who withdraws from the study prior to the analysis visit of interest (e.g. Week 52, Week 64, Week 104) and does not have a visit within  $\pm$  28 days of the target analysis visit date (excluding follow up visits).

This rule is applied consistently across all efficacy endpoints. The assessment of whether or not a subject had a visit within the  $\pm$  28 day of an analysis visit (e.g. Week 52) is performed at the domain level [e.g., a subject who had visit within 28 days for SLEDAI-2K but not a SLICC ACR assessment would be assessed on their observed data for SLEDAI-2K but would be considered withdrawn (non-responder) in SLICC ACR assessment].

#### 5.10. Treatment Failures

Treatment failures are subjects meeting any of the criteria defined below, from the time they 1<sup>st</sup> met the criteria:

- Received a protocol prohibited medication
- Arm A&B: Received immunosuppressants after Week 4 rituximab infusion visit;
   Arm C: Increased immunosuppressants (at a dose higher than at baseline and Week 12) after Week 12
- Arms A&B only: Received PI prescribed re-start belimumab medication after Week 52 visit and prior to Week 104 visit
- Started any new immunosuppressant after Day 1
- Received a prednisone equivalent corticosteroid 7-day average dose of >5 mg/day after Week 26 visit
- Received a dose above the allowable level or after a protocol specified timepoint (Section 7.7.1 of the protocol) prior to Week 52 visit

Further detail is provided in Section 15.6.15 Treatment Failure Rules During Study Conduct

### **5.11.** On Study

For Year 1, on study is defined as from 1<sup>st</sup> dose of belimumab to the earliest of:

- Week 52 visit assessment
- Study withdrawal (including LTFU and Death)

However, for subjects that withdraw during Year 1, the on treatment period could end later than the on study period. In this situation the on study period will be reset such that it ends at the same time as the on treatment period.

NOTE: Some subjects who are enrolled toward the end of the enrolment period and withdraw at or near their Week 52 assessment may have some of their Year 1 on study period reported at the end of the study (Section 5.7).

For Year 2, on study is defined as from the Week 52 visit assessment\* until the date of study completion or study withdrawal (including LTFU and death).

\*Subjects who did not complete week 52 but had not withdrawn prior to Week 52, and have post Week 52 assessments will use scheduled visit date.

For Year 1&2 on study is defined as from the 1<sup>st</sup> dose of belimumab until the date of study completion or study withdrawal (including LTFU and death).

### 5.12. On Treatment

For Year 1 on treatment is defined as from  $1^{st}$  dose of belimumab to the latter of: last dose of belimumab + 28 days or last dose of rituximab + 28 days

For Year 1&2 arm C, on treatment is defined as from 1<sup>st</sup> dose to last dose of belimumab + 28 days.

For Year 2 Arms A&B on treatment is not defined as there is no on treatment reporting (as all subjects are off treatment)

## 5.13. Race Hierarchy (minority rule)

If multiple race categories are checked on the eCRF, the subject will be assigned to a unique race group based on which of the races checked appears first in the list below:

- 1. Native Hawaiian or Other Pacific Islander
- 2. American Indian or Alaska Native
- 3. Asian
- 4. African American/African Heritage
- 5. White

For example, if African American/African Heritage and Asian are both checked, then the subject will be assigned as Asian since it appears highest in the list. Race assigned based on this minority rule will be applied to all analyses related to race (as per PSAP). In the race and racial combination details table, subjects with multiple race categories checked will be reported in the race per the minority rule as well as in the multiracial category.

# 5.14. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 15.3 | Appendix 3: Assessment Windows |
| 15.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 15.6 | Appendix 6: Derived and Transformed Data |
| 15.7 | Appendix 7: Reporting Standards for Missing Data |
| 15.8 | Appendix 8: Laboratory Parameters and Toxicity Grades |
| 15.9 | Appendix 9: Biomarkers |

### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. See Study Population shells for mock displays.

### 6.2. Disposition of Subjects

The number and percentage of subjects randomized by country and site will be summarized overall and by treatment group using the Randomized population [T11.01].

The number of subjects in each population for the primary analyses (Screened, Randomized, ITT, MITT, MITT Week 52 prior to COVID-19, MITT Week 64 prior to COVID-19, Per Protocol, Ongoing at Week 52, Ongoing on study treatment at Week 52, As Treated and PK) and for the end-of-study analysis (Ongoing at Week 64, Ongoing on study treatment at Week 64, and Completed) will be summarized overall and by treatment group [T11.02, T21.01]. A summary of the reasons for the screen failures will be provided along with a listing of the subjects who were screen failures [T11.03, L11.01]. If there are any subjects who are randomized but do not receive any study treatment, they will be included on the subject disposition listing in the Randomized population, but not the ITT population.

Subject status through Week 52 (Year 1), and over the entire study (Years 1&2 Combined) will be summarized for the ITT [T11.04, T21.02] and MITT [T11.05, T21.03] populations.

For the ITT population, a summary of treatment status and reasons for discontinuation of study treatment will be produced at Week 52 and at end of study. The number and percentage of subjects who completed the study treatment as planned as well as subjects who stopped study treatment prematurely, including reasons for treatment discontinuation, will be displayed by treatment group [T11.08, T11.09, T21.04].

The cumulative number and percentage of subjects withdrawing from the study by visit will be summarized for the ITT (T11.07) population at Week 52, and at Week 104 (T21.05) and listed (L11.03, L21.02).

A Kaplan-Meier (KM) plot of time to study withdrawal will be generated to evaluate the pattern of study withdrawals/LTFU/death over time up to Week 52 [F11.01].

Subjects who withdraw (including LTFU and death) will be considered to have experienced an event (cens=0) at:

Time to study withdrawal = withdrawal date -1<sup>st</sup> Belimumab injection date +1

Subjects ongoing at Week 52 will be considered censored (cens=1) at: Time to study withdrawal = Week 52 date -1<sup>st</sup> Belimumab injection date + 1

The figure will be repeated for the Week 104 reporting with all data from Year 1 and 2 [F21.01].

Subjects completing at Week 104 will be considered censored (cens=1) at: Time to study withdrawal = Week 104 date -1<sup>st</sup> Belimumab injection date +1

For the ITT population, the subject's study completion status will be assessed to evaluate percentages of study withdrawals by treatment group as well as the reasons for study withdrawal. The number and percentage of subjects who completed through Week 52 (Week 64 and 104) and who withdrew from the study, including reasons for withdrawal, will be displayed by treatment group and overall for Year 1 and Year 1&2 separately [T11.06, T21.06]. A listing of subjects who withdrew from the study, including reason for and time to study withdrawal will also be provided. [L11.03, L21.02].

Additionally, the cumulative number and percentage of subjects who prematurely discontinued from the planned study treatment by visit will be displayed by treatment group and overall for Year 1 and 2 separately for the ITT and MITT populations [T11.10, T11.11, T21.07, T21.08].

A listing of subject disposition will be provided showing their completion status and whether they are included in each population [L11.02, L21.01].

A shift table that summarizes the differences between the levels of each stratification factor at screening compared to values used in randomization will be provided [T11.16].

The COVID-19 environment onset and end dates will be listed (L11.15, L21.09). Current COVID-19 environment onset dates are shown in Section 15.6.16

## 6.3. Demographic and Baseline Characteristics

Continuous parameters will be summarized using descriptive statistics (mean, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum). Categorical parameters will be summarized using counts and percentages.

Demographic and baseline characteristics, as well as stratification factors, will be listed for all patients [L11.08, L11.09].

The following Demographic and baseline disease activity indicators will be summarized:

| PARAMETER | SUMMARY TYPE |
|---|---|
| Medical History | |
| Past Medical Conditions [T11.22]. and Current | Categorical: presented if past [current]. |
| Medical Conditions [T11.23]. | medical history is present |
| Family History of Cardiovascular Risk Factors | Categorical: Yes, No |
| [T11.24]. | |
| Stratification Factors at Randomization [T11.2 | |
| SLEDAI-2K (PI) | Categorical: <=9, >=10 |
| Baseline immunosuppressant use | Categorical: |
| | - Use |
| | - Non-use |
| Corticosteroid dose | Categorical: |
| (prednisone equivalent) | - ≤10 mg/day |
| | - >10 mg/day |
| Demographic [T11.17, T11.18 (MITT population | |
| Age (years) | Continuous |
| | Categorical: |
| | - <=45 years, |
| | - >45 – <65 years |
| | - >=65 years |
| | o >=65 – <75 years |
| | o >=75 years |
| Country Region | USA/Canada, |
| | Europe, |
| | Rest Of World (Section 5.5.2) |
| Country | As observed |
| Corticosteroid dose | Categorical: |
| (prednisone equivalent) | - ≤5 mg/day |
| | >5 mg/day |
| Corticosteroid dose | Categorical: |
| (prednisone equivalent) | - 0 mg/day |
| 11-1-1-4/ | >0 mg/day |
| Height (cm) | Continuous |
| Weight (kg) | Continuous |
| Body Mass Index (BMI) (kg/m²) | Continuous |
| Blood Pressure [T11.21]. | Continuous |
| Heart Rate (beats/min) [T11.21]. | Continuous |
| Sex | Categorical: Female, Male |
| Ethnicity: Hispanic or Latino origin | Categorical: Hispanic or Latino origin, Not |
| B 18 110 11 11 B 11 17 | Hispanic or Latino origin |
| Race and Racial Combination Details [T11.20]. | Categorical: White/Caucasian, Asian, African |
| | American/African Heritage, Alaskan Native |
| | or American Indian, Native Hawaiian or |
| | Other Pacific Islander, and Multiracial |

| PARAMETER | SUMMARY TYPE |
|---|---|
| Baseline Disease Activity | O MINIO MATERIAL PROPERTY OF THE PROPERTY OF T |
| SLEDAI-2K score (IBA) [T11.26, T11.27 (MITT)]. | Continuous |
| | Categorical: <=9, 10-11, >=12 |
| SLEDAI-2K score (PI) [T11.26, T11.27 (MITT)]. | Continuous |
| | Categorical: <=9, 10-11, >=12 |
| PGA score [T11.26, T11.27 (MITT)]. | Continuous |
| 01100/4000 | Categorical: 0-1, >1 – 2.5, >2.5 |
| SLICC/ACR Damage Index score [T11.26, | Continuous |
| T11.27 (MITT)]. | Categorical: 0, 1, >1 Continuous |
| SLE disease duration (years) [T11.26, T11.27 (MITT)]. | Continuous |
| SLEDAI-2K (PI) by organ domain and item at | Categorical: presented if Yes |
| baseline [T11.29]. | Categorical. presented in 165 |
| Baseline immunoglobulin levels (g/L): | Continuous value |
| IgA, IgG, and IgM [T11.30]. | Categorical: |
| | - IgA: <lln (0.81="" g="" l),="">ULN (4.63 g/L)</lln> |
| | - IgG: <lln (6.94="" g="" l),="">ULN (16.18 g/L)</lln> |
| | - IgM: <lln (0.48="" g="" l),="">ULN (2.71 g/L)</lln> |
| Baseline levels of complement: | Continuous |
| C3 [mg/dL] [T11.26, T11.27 (MITT)]. | Categorical: high (>180 mg/dL), normal (90 - |
| | 180 mg/dL), low (<90 mg/dL) |
| Baseline levels of complement: | Continuous |
| C4 [mg/dL] [T11.26, T11.27 (MITT)]. | Categorical: high (>40 mg/dL), normal (10 - |
| Complement Level (T11.26, T11.27 (MITT)) | 40 mg/dL), low (<10 mg/dL) |
| Complement Level [T11.26, T11.27 (MITT)] | Categorical: At least one low C3/C4, No low C3/C4 |
| Anti-dsDNA [IU/mL] [T11.26, T11.27 (MITT)]. | Continuous |
| / with dob/w/t [ro/mit] [111.20, 111.27 (with 1)]. | Categorical: |
| | -positive (≥ 30 IU/mL) |
| | -negative (< 30 IU/mL) |
| Complement Level and anti-dsDNA Level | Categorical: At least one low C3/C4 and anti- |
| [T11.26, T11.27 (MITT)]. | dsDNA ≥30 IU/mL; Not (At least one low |
| , , , | C3/C4 and anti-dsDNA ≥30 IU/mL) |
| Proteinuria (g/24h) [T11.26, T11.27 (MITT)] | Continuous value |
| | Categorical: |
| | <=0.5 |
| | >0.5-<1 |
| | 1-<2 |
| | >=2 |
| PARAMETER | SUMMARY TYPE |
|---|---|
| Baseline autoantibody levels [T11.31]. | |
| ANA [Titer]. | Continuous Categorical: -positive (≥ 80 Titer) -negative (< 80 Titer) |
| anti-cardiolipin (aCL) | Continuous for each of aCL-lgA, aCL-lgG, aCL-lgM Categorical (Positive is >=15): -positive (if any of the three isotypes aCL-lgG, aCL-lgA or aCL-lgM are above the upper limit of normal) -negative (if at least one is non-missing and none of the isotypes above the limit of quantification) -missing (all three isotypes are missing) |
| anti-dsDNA and/or ANA positive | Categorical: Yes, No |
| Beta-2-glycoprotein [U/mL]. for each of the | Continuous |
| isotypes IgG, IgA, and IgM | Categorical: Positive (>=21 U/mL), Negative |
| Lupus anticoagulant | Continuous |
| RNA Interferon Signature [T21.16] | Continuous |
| | Categorical: Low, High |
| B cells and T-cells at Baseline [T11.32] | |
| CD19+ Total B cells (cells/mL) B cells CD20+ (cells/mL) B cells CD20+ (%) Naive B cells IgD+ (cells/mL) Naive B cells IgD+ (%) Naive CD20+ CD27- (cells/mL) Naive CD20+ CD27- (%) Activated Total B cells CD95+ (cells/mL) Activated Total B cells CD95+ (%) Memory CD20+ CD27+ (cells/mL) Memory CD20+ CD27+ (cells/mL) Memory CD20+ CD27+ (%) Non-switched memory CD27+ IgD+ (cells/mL) Non-switched memory CD27+ IgD- (cells/mL) Switched memory CD27+ IgD- (cells/mL) Switched memory CD27+ IgD- (%) Plasmablasts CD27b CD38b (cells/mL) Plasmablasts CD20+ CD27b CD38b (cells/mL) Plasmablasts CD20- CD27b CD38b (cells/mL) Plasmablasts CD20- CD27b CD38b (%) Plasmablasts CD20- CD27b CD38b (%) | Continuous |

| PARAMETER | SUMMARY TYPE |
|---|---|
| Transitional CD10+ CD24b CD27- CD38b | |
| (cells/mL) | |
| Transitional CD10+ CD24b CD27- CD38b (%) | |
| Transitional CD24b CD27- CD38b (cells/mL) | |
| Transitional CD24b CD27- CD38b (%) | |
| CD3+ Total T cells (/uL) | |
| CD8+ T cells (/uL) | |
| CD4+ T cells (/uL) | |
| BLyS (free) [ng/mL] . | Continuous |
| | Categorical: below limit of quantification |
| | [LOQ]. (<0.05 ng/mL), above LOQ; <75th |
| | percentile, >=75 <sup>th</sup> percentile |
| Columbia Sujaida Savaritu Datina Saala (C.SS | DS) of Papalina [T44 22] |
| Columbia Suicide Severity Rating Scale (C-SS C-SSRS responses by behavior and ideation | Categorical: |
| components for lifetime and over the last six | -Ideation: categories 1-5 with corresponding |
| months | text |
| | -Behavior: categories 6-10 with |
| | corresponding text |
| | -Self-injurious behavior, no suicidal attempt |
| | · · |
| Patient Reported Outcomes (PROs) [T11.28] | |
| Patient Global Assessment (PtGA) | Continuous |
| Baseline FACIT-Fatigue scale score | Continuous |
| LuquaOal | Categorical: (<20; 20-<35; ≥35) Continuous |
| LupusQoL<br>WPAI: Lupus | Continuous |
| Allowable SLE Medication Usage at Baseline [ | |
| Allowable SLE medications by class and drug | Categorical: |
| 7 Miowable GLE medications by class and drug | Steroids, Anti-malarials, |
| | Immunosuppressants, Aspirin, NSAIDs |
| Average daily prednisone dose (mg/day) at | Continuous |
| Average daily prednisone dose (mg/day) at baseline | Continuous Categorical: (0. >0 - ≤5. >5) |
| Average daily prednisone dose (mg/day) at baseline | Continuous<br>Categorical: (0, >0 - ≤5, >5) |
| baseline Steroid, Anti-malarial and Immunosuppressant | |
| baseline | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only |
| baseline Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only |
| baseline Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only -Anti-malarial Only |
| baseline Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only -Anti-malarial Only -Steroid and Immunosuppressant Only |
| baseline Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only -Anti-malarial Only -Steroid and Immunosuppressant Only -Steroid and Anti-malarial Only |
| baseline Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only -Anti-malarial Only -Steroid and Immunosuppressant Only -Steroid and Anti-malarial Only -Immunosuppressant and Anti-malarial Only |
| Steroid, Anti-malarial and Immunosuppressant | Categorical: (0, >0 - ≤5, >5) Categorical: -Steroid Only -Immunosuppressant Only -Anti-malarial Only -Steroid and Immunosuppressant Only -Steroid and Anti-malarial Only |

Listings will be provided for current and past medical conditions [L11.10, L21.05].

The summary of demographic and baseline characteristics, baseline disease activity and allowable SLE medication will be repeated for the following subgroups:

- Age (<65 years, ≥65 years) [T11.40, T11.41, T11.42]
- Race (Black vs. Non-Black) [T11.43, T11.44, T11.45]
- Baseline SLEDAI-2K score (≤ 9 vs. ≥ 10) [T11.46, T11.47, T11.48]
- Baseline Immunosuppressant use (use vs. non-use) [T11.49, T11.50, T11.51]
- Baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day) [T11.52, T11.53, T11.54]
- Gender (Male vs Female) [T11.55, T11.56, T11.57]
- Country Region (USA/Canada, Europe, Rest of World) [T11.58, T11.59, T11.60]
- Baseline complement level (At least one low C3/C4 vs. No low C3/C4) [T11.61, T11.62, T11.63]
- Anti-dsDNA (≥ 30 IU/mL vs < 30 IU/mL) [T11.64, T11.65, T11.66]
- Baseline C3/C4 levels & anti-dsDNA (At least one low C3/C4 & anti-dsDNA ≥30 IU/mL vs. Not (At least one low C3/C4 & anti-dsDNA ≥ 30 IU/mL)) [T11.67, T11.68, T11.69]
- Baseline BLyS Protein (>=75th Percentile vs <75th Percentile) [T11.70, T11.71, T11.72]
- RNA Interferon Signature (Low vs. High) [T21.17, T21.18, TT21.19]

# 6.4. Concomitant Medications

Concomitant medications will be coded according to drug name as defined in the GSK Drug Dictionary, and classified according to the GSK-Drug ATC classification level 1 and ATC level 4. Concomitant medications are defined as medications that start on or before the first dose date of study treatment and end on or after the first dose date of study treatment, or medications that start after the first dose date of study treatment (see Section 15.4.1 for further details). Note that medications with partial or missing start and/or stop dates will be assumed to be concomitant unless there is evidence through comparison of partial dates to suggest otherwise, for example if the day is missing, then the month and year will be compared to the month and year of the first dose date of study treatment and if the month and year are the same or later, then the medication will be considered concomitant (see Section 15.7.2.1 for further details).

A summary of the number and percentage of subjects with concomitant medications by ATC level 1 term and ATC level 4 term will be displayed for both Year 1 and Year 2 separately [T11.35, T21.11]. A further summary of concomitant medications by ATC level 4 term and preferred term will be provided for both Year 1 and Year 2 [T11.36, T21.12]. A listing of all concomitant medication data will be displayed by treatment and subject [L11.11, L21.06].

Protocol-prohibited medication and allowable medication that results in treatment failure designation (see Section 7.7 of the protocol) will be summarized by treatment group. [T11.37, T21.13].

A listing of protocol-prohibited medication and allowable medication that result in treatment failure designation will be displayed by treatment and subject [L11.12, L21.07].

# 6.5. Extent of Exposure to Study Treatment

Exposure listings detail the amount of planned study medication that was taken, and restart medication (belimumab taken in Year 2 for Arms A and B). However they do not include concomitant medication of non-study belimumab or rituximab.

Exposure data for both belimumab and rituximab will be listed for:

- Year1: Arm A, B, and C for belimumab; and Arms A and B for rituximab/placebo in Year 1 [L11.13].
- Year 2: Arm A&B: Includes late Year 1 doses (taken in year 2) for Belimumab and re-start Belimumab; Arm C belimumab in Year 2 [L21.08].

See Section 15.6.2 for further details.

#### Belimumab

The extent of exposure to belimumab through Week 52 for Arm A and Arm B and through Week 104 for Arm C will be assessed by examining the duration of exposure to belimumab in days and the total number of injections a subject receives. Duration of exposure in days will be calculated as:

Duration of exposure (days) = (Last injection date - First injection date + 7).

Only complete dates will be used when calculating duration of exposure. First and last injection dates will be used, regardless of any missed doses.

Percent compliance will be calculated as:

100\* (Number of injections prescribed – Number of injections missed)/Number of injections prescribed.

The duration of exposure, the total number of injections, and the percent compliance will be summarized using descriptive statistics for the treatment phase. The total number of injections will also be summarized using counts and percentages using the following categories: 1 - 12 doses, 13 - 24 doses, 25 - 36 doses, 37 - 52 and > 52 doses (if applicable). [T11.38]. Similarly, exposure to belimumab in Arm C from Baseline to Week 104 will also be summarized using the following categories: 1 - 12 doses, 13 - 24 doses, 25 - 36 doses, 37 - 52 doses, 53 - 64 doses, 65 - 76 doses, 77 - 88 doses, 89 - 104 doses, and > 104 doses (if applicable) [T21.14].

Exposure to belimumab will also be summarized for subjects during Year 2 only. For subjects in Arms A and B this will include incorrectly taken Year 1 medication after

Week 52 and re-start medication [T21.15]. The first dose in Year 2 will be the 1<sup>st</sup> dose the subject took on the day of or after the Week 52 visit date.

Duration of exposure (days) = (Last injection date - First injection date + 7).

#### Rituximab

For subjects randomized to Arms A and B, the extent of exposure to rituximab/rituximab-placebo will be assessed by examining the dose intensity and the total number of infusions, i.e. 0, 1 or 2. Dose intensity in mg will be calculated as the cumulative actual dose divided by 2. If the total volume of an infusion is not administered, the actual dose infused for that visit will be calculated as:

Actual Dose infused (mg) = Planned Dose (mg) \* Percentage of volume infused

Dose intensity and total number of infusions will be summarized using descriptive statistics [T11.39].

#### **Data Listings**

Subjects for whom the treatment blind was broken [L11.14], or potentially the treatment blind broken (29 subjects inappropriately identified on a lab report) will be provided [L11.02].

# 6.6. Time to Study Treatment Discontinuation

This only includes the belimumab study medication as prescribed in Year 1 (and Year 2 for Arms C) i.e. this does not include re-start belimumab for subjects in Arms A&B in Year 2.

Year 1 (all arms) and Year 1&2 for Arms A&B only

- If the last dose of belimumab+10 days is prior to the Week 52 visit date (where Week 52 visit date is as observed, or predicted as day1+364 for subjects who do not have a Week 52 visit) then the subject has discontinued treatment (had the event / CENSOR=NO=0) at the earliest non-missing date of (last dose date +7, date of death, withdrawal date, LTFU date)
- If the last dose of belimumab + 10 days is on or post the Week 52 visit date (where Week 52 visit date is as observed, or predicted as day1+364 for subjects who do not have a Week 52 visit) then the subject has a censored time to discontinued treatment (does not have the event / CENSOR=Yes=1) at the earliest non-missing date of (observed or predicted Week 52 visit date, death date, withdrawal date, LTFU date)

Year 1&2 for arm C only

- If the last dose of belimumab + 10 days is prior to the Week 104 visit date (where Week 104 visit date is as observed, or predicted as day1+728 for subjects who do not have a Week 104 visit) then the subject has discontinued treatment (had the event / CENSOR=NO=0) at the earliest non-missing date of (last dose date +7, date of death, withdrawal date, LTFU date)
- If the last dose of belimumab + 10 days is on or post the Week 104 visit date (where Week 104 visit date is as observed, or predicted as day1+728 for subjects who do not have a Week 104 visit) then the subject has a censored time to discontinued treatment (does not have the event / CENSOR=Yes=1) at the earliest non-missing date of (observed or predicted Week 104 visit date, death date, withdrawal date, LTFU date)

A KM plot of time to belimumab treatment discontinuation will also be generated [F11.02]. The figures will be repeated for the Week 104 reporting with all data from Year 1 and 2 combined [F21.02]. Due to the design of the study Arms A & B will be truncated at the end of Year 1. A listing of subjects who discontinued belimumab or Rituximab treatment, including reason will be produced [L11.04, L11.05, L21.03].

#### 7. EFFICACY ANALYSES

The primary objective of the study is to demonstrate superiority (improvement in response rate) of co-administration of belimumab plus rituximab (Arm B: Combination) over belimumab monotherapy (Arm A: Control), when comparing the primary efficacy endpoint at Week 52 in subjects with SLE.

An exploratory summary of Arm B (Combination) vs Arm C (Reference) will also be shown.

SLEDAI-2K score has been measured by both the principal investigator (PI) and the independent blinded assessor (IBA). The key differences between these assessments is the frequency of assessment and awareness of the treatment allocation for Arm C:

- The principal investigator conducts a SLEDAI-2K assessment every 4 weeks in Year 1 (at least every 8 weeks in Year 2), whereas the independent blinded assessor conducts a SLEDAI-2K assessment at a reduced set of key time points (weeks baseline, 12, 26, 40, 52, 64, 80, and 104).
- The principal investigator knows which of their subjects are randomised to treatment arm C, but does not know if their remaining subjects are randomised to arm A or arm B. The independent blinded assessor however is not aware of any MITT population subject's treatment randomisation (Section 4).

Due to the level of blinding the primary and major secondary efficacy endpoints will be conducted using the independent blinded assessors' SLEDAI-2K assessment. Note however the PI assessment of SLEDAI-2K at baseline, is used as the baseline covariate in all adjusted analysis (the baseline SLEDAI-2K assessment is conducted prior to randomisation).

The other secondary endpoints analysis utilises the greater visit frequency of the principal investigator assessment. This is particularly pertinent for differentiating between treatments when considering time to response or duration of response. In by visit summaries, it also allows for the assessment of fluctuating response.

The primary and major secondary efficacy endpoints are repeated using the principal investigator assessment.

Details of the planned displays are provided in Section 15.11 and are based on GSK data standards and statistical principles. Listings of all key efficacy endpoints will be provided [L12.01 – L12.02, and L22.01-L22.02].

# 7.1. Primary Efficacy Analyses

# 7.1.1. Endpoint / Variables

The protocol defined primary endpoint is the proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (IBA), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of ≤5mg/day at Week 52 (Protocol Section 4).

The protocol Section 10.4.1 Efficacy analysis then clarifies that:

For participants who withdraw prematurely from study treatment and for who subsequent collection of data is not possible, it will be assumed for the primary analysis that they are treatment failures. A dropout/treatment failure = non-responder (DO/TF=NR) analysis will be used.

Hence when adopting the ICH Estimands and Sensitivity Analysis in Clinical Trials E9 R1 addendum terminology, this endpoint is defined as:

#### **Disease Control**

#### Responder:

- SLEDAI-2K score ≤2 (IBA); and
- Not a TF at the current or any prior visit (TF includes consideration of corticosteroids and immunosuppressants); and
- Did not withdraw from the study prior to the visit

#### Non-Responder:

- SLEDAI-2K score >2 (IBA); or
- TF at the current or any prior visit (TF includes consideration of corticosteroids and immunosuppressants); or
- Withdrew from the study prior to visit (which includes study withdrawal, lost to follow-up and death)

The derivation of SLEDAI-2K score is provided in Section 15.6.3, treatment failures are defined in Section 15.6.15. and withdrawal from the study prior to Week 52 in Section 5.9.

Note: Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint, subjects who discontinue investigational product will only be non-responders if they also meet one of the criteria above.

Note this clarification of notation does not change the protocol-specified primary analysis.

The analysis of the primary endpoint of Arm A vs Arm B will use data from treatment Arms A, and B only.

An exploratory analysis of the relative performance of Arm B vs. Arm C will also be conducted, using data from Arms B and C only.

# 7.1.2. Summary Measure

The odds ratio at Week 52 between Arm B (Combination) vs Arm A (Control).

# 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

There are 5 potential types of intercurrent events considered for this study:

- Treatment Failure
- Study Withdrawal
- Lost to Follow-up
- Death
- Investigational Product (IP) Discontinuation.

Whilst study withdrawal and lost to follow-up (LTFU) are not true intercurrent events per ICH Estimands and Sensitivity Analysis in Clinical Trials E9 R1 addendum terminology; they are included in the reporting here to allow for backward compatibility to the study Protocol (see Section 7.1.1).

Four intercurrent event strategies are employed:

- Hybrid strategy considers all data while the subject is continuing in the study
  irrespective of IP discontinuation. Treatment failure and study withdrawal (including
  LTFU and death) are components of the endpoint definition. Subjects who
  discontinue investigational product (belimumab) are encouraged to continue in the
  study.
- <u>Composite strategy</u> considers data collected only while the subject is continuing to receive study treatment. Treatment failure and study withdrawal (including LTFU and death), and IP discontinuation are components of the endpoint definition.
- Hybrid on treatment strategy considers data collected only while the subject is receiving study treatment. Treatment failure and study withdrawal (including LTFU and death), are components of the endpoint definition. IP discontinuation are excluded (unless already experienced treatment failure).
- <u>Treatment Policy</u> strategy considers all data while the subject is continuing in the study irrespective of IP discontinuation or Treatment Failure. Study withdrawal (including LTFU and death), are components of the endpoint definition

The main estimand of this endpoint, is a Hybrid strategy, subjects who discontinue investigational product will continue in the study, assessments after treatment discontinuation will be included in the main estimand. Subjects who are a treatment failure or withdraw from the study will be a non-responder for this estimand.

An analysis of 3 supportive estimands will also be conducted using the alternative intercurrent event strategies, namely:

Composite,

This will include IP discontinuation as an intercurrent event resulting in the subject being a non-responder.

• Hybrid On treatment,

This will only include subjects whilst they are on treatment, or if they have met the definition of a non-responder prior to discontinuing treatment.

• Treatment Policy,

Assessments after IP discontinuation and assessments after Treatment Failure will be included. Subjects who withdraw from the study will be non-responders.

The impact of the different IP discontinuation components of the endpoint for the Hybrid and composite estimands is summarised by considering 6 hypothetical scenarios:

Table 2 Scenarios for the components of the Hybrid and composite endpoint

| Example<br>Subject | SLEDAI-2K score at Week 52 | Study<br>Withdrawal(including<br>Lost to Follow-up, or<br>Death) prior to Week 52 | Treatment<br>Failure<br>prior to<br>Week 52 | IP<br>Discontinuation<br>prior to Week<br>52 | Main Estimand<br>Hybrid | Supplemental<br>Estimand<br>Composite |
|---|---|---|---|---|---|---|
| 1 | >2 | N | N or Y | N or Y | NR | NR |
| 2 | <=2 | N | N | N | R | R |
| 3 | <=2 | N | N | Υ | R | NR |
| 4 | <=2 | N | Υ | N or Y | NR | NR |
| 5 | Incomplete* or entirely missing Missing - does not exist due to | N | N or Y | N or Y | NR | NR |
| 6 | study withdrawal | Υ | N or Y | Υ | NR | NR |

R = Responder; NR = Non-Responder

A full breakdown of scenarios 'by subject type' and including Hybrid On Treatment and Treatment Policy is provided in Section 15.6.4

<sup>\*</sup>Incomplete: does not include partial scores where it is possible to determine that the total score must be >2, or that the maximum possible score (assuming worst case for missing data) is <=2 (see Section 15.6.4 Partial but informative SLEDAI-2K score).

# 7.1.5. Statistical Analyses / Methods

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

• The proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (IBA), achieved without treatment failure or study withdrawal

#### Derivation

• Derivation of the endpoint for Arms A, B and C is provided in Section 15

# **Model Specification**

- Logistic regression model.
- Terms in the model:
  - **Dependent:** response (yes/no)
  - Categorical: treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day).

#### **Model Checking & Diagnostics**

- If any factor fails to converge it will be removed from the logistic model.
- If the logistic model fails to converge, e.g., due to a small number of responders, the primary endpoint will be analyzed using a Fishers exact test.
- If the model diagnostics raise questions about the validity of the analysis additional nonparametric analysis will also be conducted.

#### **Model Results Presentation**

- The table [T12.01] will display:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group,
  - the observed difference in percentage of responders for the comparison of Arm B vs Arm A; and Arm B vs Arm C,
  - the stratified (baseline SLEDAI-2K score, baseline immunosuppressant use, baseline corticosteroid dose) Cochran-Mantel-Haenszel treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A.
- A table [T12.02]. showing the details from the logistic regression will also be presented; including:
  - the parameter estimate and standard error for each of the terms in the model
  - the odds ratio and 95% CI and p-value for each covariate in the model
  - the parameter estimate, standard error, odds ratio, 95% CI and p-value for the comparison of Arm B vs Arm A

- the parameter estimate, standard error, odds ratio, and 95% CI for the comparison of Arm B vs Arm C
- the odds ratio and 95% CI for the comparison of Arm A vs Arm C
- The proportion of participants with a state of disease control at Week 52 will be displayed in a point estimate +/- SE figure, by treatment group [F12.01].

# **Subgroup Analyses**

The comparison of the primary efficacy endpoint between Arm B vs. Arm A will be performed by the following subgroups [F12.02]:

- Age (<65 years vs. ≥65 years) [T12.16].
- Race (Black vs. Non-Black) [T12.17].
- Gender (Male vs. Female) [T12.18]
- Baseline SLEDAI-2K score (≤ 9 vs. ≥ 10) [T12.19].
- Baseline immunosuppressant use (use vs. non-use) [T12.20].
- Baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day) [T12.21].
- Baseline C3/C4 levels & anti-dsDNA (At least one C3/C4 low & anti-dsDNA >= 30 IU/mL vs. NOT (At least one C3/C4 low & anti-dsDNA >= 30 IU/mL)) [T12.24].
- BLyS Protein at baseline (>= 75<sup>th</sup> Percentile vs. < 75<sup>th</sup> Percentile) [T12.25].
- Country Region (USA/Canada vs. Europe vs. Rest of World) [T12.26].
- Baseline complement level (At least one low C3/C4 vs. No low C3/C4) [T12.22].
- Anti-dsDNA (<30 IU/mL vs. >=30 IU/mL) [T12.23]
- RNA Interferon Signature at baseline (Low vs. High) [T22.34] (note this assessment of subgroups for the primary endpoint will be reported at the end of the study).

Each of the subgroups will be analysed separately using a logistic regression model with adjustment for the stratification factors, using the Intercurrent event strategy: Hybrid. If the model fails to converge the relevant stratification factor(s) will be removed from the model.

To further assess each subgroup, the interaction between treatment and the subgroup will be tested by fitting a logistic regression model to the data (all subgroups combined). The model, will include the stratification factors, the variable for the subgroup, and the interaction term between treatment group and the subgroup. The summary table will include the p-value for the interaction that tests the of stability of Arm B vs Arm A over the 2 (or more) levels of the subgroup. If the logistic model fails to converge then the interaction p-value will not be presented.

# Supportive Analyses

- The disposition of the primary endpoint, detailing the reasons why a subject was a non-responder will be summarized (n,%) [T12.03, T12.04].
- The components of the primary endpoint will be summarized [T12.05]. i.e. proportion of participants with:
  - SLEDAI 2K-score ≤2 (IBA)
  - Treatment failure due to corticosteroid use
  - Treatment failure due to immunosuppressant use
  - Treatment failure due to anti-malarial, NSAID, Aspirin or other prohibited medication use
  - Study withdrawal
- The table will include

- the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group
- the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
- the p-value for the odds ratio the treatment difference for Arm B vs Arm A
- The primary efficacy analysis at Week 52 will be repeated to assess the robustness of the primary efficacy results:
  - ITT population –Including subjects where the independent blinded assessor was potentially unblinded at Week 52. Intercurrent event strategy: Hybrid [T12.06].
  - Unadjusted for covariates, the only independent variable in the model will be treatment group. Intercurrent event strategy: Hybrid [T12.07].
  - Composite. Intercurrent event strategy: Composite [T12.08].
  - Hybrid On treatment. Intercurrent event strategy: Hybrid On Treatment [T12.10].
  - Treatment Policy. Intercurrent event strategy: Treatment Policy [12.11].
  - Per Protocol population. Intercurrent event strategy: Hybrid[T12.09].
  - Ongoing on study treatment at Week 52 population. Intercurrent event strategy: Hybrid on Treatment [T12.12].
- A supportive analysis that considers all the data from Arms A, B, and C in the same model will
  also be conducted. Estimates of the treatment effect will be made for comparison of Arms A vs
  B and Arms B vs C. Intercurrent event strategy: Hybrid (T12.13)
- Two tipping point analyses may be performed if there is a significant treatment difference, including all recorded data up to the time of study withdrawal, and using differing assumptions regarding data missing following study withdrawal (Section 7.1.6). Intercurrent event strategy: Hybrid [T12.14, F12.03]. Intercurrent event strategy: Treatment Policy [T12.15, F12.04].

# 7.1.6. Tipping Point Analysis

Tipping point analyses will be performed for the primary endpoint if the endpoint is statistically significant and it is plausible that missing data caused by study withdrawal could alter the conclusions of the analysis (treatment p-value is  $\leq 0.05$  and > 0.001). If the tipping point analyses are needed, they will be performed shortly after the Statistical Analysis Complete milestone has been met and will be presented in the clinical study report.

The tipping point analyses will be based on the Intent-to-Treat population. Only the subjects in the belimumab plus placebo, and belimumab plus rituximab arms will be considered.

For the primary analysis, subjects for whom the Week 52 disease control status cannot be determined due to study withdrawal (including lost to follow-up, and death) are imputed as non-responders. In contrast, the missing data due to study withdrawal in the tipping point analysis is evaluated using multiple imputation methods, by simulating all combinations of response probability in the treatment arms independently.

The first tipping point analysis will use the Hybrid strategy (as described in Section 7.1.4 as per the primary estimand). If a subject's study withdrawal is subsequent to treatment failure the subject will still be considered as a non-responder, i.e. the non-responder assumption will only be varied for withdrawn subjects that were not treatment failures.

The second tipping point analysis will use the treatment policy strategy (Section 7.1.4). In this approach, treatment failure data is ignored, i.e. the non-responder assumption is varied for all withdrawn subjects regardless of treatment failures.

The tipping point analyses will not consider covariates. However, if the conclusions of the primary analysis adjusting for covariates differ from the conclusions of the unadjusted analysis, a post hoc analysis assessing the impact of covariate adjustment in the tipping point analyses may be performed.

The following multiple imputation method will be implemented:

- 1. For subjects in Arm A (belimumab plus placebo) and Arm B (belimumab plus rituximab) with missing Bernoulli outcomes, a grid of the probability of response varying from 0.025 to 0.975 by 0.025 will be created. This will create all combinations, from low to high response probability, for subjects with a missing response.
- 2. For a given of probability (e.g., 0.025 for Arm A, 0.500 for Arm B)
  - a. An incidence of the number of additional responders for Arm A (Arm B) given the number of Arm A (Arm B) subjects with missing outcome and the probability assumed (e.g., 0.025 (e.g., 0.500)) will be simulated using the binomial distribution.
  - b. The statistics (sample mean and standard error) will be calculated and used to construct the Mantel-Haenszel Chi-Square test.

Steps 2a and 2b will be repeated 1000 times, and Rubin's rules applied to combine them, in order to obtain a single p-value for each given probability combination.

Heat maps will be produced (Figure 2) to show the results of the multiple imputation tipping point analyses for disease control at Week 52. The black lines on each heat map will represent a plausible scenario whereby the probability of response for the missing data in Arms A and B will be equal to the observed case response rate on the control arm (Arm A: belimumab plus placebo).



Figure 2 Tipping Point for Disease Control at Week 52

Percentage of Belimumab SC plus Rituximab IV responders

A tipping point analysis will also be performed for the key secondary endpoints if there is hierarchical significance for the endpoint, and it is plausible that the imputation strategy for missing data could alter the conclusions of the analysis (treatment p-value is  $\leq 0.05$  and > 0.001).

# 7.1.7. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the Primary Endpoint

Additional analyses will be carried out to assess the impact of the COVID-19 pandemic on the primary endpoint. The additional analyses will utilise the COVID-19 environment onset date (Section 15.6.16) to establish which data might be affected by COVID-19.

# 7.1.7.1. COVID Attributed – Observed Data until Intercurrent Events That Could be Attributable to the COVID-19 Pandemic

The first additional analysis (T12.40) uses the observed SLEDAI-2K data, as long the subject has not experienced a treatment failure or study withdrawal that could have been attributable to COVID-19 (i.e. after the COVID-19 environment onset date).

A Hypothetical estimand will be used to estimate the treatment effect had the COVID-19 pandemic not occurred. The difference in response rates between Arm A and Arm B at Week 52 will be assessed for subjects who:

- achieve a SLEDAI 2K-score ≤2 (IBA),
- without immunosuppressants that could be attributable to the COVID-19 pandemic and
- with corticosteroids at a prednisone equivalent dose of ≤5mg/day, in the absence of higher doses that could be attributable to the COVID-19 pandemic

The full MITT population will be used, with the following attributes:

- A strategy that matches the primary analysis (Hybrid) will be used for the following Intercurrent Events to classify the subject as a Non-Responder:
  - Study Withdrawal (includes Lost to Follow Up) that occurs prior to the COVID-19 environment onset date
  - Treatment Failure (includes consideration of corticosteroids and immunosuppressants) that occurs prior to the COVID-19 environment onset date
  - Death that occurs at any time
- A hypothetical strategy will be used for any subject who has their Week 52 assessment scheduled to be on or after the COVID-19 environment onset date, who has not been classified as a Non-Responder using the strategy above, and has any of the following Intercurrent Events on or after the COVID-19 onset date:
  - Study Withdrawal (includes Lost to Follow Up)
  - Treatment Failure (includes consideration of corticosteroids and immunosuppressants)
  - Missing SLEDAI-2K score (IBA)

The response status for these subjects will be treated as a missing value and will be assumed to be Missing At Random (MAR). It will be imputed using Multiple Imputation methods, which take into account the subjects baseline characteristics and their existing pre-COVID-19 data.

 Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint.

#### **Imputation of Missing Data**

- A bayesian repeated measures logistic regression model will be fitted to the observed data, using a Markov Chain Monte Carlo (MCMC) approach, adjusting for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10 ), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day). Non-informative priors will be used.
- Samples will be drawn from the posterior distribution of the model parameters of the Bernoulli
  distribution for each treatment group and each missingness pattern.
- Each sample leads to a separate imputed dataset, in which the missing values are replaced by
  values drawn randomly from their conditional distribution. This distribution is based on the
  observed data and the covariates for that subject using the imputation model and the sampled
  parameter values.
- These steps will be repeated at least 1000 times.

# **Model Specification**

- Each imputed dataset will be analyzed using logistic regression to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10 ), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day).
- The resulting Odds Ratios and their Standard Errors will be combined across imputations using Rubin's rules.

#### 7.1.7.2. COVID Environment – Observed Data Until the COVID-19 Pandemic

The second additional analysis assumes that all data after the COVID-19 environment onset date may either be missing due to the pandemic or affected by the pandemic. There may be intangible ways that

the data may have been affected even if it has been collected, therefore this analysis accepts that we cannot distinguish between affected and unaffected data after the COVID-19 environment onset date.

A Hypothetical estimand will be used to estimate the treatment effect had the COVID-19 pandemic not occurred. The difference in response rates between Arm A and Arm B at Week 52 will be assessed for subjects who:

- achieve a SLEDAI 2K-score ≤2 (IBA),
- without immunosuppressants and
- with corticosteroids at a prednisone equivalent dose of ≤5mg/day and
- in the absence of any Intercurrent Events that could be attributable to the COVID-19 pandemic, based on the COVID-19 environment onset date.

The full MITT population will be used, with the following attributes:

- A strategy that matches the primary analysis (Hybrid) will be used for the following Intercurrent Events to classify the subject as a Non-Responder:
  - Study Withdrawal (includes Lost to Follow Up and death) that occurs prior to the onset date
  - Treatment Failure (includes consideration of corticosteroids and immunosuppressants) that occurs prior to the onset date

0

- A hypothetical strategy using the COVID-19 environment onset date as the Intercurrent Event
  will be used for any subject who has their Week 52 assessment scheduled to be on or after the
  COVID-19 environment onset date, who has not already been classified as a Non-Responder
  using the strategy above. The response status for these subjects will be treated as a missing
  value and will be assumed to be Missing At Random (MAR). It will be imputed using Multiple
  Imputation methods, which take into account the subjects baseline characteristics and their
  existing pre-COVID data.
- Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint.

The statistical methods will match the first additional analysis (Section 7.1.7.1) [T12.41].

# 7.1.7.3. Pre-COVID – MITT Population Prior to the COVID-19 Pandemic

The third additional analysis will use the "MITT Week 52 prior to COVID-19" analysis population. This will assess the treatment difference on the subset of subjects who completed Week 52 before the COVID-19 environment onset date and hence have no possible COVID-19 impact on any of their assessments.

A Hybrid estimand will be used to estimate the treatment effect in the population of subjects for which the COVID-19 pandemic not occurred. The difference in response rates between Arm A and Arm B at Week 52 will be assessed for subjects who complete Week 52 prior to the COVID-19 environment onset date and who:

- achieve a SLEDAI 2K-score ≤2 (IBA),
- without immunosuppressants and
- with corticosteroids at a prednisone equivalent dose of ≤5mg/day.

The "MITT Week 52 prior to COVID-19" population will be used, with the following attributes:

- A strategy that matches the primary analysis (Hybrid) will be used for the following Intercurrent Events to classify the subject as a Non-Responder:
  - Study Withdrawal (includes Lost to Follow Up and Death)
  - o Treatment Failure (includes consideration of corticosteroids and immunosuppressants)
- Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint.

The statistical methods will match the primary analysis (Section 7.1.5) for the endpoint definition, derivation, model specification, model checking and diagnostics and the model results presentation [T12.42].

# 7.1.7.4. Graphical Representation of the Additional Analyses

Table 3 shows a graphical representation of specific scenarios for individual subjects, in terms of their completion status or any Intercurrent Events, and the timing of them in relation to the COVID-19 environment onset date (Section 15.6.16). The way in which the data for subjects in each scenario will be used is presented for the primary analysis, plus each of the three pre-specified additional analyses to investigate the COVID-19 pandemic.

Table 3 Graphical Representation of the Additional Analyses

| COVID-19 e | environment<br>et date | Description | Primary<br>Analysis<br>Hybrid | COVID<br>Attributed | COVID<br>Environment | Pre-<br>COVID |
|---|---|---|---|---|---|---|
| X——0 Comp. | | Subject Completes Week 52 prior to onset date | R/NR | R/NR | R/NR | R/NR |
| X—0 WD/Death | | Subject had scheduled Week 52 prior to COVID-19 environment onset date, but Withdraws / LTFU / Dies prior to COVID-19 environment onset date | NR | NR | NR | NR |
| X0 TF | | Subject had scheduled Week 52 prior to onset date, but has Treatment Failure prior to onset date | NR | NR | NR | NR |
| X | 0 Comp. | Subject Completes on or after COVID-19 environment onset date | R/NR | R/NR | Imputed | Excluded |
| X——0<br>WD/Death | | Subject had scheduled Week 52 on or after onset date, but Withdraws/Dies prior to onset date | NR | NR | NR | Excluded |
| X0 | | Subject had scheduled Week 52 on or after onset date, but has Treatment Failure prior to onset date | NR | NR | NR | Excluded |

| X | <del>0</del> WD | Subject Withdraws on or after onset date | NR | Imputed | Imputed | Excluded |
|---|---|---|---|---|---|---|
| Χ | <del>0</del> Death | Subject Dies on or after onset date | NR | NR | Imputed | Excluded |
| X | <del>0</del> TF | Subject has Treatment Failure on or after onset date | NR | Imputed | Imputed | Excluded |

Comp. = Completed; WD = Study Withdrawal (includes Lost to Follow Up); TF = Treatment Failure (includes consideration of corticosteroids and immunosuppressants); R/NR = Responder/Non-Responder based on SLEDAI-2K criteria; NR = Non-Responder

# 7.2. First Major Secondary Efficacy Analyses

# 7.2.1. Endpoint / Variables

The proportion of participants with a state of clinical remission defined as a Clinical SLEDAI-2K score =0 (IBA) (Section 15.6.3), achieved without immunosuppressants and corticosteroids at a prednisone equivalent dose of 0 mg/day at Week 64.

The protocol Section 10.4.1 Efficacy analysis then clarifies that:

For participants who discontinue prematurely from study treatment and for who subsequent collection of data is not possible, it will be assumed for the primary analysis that they are treatment failures. A dropout/treatment failure = non-responder (DO/TF=NR) analysis will be used.

Hence when adopting the ICH Estimands and Sensitivity Analysis in Clinical Trials E9 R1 addendum terminology, this endpoint is defined as:

#### **Clinical Remission**

#### Responder:

- Clinical SLEDAI-2K score =0 (IBA); and
- 7-day average prednisone equivalent dose of 0mg/kg at the visit; and
- Not a TF at the current or any prior visit (TF includes consideration of corticosteroids and immunosuppressants); and
- Did not Withdraw from the study prior to the visit

#### Non-Responder:

- Clinical SLEDAI-2K score >0 (IBA); or
- 7-day average prednisone equivalent dose > 0mg/kg at the visit; or
- TF at the current or any prior visit (TF includes consideration of corticosteroids and immunosuppressants); or
- Withdrew from the study prior to the visit (includes lost to follow-up and death)

The derivation of Clinical SLEDAI-2K score is provided in Section 15.6.3.

Treatment failures are defined in Section 15.6.15. and includes the use of re–start belimumab for Arms A&B. Re-start belimumab is principal investigator prescribed belimumab, it does not include late dosing of Year 1 (prescribed pre Week 52) belimumab injections that were taken incorrectly after Week 52.

Withdrawal from the study prior to Week 64 is defined in Section 5.9.

Note: Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint, subjects who discontinue investigational product will only be non-responders if they also meet 1 of the criteria above.

Note this clarification of notation does not change the protocol-specified analysis.

The analysis of Arm A vs Arm B will use data from treatment Arms A, and B only. An exploratory analysis of the relative performance of Arm B vs. Arm C will also be conducted, using data from Arms B and C only.

Note: A subject can be a responder for this key secondary endpoint without being a responder for the primary endpoint.

# 7.2.2. Summary Measure

The odds ratio at Week 64 between Arm B (Combination) vs Arm A (Control).

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent event strategies used for the primary endpoint (as defined in Section 7.1.4) will be used for this major secondary endpoint.

Subjects in Arms A and B will not receive investigational product post Week 52, these subjects will be considered as on treatment if they completed treatment through Week 52.

The main estimand of this endpoint, is a Hybrid strategy, subjects who discontinue investigational product will continue in the study, assessments after treatment discontinuation will be included in the main estimand.

# 7.2.5. Statistical Analyses / Methods

#### 7.2.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

 The proportion of participants with a state of clinical remission defined as a Clinical SLEDAI-2K score = 0 (IBA), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day at Week 64, and without treatment failure or study withdrawal

#### **Model Specification**

• The proposed statistical analyses planned for the primary endpoint will be repeated for this major secondary endpoint.

#### **Model Checking & Diagnostics**

 The model and diagnostics checks proposed for the primary endpoint will be repeated for this major secondary endpoint.

#### **Model Results Presentation**

 The proposed tables and figure for the primary endpoint will be repeated for this major secondary endpoint [T22.01, T22.02, F22.01].

#### **Subgroup Analyses**

Subgroup analyses will not be conducted for major secondary endpoints.

#### **Supportive Analyses**

- The disposition of the endpoint, detailing the reasons why a subject was a non-responder will be summarized (n,%) [T22.03].
- The components of the endpoint will be summarized [T22.04]. i.e. proportion of participants with
  - Clinical SLEDAI-2K score =0 (IBA)
  - Treatment failure due to corticosteroid use
  - Corticosteroids at a prednisone equivalent dose of >0mg/day and <=5mg/day</li>
  - Treatment failure due to immunosuppressant use
  - Treatment failure due to anti-malarial, NSAID, Aspirin or other prohibited medication use
  - Study withdrawal
- The table will include:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group,
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the stratified (baseline SLEDAI-2K score, baseline immunosuppressant use, baseline corticosteroid dose) Cochran-Mantel-Haenszel treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A
- This key Secondary efficacy analysis at Week 64 will be repeated to assess the robustness of the results:
  - Including subjects where the independent blinded assessor was potentially unblinded, at Week 64 (i.e. ITT population). Intercurrent event strategy: Hybrid [T22.05].
  - Unadjusted for covariates. The only independent variable in the model will be treatment group. Intercurrent event strategy: Hybrid [T22.06].

Tipping point analyses may be performed, including all recorded data up to the time of study withdrawal, and using differing assumptions regarding data missing following withdrawal from the study as detailed in Section 7.1.6. Intercurrent event strategy: Hybrid [T22.07, F22.12].

# 7.2.6. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the First Major Secondary Endpoint

Additional analyses will be carried out to assess the impact of the COVID-19 pandemic on the first major secondary endpoint.

# 7.2.6.1. COVID Attributed – Observed data until Intercurrent Events that could be attributable to the COVID-19 pandemic

The first additional analysis specified for the primary endpoint (Section 7.1.7.1) will be repeated for the first major secondary endpoint [T22.35].

#### 7.2.6.2. COVID Environment – Observed data until the COVID-19 pandemic

The second additional analysis specified for the primary endpoint (Section 7.1.7.2) will be repeated for the first major secondary endpoint [T22.36].

#### 7.2.6.3. Pre-COVID – MITT Population prior to the COVID-19 pandemic

The third additional analysis specified for the primary endpoint (Section 7.1.7.3) will be repeated for the first major secondary endpoint [T22.37] using the "MITT Week 64 prior to COVID-19" population.

# 7.3. Second Major Secondary Efficacy Analyses

#### 7.3.1. Endpoint / Variables

The proportion of participants with a state of disease control defined as a SLEDAI-2K score  $\leq 2$  (IBA), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of  $\leq 5$ mg/day at Week 104.

This endpoint is as defined for the primary endpoint (Section 7.1) but at Week 104.

The primary comparison is Arm B (Combination) vs Arm A (Control), and an exploratory summary of Arm B (Combination) vs Arm C (Reference) will also be shown.

Note: A subject can be a responder for this key secondary endpoint without being a responder for the primary endpoint or the first major secondary endpoint.

#### 7.3.2. Summary Measure

The odds ratio at Week 104 between Arm B (combination) vs Arm A (control).

# 7.3.3. Population of Interest

The secondary efficacy analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

### 7.3.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent event strategies used for the primary endpoint (see as defined in Section 7.1.4) will be used for this major secondary endpoint.

Subjects in Arms A and B will not receive investigational product post Week 51, these subjects will be considered as on treatment if they completed treatment through Week 52.

The main estimand of this endpoint, is a Hybrid strategy, subjects who discontinue investigational product will continue in the study, assessments after treatment discontinuation will be included in the main estimand.

# 7.3.5. Statistical Analyses / Methods

# 7.3.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

The proportion of participants with a state of disease control defined as a SLEDAI-2K score
 ≤2 (IBA), without treatment failure or study withdrawal

#### **Model Specification**

• The proposed statistical analyses planned for the primary endpoint will be repeated for this major secondary endpoint.

#### **Model Checking & Diagnostics**

• The model and diagnostics checks proposed for the primary endpoint will be repeated for this major secondary endpoint.

#### Model Results Presentation

 The proposed tables and figure for the primary endpoint will be repeated for this major secondary endpoint [T22.10, T22.11, F22.04].

# **Subgroup Analyses**

Subgroup analyses will not be conducted for major secondary endpoints.

#### **Supportive Analyses**

• The disposition of the endpoint, detailing the reasons why a subject was a non-responder will be summarized (n,%) [T22.12].

The components of the endpoint will be summarized [T22.13]. i.e. proportion of participants with:

- SLEDAI-2K score <=2 (IBA)</li>
- Treatment failure due to corticosteroid use
- Treatment failure due to immunosuppressant use

- Treatment failure due to anti-malarial, NSAID, Aspirin or other prohibited medication use
- Study withdrawal
- The table will include:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group,
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the stratified (baseline SLEDAI-2K score, baseline immunosuppressant use, baseline corticosteroid dose) Cochran-Mantel-Haenszel treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A
- This key Secondary efficacy analysis at Week 104 will be repeated to assess the robustness of the results:
  - Including subjects where the independent blinded assessor was potentially unblinded, at Week 104 (i.e. ITT population). Intercurrent event strategy: Hybrid [T22.14].
  - Unadjusted for covariates. The only independent variable in the model will be treatment group. Intercurrent event strategy: Hybrid [T22.15].

Tipping point analyses may be performed, including all recorded data up to the time of study withdrawal, and using differing assumptions regarding data missing following withdrawal from the study, as detailed in Section 7.1.6. Intercurrent event strategy: Hybrid [T22.16, F22.13].

# 7.3.6. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the Second Major Secondary Endpoint

Additional analyses will be carried out to assess the impact of the COVID-19 pandemic on the second major secondary endpoint. It may not be possible to conduct all the proposed analysis, the feasibility of the analysis is dependent on the number of observed intercurrent events after the COVID-19 environment onset date or quantity of missed assessments.

# 7.3.6.1. COVID Attributed – Observed Data Until Intercurrent Events That Could be Attributable to the COVID-19 Pandemic

The first additional analysis specified for the primary endpoint (Section 7.1.7.1) will be repeated for the second major secondary endpoint [T22.38].

# 7.3.6.2. COVID Modified – SLEDAI 2K-Score ≤2 (IBA), Without Current Immunosuppressants, Without Current Belimumab (arms A&B), and prednisone equivalent dose of ≤5mg/day at Week 104

This is an additional endpoint to that specified in the protocol, using a modified definition of disease control. It will be defined as a SLEDAI-2K score  $\leq 2$  (IBA), without **Current** Immunosuppressants

or **Current** Belimumab dosing (Arms A and B) and corticosteroids at a prednisone equivalent dose of ≤5mg/day at Week 104.

It is possible that subjects may take extra immunosuppressants/corticosteroids/Belimumab during the COVID-19 environment, which would class them as a Treatment Failure and therefore a Non-Responder for the main analysis. This additional analysis will allow the subjects to take these concomitant medications / re-start Belimumab during the study, as long as their dose is back to the pre-defined levels for an adequate period prior to Week 104. Therefore, these subjects will not automatically be classed as a Treatment Failure (Non-Responder) for this additional analysis.

#### Disease Control without Treatment Failure

#### Responder:

- SLEDAI 2K-score ≤2 (IBA); and
- Did not withdraw from the study prior to the visit; and
- Did not receive a protocol non-allowed immunosuppressant or change in immunosuppressant on the day of the visit or the 55 days prior; and
- Did not receive corticosteroids at a prednisone equivalent dose of >5mg/day (7day average) on the day of the visit or the 6 days prior; and
- Did not have a Belimumab dose on the day of the visit or the 112 days (16 weeks) prior (Arms A and B).

#### Non-Responder:

- SLEDAI 2K-score >2 (IBA); or
- Withdrew from the study prior to Week 104 (which includes study withdrawal, lost to follow-up and death); or
- Received a protocol non-allowed immunosuppressant or change in immunosuppressant on the day of the visit or the 55 days prior; or
- Received corticosteroids at a prednisone equivalent dose of >5mg/day (7day average) on the day of the visit or the 6 days prior; or
- Had a Belimumab dose on the day of the visit or the 112 days (16 weeks) prior (Arms A and B).

The derivation of SLEDAI-2K score is provided in Section 15.6.3 and withdrew from the study prior to Week 104 in Section 5.9.

Note: Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint, subjects who discontinue investigational product will only be non-responders if they also meet one of the criteria above.

The statistical methods will match the primary analysis (Section 7.1.5 Hybrid strategy) for the model specification, model checking and diagnostics and the model results presentation at Week 104 [T22.39].

# 7.4. Lupus Low Disease Activity State (LLDAS)

# 7.4.1. Endpoint / Variables

The LLDAS endpoint is derived based on [Franklyn, 2016] and [Oon, 2019] given the available data in this study, namely:

- SLEDAI-2K ≤4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity;
- o no new features of lupus disease activity compared with the previous assessment;
- o PGA (scale 0-3)  $\leq 1$ ;
- o current prednisolone (or equivalent) dose ≤7.5 mg daily; and
- o well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents, excluding investigational drugs.
- Not study withdrawal (including death and lost to follow-up)

Further details of the derivation that is applied to this study is provided in Section 15.6.9 Lupus Low Disease Activity State (LLDAS). The principal investigators assessment of the SLEDAI-2K is used in the derivation of LLDAS. Treatment Failures (TF) is not a component of the endpoint.

# 7.4.2. Summary Measure

The odds ratio between Arm B (Combination) vs Arm A (Control).

#### 7.4.3. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

#### 7.4.4. Strategy for Intercurrent (Post-Randomization) Events

The definition of the endpoint includes consideration for the intercurrent events of study withdrawal (including LTFU and death)(as defined in Section 7.1.4). Treatment failure is not a component of the endpoint and is not considered as an intercurrent event. Data from subjects who discontinue IP is included in this secondary endpoint.

Subjects in Arms A and B will not receive investigational product post Week 52, these subjects will be considered as on treatment if they completed treatment through Week 52.

Subjects who discontinue investigational product will continue in the study, assessments after treatment discontinuation will be included in the estimand.

# 7.4.5. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

# 7.4.6. Statistical Methodology Specification

# **Endpoint / Variables**

- Proportion of participants that meet the Lupus Low Disease Activity State (LLDAS) response criteria by Visit [T12.37, T22.31]
- Proportion of participants for each component of the Lupus Low Disease Activity State (LLDAS) response criteria at Weeks 52, 64, and 104 [T12.38,T22.32]

# **Model Specification**

 The proposed statistical analyses planned for the primary endpoint will be repeated for LLDAS.

#### **Model Checking & Diagnostics**

 The model and diagnostics checks proposed for the primary endpoint will be repeated for the LLDAS endpoints.

#### **Model Results Presentation**

- The table will display:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

# 7.5. Other Secondary Efficacy Analyses - Proportion Endpoints (Hybrid)

# 7.5.1. Summary Measure

The odds ratio between Arm B (combination) vs Arm A (control).

#### 7.5.2. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

# 7.5.3. Strategy for Intercurrent (Post-Randomization) Events

The same intercurrent event strategy as used for the primary endpoint (Section 7.1.4) will also be used for other secondary endpoints.

# 7.5.4. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

# 7.5.5. Statistical Methodology Specification

# **Endpoint / Variables**

- The proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (IBA), achieved without treatment failure or study withdrawal by visit (T12.27, T22.17, F12.05, F22.05).
- Proportion of participants with a state of clinical remission, defined as a Clinical SLEDAI-2K score = 0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit. (T22.08, F22.02)
- Proportion of participants with a state of complete remission, defined as SLEDAI-2K score = 0 (PI), achieved without treatment failure or study withdrawal, and with corticosteroids at a prednisone equivalent dose of 0 mg/day, sustained for at least 24 weeks.(T22.19)
- Proportion of participants with a state of clinical remission, defined as Clinical SLEDAI-2K score =0 (PI) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, sustained for at least 24 weeks. (T22.20)
- Proportion of participants with a state of complete remission, defined as a SLEDAI-2K score =0 (PI), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit (T22.21,F22.08)
- The proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (PI), achieved without treatment failure or study and with corticosteroids at a prednisone equivalent dose of ≤5mg/day by visit (T12.28, T22.18, F12.06).
- The proportion of participants with a state of clinical remission defined as a Clinical SLEDAI-2K score =0 (PI) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit (T22.18,F22.03).

#### **Model Specification**

• The proposed statistical analyses planned for the primary endpoint (Hybrid) will be repeated for the other binary secondary endpoints.

#### **Model Checking & Diagnostics**

• The model and diagnostics checks proposed for the primary endpoint will be repeated for the other binary secondary endpoints.

#### **Model Results Presentation**

For each endpoint a table will display:

- the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group
- the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
- the p-value for the odds ratio the treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

# 7.6. Other Secondary Efficacy Analyses - Proportion Endpoints (Observed Case)

# 7.6.1. Summary Measure

The odds ratio between Arm B (combination) vs Arm A (control).

# 7.6.2. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

# 7.6.3. Strategy for Intercurrent (Post-Randomization) Events

Treatment failure and study withdrawal will not be considered as components of the endpoint and an observed case analysis will be conducted.

# 7.6.4. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

# 7.6.5. Statistical Methodology Specification

#### **Endpoint / Variables**

- Proportion of participants with SLEDAI-2K (PI) organ improvement by visit (T12.31, T22.27)
- Proportion of participants with SLEDAI-2K (PI) organ worsening by visit (T12.32,T22.28)
- Proportion of participants with any SLICC Damage Index worsening (change >0) compared with baseline at Week 52 and Week 104 (Worst Observation Carried Forward for observed visits) (T12.36, T22.30). Note: The scoring of the SLICC Damage Index is such that it should not be possible for a subject to improve. Hence the WOCF is used to ensure the correct scoring has been applied the highest score for an individual item is carried forward to subsequent observed visits, it does not impute missing visits. Only observed (but potentially corrected by WOCF) data will be analysed, irrespective of treatment failure or IP discontinuation (all data reported will be included).

# **Model Specification**

The proposed statistical analyses planned for the primary endpoint will be repeated for the
other binary secondary endpoints. The SLICC Damage Index worsening will also include
SLICC DAMAGE index score at baseline as a covariate.

# **Model Checking & Diagnostics**

 The model and diagnostics checks proposed for the primary endpoint will be repeated for the other binary secondary endpoints.

#### **Model Results Presentation**

- For each endpoint a table will display:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group
- For the SLICC analysis (T12.36, T22.30) the table will also display:
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A at weeks 52, 64 and 104.

# 7.7. Other Secondary Efficacy Analyses - Time to Event Endpoints

# 7.7.1. Summary Measures

The hazard ratio of Arm B (combination) and Arm A (control).

# 7.7.2. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

#### 7.7.3. Strategy for Intercurrent (Post-Randomization) Events

Subjects without an event will be considered censored at the last observed timepoint.

# 7.7.4. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

# 7.7.5. Statistical Methodology Specification for Time to Event Endpoints

#### **Endpoints**

• Time to first severe flare (as measured by the modified SLE Flare Index) [T12.33, T22.22, F12.12,F22.06]

- Time to first flare (as measured by the modified SLE Flare Index) [T12.34, T22.23,F12.09,F22.07]
- Time to disease control sustained to Week 104, defined as SLEDAI-2K score ≤2 (PI), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of ≤5 mg/day.[T22.24,F22.09].
- Time to clinical remission sustained to Week 104, defined as Clinical SLEDAI-2K score=0
  (PI) (Section 15.6.3), achieved without immunosuppressants and with corticosteroids at a
  prednisone equivalent dose of 0 mg/day [T22.33].

#### Derivation

#### Flare Endpoints

| Subject | Time to defined as: | Censored |
|---|---|---|
| Flare | Date of 1st flare – trt start date +1 | No = 0 |
| TF before or without flare | Date of 1st TF – trt start date +1 | No = 0 |
| Subjects without a Flare or TF | Subjects without a Flare or TF who have an intercurrent event: | |
| Withdraw | Date of last Flare assessment prior to | Yes =1 |
| Lost to Follow-up | intercurrent event – trt start date +1 | |
| Die | Date of Death – trt start date +1 | Yes =1 |
| For Year 1 reporting: | | |
| Subject completes Week 52 | Date of Week 52 visit – trt start date +1 | Yes =1 |
| For Year 2 reporting: | | |
| Subject completes Week 104 | Date of Week 104 visit – trt start date +1 | Yes =1 |

- The flare criteria will be programmed from the SLEDAI-2K irrespective of data recorded on the SFI form
- Flares recorded as severe on the SFI form will be downgraded to not severe in the programmed endpoint if the only cause of the severe flare was SLEDAI-2K>12
- Only post baseline flares will be included in the analysis (Flares on Day 1 will not be considered)
- Treatment failure is considered as a severe flare.
- Subjects who do not have a flare assessment post baseline will be censored at Day 1 and hence reported as 'time to' defined as 1 and censor =Yes = 1

#### **Time to Response Endpoints**

| Subject | Time to defined as: | Censored |
|---|---|---|
| Sustained response | Date of 1st sustained response – trt start date +1 | No = 0 |
| Subjects without a sustained response | | |

| Withdraw | Date of last visit prior to intercurrent event – trt | Yes =1 |
|---|---|---|
| Lost to Follow-up | start date +1 | |
| Treatment Failure | | |
| Die | Date of Death – trt start date +1 | Yes =1 |
| For Year 1 reporting: | | |
| Subject completes Week 52 without treatment failure | Date of Week 52 visit – trt start date +1 | Yes =1 |
| For Year 2 reporting: | | |
| Subject completes Week 104 without treatment failure | Date of Week 104 visit – trt start date +1 | Yes =1 |

Further detail is provided in Section 15.6.7.

#### **Model Specification**

A Cox proportional hazards model controlling for treatment group, baseline SLEDAI-2K score ( $\leq$ 9 vs.  $\geq$ 10 ), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent  $\leq$ 10 mg/day vs. >10 mg/day) will be used to evaluate time to event endpoints.

Ties will be managed using Efron's approximation.

#### **Model Checking & Diagnostics**

Overall model Goodness of fit tests using the -2 Log Likelihood, Akaike's Information Criterion (AIC), and Schwarz Bayesian criterion (SBC) tests will be performed. The AIC and SBC statistics offer two different ways of adjusting the -2 log likelihood statistic for the number of terms in the model and the number of observations used. Lower values in these statistics represent a more desirable model. These tests will aid in the assessment of model fit but the final decision regarding goodness of fit will be based on statistician review. If the model fit is considered inadequate additional analysis will be conducted.

#### **Model Results Presentation**

A table for each endpoint [as above] will present:

- The number and percentage of subjects with an event and the median, 25<sup>th</sup> percentile, and 75<sup>th</sup> percentile of days to event by treatment group,
- the hazard ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C.
- the p-value for the hazard ratio for Arm B vs Arm A.
- the median, 25<sup>th</sup> percentile, and 75<sup>th</sup> percentile of days, min and max for the study day of 1<sup>st</sup> event

A Kaplan-Meier plot of time to event for each endpoint will be displayed by treatment group.

#### **Subgroup Analyses**

Subgroup analyses will not be conducted for secondary endpoints.

# 7.8. Other Secondary Efficacy Analyses - Duration Endpoints

# 7.8.1. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

# 7.8.2. Strategy for Intercurrent (Post-Randomization) Events

A Hybrid strategy will be adopted

# 7.8.3. Endpoint / Variables

The endpoint points are defined as per the primary (Section 7.1) and secondary (Section 7.2) endpoints. The duration is defined as the longest period between any 2 assessments that the subject remains a responder throughout (missing assessments are not considered).

# 7.8.4. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

# 7.8.5. Statistical Methodology Specification for Duration Endpoints

# **Endpoints**

- Duration of disease control, defined as SLEDAI-2K score ≤2 (PI), achieved without treatment failure or study withdrawal [T12.29].
- Duration of clinical remission, defined as Clinical SLEDAI-2K score =0 (PI) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day. [T22.25].

#### **Imputation of Missing Data**

**Duration endpoints:** 

There will be no imputation of missing data, only observed data will be considered. Duration will be derived based on the date of the assessment as:

Date of last visit meeting criteria - Date of first visit meeting criteria +1

#### **Model Specification**

 Duration endpoints will be analyzed using ANCOVA to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day).

#### **Model Checking & Diagnostics**

The Kolmogorov-Smirnov D statistic will be used to test the assumption of normality.
 Residuals will be reviewed to assess the homogeneity of variance assumption. If the model fit is inadequate additional analysis will be conducted.
### **Model Results Presentation**

The tables will display:

- Baseline: the number of subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, maximum for each arm
- At each visit:
  - the number subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum,
  - LS Mean, and standard error of the LS Mean for each arm at Weeks 52, 64 and 104.
  - o the treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
  - the p-value for treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

## 7.9. Other Secondary Efficacy Analyses Continuous Endpoints

## 7.9.1. Endpoint / Variables

Change from baseline in SLEDAI-2K (PI) score and change from baseline in Physician Global Assessment (PGA) by visit.

## 7.9.2. Summary Measure

The difference in mean change from baseline between Arm B (Combination) vs Arm A (Control).

## 7.9.3. Population of Interest

The secondary efficacy analyses will be based on the modified Intent-To-Treat population, unless otherwise specified.

## 7.9.4. Strategy for Intercurrent (Post-Randomization) Events

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subjects not withdrawn from the study . Data collected after TF will be used in the analysis.

#### 7.9.5. Subgroup, Supportive and Sensitivity Analyses

There are no planned subgroup, supportive or sensitivity analyses for other secondary endpoints.

## 7.9.6. Statistical Methodology Specification for Continuous Endpoints

## **Endpoints**

- Change from baseline in SLEDAI-2K (PI) score by visit.[T12.30, T22.26,F12.07, F22.10].
- Change from baseline in Physician Global Assessment (PGA) by visit [T12.35,T22.29, F12.08, F22.11].

## Imputation of Data for Missed Visits and Following Study Withdrawal

- A bayesian repeated measures normal model will be fitted to the data collected prior to study withdrawal, using a Markov Chain Monte Carlo approach, adjusting for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day). Non-informative priors will be used.
- Quasi-independent samples will be drawn from the posterior distributions for the parameters
  of the multivariate normal distribution for each treatment group and each missingness
  pattern.
- Each sample leads to a separate imputed dataset, in which the missing values are replaced by values drawn randomly from their conditional distribution. This distribution is based on the observed data and the covariates for that subject using the imputation model and the sampled parameter values.
- These steps will be repeated at least 1000 times.

## **Imputation of Data Following Partially Missing SLEDAI-2K**

The same imputation approach will be used for subjects with partially completed SLEDAI-2K scores (i.e. some missing items) however imputed values that are below the minimum possible score (determined from the completed items) will be replaced with the known minimum score. Similarly, imputed values that are above the maximum possible score will be replaced with the known maximum score

Minimum and maximum possible SLEDAI-2K scores are detailed in Section 15.6.3.

## **Model Specification**

- Each imputed dataset will be analyzed using ANCOVA to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day).
- The resulting treatment differences and their SEs will be combined across imputations using Rubin's rules.
- The models for the SLEDAI-2K endpoints will include the baseline (PI) SLEDAI-2K score (continuous) rather that the stratification factor (≤9 vs. ≥10).
- The model for PGA endpoints will also include the baseline PGA score (continuous).

#### **Model Checking & Diagnostics**

The Kolmogorov-Smirnov D statistic will be used to test the assumption of normality. Residuals will be reviewed to assess the homogeneity of variance assumption. If the model fit is inadequate additional analysis will be conducted

### **Model Results Presentation**

The tables will display:

- Baseline: the number of subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, maximum for each arm
- At each visit:
  - the number subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum
  - LS Mean, and standard error of the LS Mean for each arm at Weeks 52, 64 and 104.
  - o the treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
  - the p-value for treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

For change from baseline endpoints, a plot of LS means +/- SE by visit and treatment group will be provided.

# 7.10. Other Secondary Efficacy Analyses: SLEDAI-2K Score ≤2 (IBA), Without Current Immunosuppressant and Corticosteroids <=5mg/day

## 7.10.1. Endpoint / Variables

This is an additional endpoint to that specified in the protocol. The proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (IBA), achieved without current immunosuppressants and with current corticosteroids at a prednisone equivalent dose of ≤5mg/day at Week 52. Immunosuppressant use and corticosteroid reduction are key components of the endpoint in the protocol and are included in the synopsis definition without referring to treatment failure. Hence a supportive analysis that considers immunosuppressant use and corticosteroids without other treatment failure criteria will be conducted.

## Disease Control without Treatment Failure

#### Responder:

- SLEDAI-2K score ≤2 (IBA); and
- Did not withdraw (including LTFU and death) from the study prior to the visit; and
- Did not receive a protocol non-allowed immunosuppressant or change in immunosuppressant on the day of the visit or the 55 days prior; and
- Did not receive corticosteroids at a prednisone equivalent dose of >5mg/day (7day average) on the day of the visit or the 6 days prior.

### Non-Responder:

- SLEDAI-2K score >2 (IBA); or
- withdrew from the study prior to Week 52 (including, LTFU and death); or
- Received a protocol non-allowed immunosuppressant or change in immunosuppressant on the day of the visit or the 55 days prior; or

Received corticosteroids at a prednisone equivalent dose of >5mg/day (7day average) on the day of the visit or the 6 days prior.

The derivation of SLEDAI-2K score is provided in Section 15.6.3 and withdrawal from the study prior to Week 52 in Section 5.9.

Note: Discontinuation of study investigational product (belimumab or rituximab) is NOT a component of this endpoint, subject who discontinue investigational product will only be non-responders if they also meet 1 of the criteria above.

## 7.10.2. Summary Measure

The odds ratio at Week 52 between Arm B (Combination) vs Arm A (Control).

## 7.10.3. Population of Interest

The efficacy analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

## 7.10.4. Strategy for Intercurrent (Post-Randomization) Events

The definition of the endpoint includes consideration for the intercurrent events of study withdrawal (including LTFU and death)(as defined in Section 7.1.4). Treatment failure is not a component of the endpoint and is not considered as an intercurrent event. Data from subjects who discontinue IP is included in this secondary endpoint.

## 7.10.5. Statistical Analyses / Methods

### 7.10.5.1. Statistical Methodology Specification

## **Endpoint / Variables**

• The proportion of participants with a state of disease control defined as a SLEDAI-2K score ≤2 (IBA), achieved without study withdrawal, without current immunosuppressants, and with current corticosteroids at a prednisone equivalent dose of ≤5mg/day

#### **Derivation**

Derivation of the endpoint for Arms A, B and C is provided in Section 15.6.4

#### **Model Specification**

- Logistic regression model.
- Terms in the model:
  - **Dependent:** response (yes/no)
  - Categorical: treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day).

## **Model Checking & Diagnostics**

• The model and diagnostics checks proposed for the primary endpoint will be repeated for the other binary secondary endpoints.

## **Model Results Presentation (T12.39)**

- the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group
- the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Week 52.
- the p-value for the odds ratio the treatment difference for Arm B vs Arm A at Week 52.

## 7.11. Additional Efficacy Analyses

A scatter plot will be produced to assess the degree to which the Principal Investigators assessment of SLEDAI-2K differs from that of the Independent Blinded Assessor at Week 52 [F12.10].

This will only include subjects who have both a PI and IBA SLEDAI-2K total score at Week 52. The scatter plot will show the PI SLEDAI-2K total score on the x-axis and IBA SLEDAI-2K total score on the y-axis. No formal statistical testing will be conducted. Different colours (and symbols) will be used for the following groups of subjects:

- Arm A
- Arm B
- Arm C included in MITT population
- Arm C excluded from MITT population

A Bland-Altman plot of the differences between the IBA and PI scores against the mean of the IBA and PI scores will also be produced at Week 52 [F12.11].

If the conclusions of the analysis of the comparison between Arm A and Arm B for disease control differ between SLEDAI-2K score based on the IBA assessment and the PI assessment at Week 52, then additional analysis may be performed. Additional analysis of endpoints at Week 52 will be performed after the Week 52 Statistical Analysis Complete milestone has been met and will be presented in the Week 52 clinical study report. Analysis of endpoints post Week 52 will be performed as part of the Week 104 reporting.

A difference in conclusion will be determined by the study team after reviewing the complete Week 52 SAC outputs. Consideration will be given to the comparison of the magnitude of the odds ratio in the analysis of:

- The proportion of participants with a state of disease control (IBA)
- The proportion of participants with a state of disease control (PI)

with consideration to the related C.I.s and p-values for the comparison between Arms A and B.

The additional analyses will consider some or all of the following endpoints depending on the results by endpoint for the Week 52 reporting:

- Proportion of participants with a state of clinical remission, defined as a Clinical SLEDAI-2K score =0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit.
- Proportion of participants with a state of complete remission, defined as SLEDAI-2K score=0 (IBA), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, sustained for at least 24 weeks
- Proportion of participants with a state of clinical remission, defined as Clinical SLEDAI-2K score =0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, sustained for at least 24 weeks.
- Proportion of participants with a state of complete remission, defined as a SLEDAI-2K score =0 (IBA), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day, by visit
- Proportion of participants with SLEDAI-2K (IBA) organ improvement by visit (TP, Observed)
- Proportion of participants with SLEDAI-2K (IBA) organ worsening by visit (TP, Observed)
- Time to disease control sustained to Week 104, defined as SLEDAI-2K score ≤2 (IBA), achieved without treatment failure or study withdrawal.
- Time to clinical remission sustained to Week 104, defined as Clinical SLEDAI-2K score=0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day.
- Duration of disease control, defined as SLEDAI-2K score ≤2 (IBA), achieved without treatment failure or study withdrawal..
- Duration of clinical remission, defined as Clinical SLEDAI-2K score =0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day.
- Change from baseline in SLEDAI-2K (IBA) score by visit.
- Duration of disease control, defined as SLEDAI-2K score ≤2 (IBA), achieved without treatment failure or study withdrawal.
- Duration of clinical remission, defined as Clinical SLEDAI-2K score =0 (IBA) (Section 15.6.3), achieved without treatment failure or study withdrawal and with corticosteroids at a prednisone equivalent dose of 0 mg/day.
- Change from baseline in SLEDAI-2K (IBA) score by visit.
- Proportion of participants that meet the Lupus Low Disease Activity State (LLDAS) response criteria by Visit based on the IBA assessment.

The analysis will be based on the modified Intent-To-Treat population and use the same intercurrent event strategy (Hybrid as used for the primary endpoint (Section 7.1.4). The analysis will be conducted as specified in Section 7.4.4, Section 7.4.5, Section 7.4.6)

Similarly if there is a difference in the conclusions of the analysis of clinical remission based on the IBA and PI assessment at Week 64, or analysis of disease control based on the IBA and PI assessment at Week 104; then additional analyses will be performed shortly after the Week 104 Statistical Analysis Complete milestone has been met and will be presented in the Week 104 clinical study report. The additional post Week 104 SAC analysis will repeat the analysis of the other secondary endpoints but utilising the IBA assessment instead of the PI assessment. The endpoints to be assessed will potentially include all those previously listed in the Section 7.11.

Note that in the event that the Week 52 reporting does not identify a treatment benefit an abridged set of analysis may be conducted at the end of the study (Week 104).

# 7.12. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic on the Secondary Efficacy Endpoints

There will not be any prospective additional analyses carried out to assess the impact of the COVID-19 pandemic on the secondary (non-major) endpoints. However, if the additional analysis of the primary endpoint indicates a major impact of the COVID-19 pandemic, then additional post-SAC analyses will be performed on the secondary endpoints after the Week 52 Statistical Analysis Complete milestone has been met and will be presented in the Week 52 clinical study report.

Similarly, if the additional analysis of the key secondary endpoints indicates a major impact of the COVID-19 pandemic, then additional post-SAC analyses will be performed on the other secondary endpoints after the Week 104 Statistical Analysis Complete milestone has been met and will be presented in the Week 104 clinical study report.

## 8. SAFETY ANALYSES

The safety analyses will be based on the ITT population. However, if there are more than 5% of subjects who receive a rituximab/placebo infusion that is different from the randomized treatment for one or both doses, safety analysis will be performed on the As Treated population.

## 8.1. Adverse Events

## 8.1.1. Reporting Phases

Adverse events will be reported for Year 1 and Year 2 study period:

#### 8.1.1.1. Pre Treatment

Adverse events starting prior to the 1<sup>st</sup> dose of belimumab.

### 8.1.1.2. On Treatment (Year 1 only)

As defined in Section 5.12

## 8.1.1.3. On Study

As defined in Section 5.11

Year 2 reporting will include all events starting on or after Week 52 visit + 1 day and at or prior to the Week 104 visit.

Year 1&2 reporting will include all events starting on or after the 1<sup>st</sup> dose of belimumab and at or prior to the Week 104 visit.

The tabular summary for each category of AE listed below will include the number of events, number of subjects who reported at least one event, and percentage of subjects who reported at least one AE (incidence) by treatment group for each SOC (where applicable), each PT, and overall.

#### 8.1.1.4. Post Withdrawal/Completion

Adverse events starting after the on study period (Section 5.11 / Section 8.1.1.3) will be reported separately.

## 8.1.2. Adverse Events Analyses

- Adverse events analyses including the analysis of adverse events (AEs), Serious
  Adverse Events (SAEs) and AEs of special interest (AESIs) will be based on GSK
  Core Data Standards
- All subjects will be followed for safety through at least 8 weeks post-treatment.

- A table summarizing AEs that occurred prior to treatment start date will be presented, for each system organ class (SOC) and preferred term (PT) by treatment group [T13.01].
- All AEs will be classified using the current standard GSK Medical Dictionary for Regulatory Activities (i.e. MedDRA version in use at the time of reporting), and grouped by SOC and PT, unless otherwise stated. MedDRA version is detailed on every table that uses MedDRA. The Year 1 report will be based on MedDRA dictionary version 23. The Year 2 report will use the MedDRA dictionary current at the time of reporting the Year 2 data (anticipated to be version 25) and hence will be different to Year 1. Dictionary coding changes between Year 1 and Year 2 will be listed (L23.13) and any impact on the interpretation will be detailed in the Year 2 clinical study report (CSR). The investigator will evaluate all AEs with respect to seriousness, severity, and causality. The severity of an AE is to be determined using the Assessment of Intensity provided in Appendix 7 of the protocol, if a grade is provided for the AE of interest.
- AEs during Year 1 that are not reported until Year 2; and AEs that have their reporting details (e.g. onset date, severity etc) changed after Year 1, will be reported in Year 2 with the latest details. Changes will be listed and summarised as appropriate.
- All treatment-emergent AEs will be summarized for both the double-blind phase (Year 1) and the observational phase (Year 2) separately. Selected tables will also be produced for Years 1 and 2 combined. See Section 8.1.1 for definitions of phases.
- An overall summary of AEs will be presented showing the number and percent of subjects with at least one: AE, related AE, serious AE (SAE), severe AE, AE resulting in study treatment discontinuation, and deaths [On Treatment:T13.02, and On Study: T13.03, T23.01,T23.02, L13.05, L13.06, L23.12].
- Common AEs will be defined as  $\geq 5\%$  incidence in any treatment group.
- The number and percentage of subjects experiencing an AE and the total number of AEs will be summarized for each of the following AE categories:
  - All AEs (by SOC and PT) [On Treatment: T13.04; On Study: T13.05, T23.03, T23.04].
  - AEs (by PT) [On Treatment:T13.06; On Study: T23.05]. (ordered on total incidence Arms A+B+C)
  - Study treatment Related AEs (by SOC and PT) belimumab only [on Treatment:T13.07; on Study: T23.06].
  - Study treatment Related AEs (by SOC and PT) rituximab only [on Treatment:T13.08; on Study: T23.07].
  - Study treatment Related AEs (by SOC and PT) Both belimumab and rituximab [on Treatment: T13.09; on Study: T23.08].
  - Severe AEs (by SOC and PT) [On Treatment:T13.11, on Study T23.27].
  - Serious AEs (by SOC and PT) [On Treatment:T13.21, and on Study:T13.22, T23.19, T23.20]

- AEs leading to permanent discontinuation of study treatment (by SOC and PT) [on Study:T13.26, T13.27; on Study: T23.21, T23.22].
- Deaths (by Category and PT) [on Study: T13.20, T23.18].
- Common Non-Serious AEs (by SOC and PT) [on Study: T13.28; T23.23].
- Study treatment Related Serious AEs (by SOC and PT) [On Treatment:T13.23, T13.24, T13.25; on Study: T23.24, T23.25, T23.26].
- Fatal Serious AEs (by SOC and PT) and Study treatment Related Fatal Serious AEs (by SOC and PT) [On Treatment:T13.29; on Study:T23.28].
- By default, adverse events will be sorted by MedDRA SOCs, in descending order from the SOC with the highest total incidence (i.e., summed across all treatment groups) for any adverse event within the class, to the SOC with the lowest total incidence. If the total incidence for any two or more adverse events is equal, the events will be presented in alphabetical order. Only SOCs with observed AE PTs will be presented. Repeat sort order for MedDRA PTs within each SOC.
- The table for all AEs by SOC and PT will be repeated for the following subgroups:
  - Age group (<65, >=65), [On Treatment: T13.12; On Study: T23.10].
  - Race (Black, non-Black), [On Treatment: T13.13; On Study: T23.11].
  - Country region, [On Treatment: T13.14; On Study: T23.12].
  - Baseline C3/C4 levels & anti-dsDNA subgroup [On Treatment: T13.15; On Study: T23.13].
  - Baseline SLEDAI-2K (<=9, >=10) [On Treatment: T13.16; On Study: T23.14].
  - Baseline Immunosuppressant use (Y,N) )[ On Treatment: T13.17; On Study: T23.15].
  - Baseline Corticosteroid dose (<=10 mg/day, >10 mg/day) )[ On Treatment: T13.18; On Study: T23.16].
  - Gender, [On Treatment: T13.19; On Study: T23.17].
- For Year 1 reporting, the table of deaths by category and PT will include deaths that occurred during Year 1 and fatal SAEs that started during Year 1 and resulted in death during Year 2 by the time of the data cut [On Treatment:T13.20]. For Year 2 reporting, the table of deaths by category and PT will include deaths that occurred during Year 2 (and 8-week Follow-up) that have not been previously reported in Year 1 as a result of a fatal SAE [On Study: T23.22].
- A summary of AEs by SOC, PT and severity will also be provided by treatment group. The number and percentage of subjects will be summarized as mild, moderate or severe based on the maximum severity observed within each PT, and within each SOC [On Treatment: T13.10; On Study: T23.09].
- The hierarchical relationship between MedDRA SOCs, PTs, and verbatim text will be displayed in a listing for all AEs [L13.01, L23.01].
- A listing of all AEs [On Study: L13.02, L23.02], study treatment related AEs [On Study: L13.03, L13.04, L23.03, L23.04], and AEs resulting in study treatment

discontinuation [On Study: L13.05, L13.06, L23.05] and post withdrawal [L13.07,23.06] will be presented, including duration, study day of onset/resolution and days since 1<sup>st</sup> / last belimumab dose.

- If a Year 1 adverse events is reported after year 1 database lock it will be reported in year 2 (L23.07].
- A summary of Adverse Events including Exposure-Adjusted Incidence Rates will be produced for Year 1 On Treatment (Section 5.12) [T13.44] and Years 1&2 combined On Study (Section 5.11) [T23.37]. These will present Adverse Events Overall and by System Organ Class and Preferred Term and will display:
  - the number of subjects experiencing the event (n);
  - For Year 1: the sum of the total time to the first event or total on treatment time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On Treatment Exposure (Year 1);
  - For Years 1&2 combined: the sum of the total time to the first event or total onstudy time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On-Study Exposure (Years 1&2 Combined);
  - the exposure adjusted subject rate per 100 subject years (r = (n/e)\*100).
- A summary of Adverse Events leading to Permanent Discontinuation of Belimumab Study Drug including Exposure-Adjusted Incidence Rates will be produced for Year 1 On Treatment (Section 5.12) [T13.45] and Years 1&2 combined On Study (Section 5.11) [T23.39]. These will present Adverse Events Overall and by System Organ Class and Preferred Term and will display:
  - the number of subjects experiencing the event (n);
  - For Year 1: the sum of the total time to the first event or total on treatment time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On Treatment Exposure (Year 1);
  - For Years 1&2 combined: the sum of the total time to the first event or total onstudy time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On-Study Exposure (Years 1&2 Combined);
  - the exposure adjusted subject rate per 100 subject years (r = (n/e)\*100).

## 8.1.3. Deaths, Serious Adverse Events, and Survival Status

In addition to the tabular summaries of AEs described in Section 8.1.2, listings for all SAEs [L13.08, L23.08], all deaths [L13.09, L23.09] and all non-fatal SAEs [L13.10, L23.10] will be produced (which will also identify on study events). The categorization of the cause of death will be adjudicated by GSK.

A listing of reasons for considering an AE as serious will be provided [L13.11, L23.11].

A summary of Serious Adverse Events including Exposure-Adjusted Incidence Rates will be produced for Year 1 On Treatment (Section 5.12) [T13.46] and Years 1&2 combined

On Study (Section 5.11) [T23.38]. These will present Serious Adverse Events Overall and by System Organ Class and Preferred Term and will display:

- the number of subjects experiencing the event (n);
- For Year 1: the sum of the total time to the first event or total on treatment time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On Treatment Exposure (Year 1);
- For Years 1&2 combined: the sum of the total time to the first event or total onstudy time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On-Study Exposure (Years 1&2 Combined);
- the exposure adjusted subject rate per 100 subject years (r = (n/e)\*100).

A summary of Deaths including Exposure-Adjusted Incidence Rates will be produced for Year 1 On Treatment (Section 5.12) [T13.47] and Years 1&2 combined On Study (Section 5.11) [T23.40]. These will present Deaths Overall and by Category and Preferred Term and will display:

- the number of subjects experiencing the event (n);
- For Year 1: the sum of the total time to the first event or total on treatment time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On Treatment Exposure (Year 1);
- For Years 1&2 combined: the sum of the total time to the first event or total onstudy time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On-Study Exposure (Years 1&2 Combined);
- the exposure adjusted subject rate per 100 subject years (r = (n/e)\*100)

Survival status will also be summarized at Weeks 52 and 104. The number and percentage of subjects will be summarized for each of the following categories for Year 1 and Year 1&2 [T13.30, T23.29].

- Alive
- Consent Withdrawn
- Lost to Follow-up
- All Deaths based on the date of death relative to the planned or actual Week 52 visit.
  - For Year 1 reporting, include deaths that occur at or prior to the observed Week 52 visit.
  - For Year 2 reporting (after the actual Week 52 visit):
    - Include all deaths

## 8.1.4. Adverse Events of Special Interest Analyses

To ensure consistency across belimumab studies, AESI will be defined per the version of the PSAP and MedDRA in effect at the time of DBR.

The Benlysta Program Safety Analysis Plan (PSAP) has been developed to include an adverse event of special interest (AESI) analysis for consistent reporting across belimumab studies. Categorizations for the AESIs are defined in the PSAP.

The milestone defined in the PSAP (i.e. before database release) for adjudications will be "primary analysis database release" (Year 1) and "end of study database release" (Year 2).

Events with a start date on or prior to the week 52 visit date will be attributed to Year 1; otherwise events will be attributed to Year 2. Events will only be reported once even if the event does not resolve by the Week 52 visit.

An overall summary of AESIs will be presented and each specific category of AESI will be presented separately by PT. The number and percentage of subjects with at least one occurrence and the number of events of the following AESIs will be provided [On Treatment: T13.31; On Study: T23.30].

A summary of AESI including Exposure-Adjusted Incidence Rates will be produced for Year 1 On Treatment (Section 5.12) [T13.48] and Years 1&2 combined On Study (Section 5.11) [T23.xxx]. These will present AESI Overall and by each specific category and Preferred Term and will display:

- the number of subjects experiencing the event (n);
- For Year 1: the sum of the total time to the first event or total on treatment time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On Treatment Exposure (Year 1);
- For Years 1&2 combined: the sum of the total time to the first event or total onstudy time\* if no event (years) across all subjects (e), \* defined in Section 15.6.2: On-Study Exposure (Years 1&2 Combined);
- the exposure adjusted subject rate per 100 subject years (r = (n/e)\*100).

The following AESI will be identified and adjudicated as detailed in the PSAP.

### **Adverse Events**

#### Adverse Events of Special Interest (AESI)

AESI will be defined per the version of the PSAP/MedDRA in effect at the time of DBR. Malignant Neoplasms

- Malignancies Excluding non-melanoma skin cancer (NMSC)
- Malignancies Including NMSC
  - Solid Tumour
  - Hematologic

#### **Adverse Events**

## **Adverse Events of Special Interest (AESI)**

- Skin (All)
  - NMSC
  - Excluding NMSC
- Tumours of unspecified malignancy adjudicated as malignant per GSK Post-Injection Systemic Reactions (PISR)
  - PISR per Anaphylactic Reaction Customized MedDRA Query (CMQ) narrow search
  - PISR per Anaphylactic Reaction CMQ broad search
  - PISR per Anaphylactic Reaction CMQ algorithmic search
  - Serious Anaphylaxis per Sampson Criteria per GSK adjudication
  - Serious Acute PISR/Hypersensitivity Per GSK adjudication
    - Serious Acute PISR Excluding Hypersensitivity per GSK adjudication
    - Serious Acute Hypersensitivity Reactions per GSK adjudication
  - Serious Delayed Acute Hypersensitivity Reactions per GSK adjudication
  - Serious Delayed Non-Acute Hypersensitivity Reactions per GSK adjudication

All Infections of Special Interest (Opportunistic Infections (OI), Herpes Zoster (HZ), Tuberculosis (TB), And Sepsis; All and Serious, separately)

- All opportunistic infections (OI) per GSK adjudication
- OI per GSK adjudication excluding Tuberculosis and Herpes Zoster
- Active Tuberculosis
  - Non-Opportunistic
  - Opportunistic
- Herpes Zoster
  - Non-Opportunistic
  - Opportunistic
    - Recurrent
    - Disseminated
- Sepsis

<u>Depression (including mood disorders and anxiety)/suicide/self-injury (All and Serious, separately)</u>

- Depression (including mood disorders and anxiety) (excluding suicide and self-injury)
- Suicide/self-injury
- Serous suicide/self-injury per GSK adjudication
  - Suicidal Behavior
    - Completed Suicide
  - Suicidal Ideation
  - Self-injurious Behavior without Suicidal Intent
- Deaths

Malignant neoplasm events identified as "tumours of unspecified malignancy" will be reviewed for classification as malignant per GSK adjudication and will be presented by category and PT [On Treatment: T13.32; On Study: T23.31].

Post-injection systemic reactions and serious post-injection systemic reactions will be presented using nine different definitions as indicated above. These will be presented by category and PT [On Treatment: T13.33, T13.34; On Study: T23.32, T23.33].

Infection AESIs will be presented by Category and PT for all infections and for infections leading to study treatment discontinuation [On Treatment: T13.41, T13.42; On Study: T23.34, T23.35].

Depression, suicide and self-injury as defined in the PSAP will be presented by Category and PT [On Treatment: T13.43; On Study: T23.36].

All AESI will be presented in a listing [L13.12, L23.12]. Post-Treatment AESIs will be summarized and presented by Category.

## 8.1.5. Post-Injection Systemic Reactions

Summaries of post-injection systemic reactions that occur on the day of an injection or within 3 days after an injection will be presented by treatment group, by the first six injections and over all injections, and PT for the following:

- Post-Injection Systemic Reactions Adverse Events of Special Interest by Category and PT [T13.33, T23.32].
- Serious Post-Injection Systemic Reactions Adverse Events of Special Interest by Category and PT [T13.34, T23.33].
- Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the injection or within 3 days after the Belimumab injection) by PT in the first six injections [On treatment:T13.35].
- Serious Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the injection or within 3 days after the Belimumab injection) by PT in the first six injections [on Treatment: T13.36].
- Serious Acute Post-Injection Systemic Reactions/Hypersensitivity per GSK Adjudication by PT in the First Six Injections [On Treatment: T13.37].
- Serious Delayed Acute Hypersensitivity Reactions per GSK Adjudication by PT in First Six Injections [On Treatment:T13.38].
- Serious Delayed Non-Acute Hypersensitivity Reactions per GSK Adjudication by PT in First Six Injections [On Treatment: T13.39].
- Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the injection or within 3 days after the Rituximab infusion) by PT [On treatment:T13.40].

## 8.1.6. Additional Adverse Event Summaries to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic

Additional adverse event summaries will be produced to further understand the safety profile and/or impact of the COVID-19 pandemic on safety.

Two listings will be produced to show the number of subjects with a suspected, probable or confirmed COVID-19 infection. The first listing will present data for Year 1 On Treatment (Section 5.12) [L13.26]; the second listing will present data for Years 1 and 2 combined On-Study (Section 5.11) [L23.27]. Both listings will also show the number of subjects who had a COVID-19 diagnosis test performed and the number of subjects with positive, negative, or indeterminate results. The listings will be based on information collected on the COVID-19 Coronavirus Infection Assessment CRF page.

Extra tables will be produced to display the incidence of Adverse Events over the time course of the trial. Event rates will be reported by calendar time defined as either pre or during the COVID-19 pandemic (or post the pandemic if applicable by the Year 2 reporting). The COVID-19 environment onset date will be used to define pre and during the COVID-19 pandemic (Section 15.6.16).

The following Tables will summarise the Year 1 On Treatment (Section 5.12) events for pre or during the COVID-19 pandemic. Event rates will be adjusted for on treatment exposure (Section 15.6.2, On -Treatment exposure in the relevant pandemic phase (Year 1)).

- The overall rates of AEs, SAEs and severe AEs [T13.49]
- The overall rates of AEs, SAEs and severe AEs, presented by Country Region (USA/Canada vs. Europe vs. Rest of World) (Section 5.5.2.) [T13.50]
- The most frequent Adverse Events (≥ 5% incidence in any treatment group) by Preferred Term [T13.51]

The following Tables will summarise the Year 1 and 2 combined On-Study (Section 5.11) events for pre or during the COVID-19 pandemic. Note that if a date is defined prior to the Year 2 reporting for the 'end of the pandemic' then this output will split events into pre, during or post the COVID-19 pandemic. Event rates will be adjusted for on-study exposure in the relevant pandemic phase (Section 15.6.2, On-Study exposure (Years 1&2 combined)).

- The overall rates of AEs, SAEs and severe AEs [T23.42]
- The overall rates of AEs, SAEs and severe AEs, presented by Country Region (USA/Canada vs. Europe vs. Rest of World) (Section 5.5.2.) [T23.43]
- The most frequent Adverse Events (≥ 5% incidence in any treatment group) by Preferred Term [T23.44]

## 8.2. Columbia-Suicide Severity Rating Scale (C-SSRS)

For suicidal ideation, the pre-treatment reference period is the lifetime history, current history and baseline (for further detail refer to the IDSL documentation). For suicidal behavior, the pre-treatment reference period is the lifetime history and baseline (note: suicidal behavior is not re-assessed for the current history time period).

Suicidal ideation and suicidal behavior will be considered as distinct categories and assessed independently of each other. Treatment emergence will be assessed for the on treatment period and the on-study period.

Suicidal ideation will be assessed using responses to C-SSRS ideation questions (categories 1 to 5) only. Suicidal behavior will be assessed using responses to C-SSRS behavior questions (categories 6 to 10) only.

- Treatment emergent suicidal ideation will be assessed using the maximum ideation score pre-treatment, compared to the maximum ideation score post-treatment (Year 1 or Year 2 as appropriate). If the maximum ideation score worsens relative to the pre-treatment reference period then this will be considered a treatment emergent suicidal ideation. This is derived from responses to suicidal ideation questions (categories 1 to 5).
- Treatment emergent suicidal behavior will be assessed using the maximum behavior score pre-treatment, compared to the maximum behavior score post-treatment (Year 1 or Year 2 as appropriate). If the maximum behavior score worsens relative to the pre-treatment reference period then this will be considered a treatment emergent suicidal behavior. This is derived from responses to suicidal behavior questions (categories 6 to 10).
- Treatment emergent suicidal ideation or behavior will be defined as a subject having a treatment emergent suicidal ideation (as defined above) and/or a treatment emergent suicidal behavior (as defined above).

## Suicidal Ideation (categories):



## **Suicidal Behavior (categories):**

CCI - This section contained Clinical Outcome
Assessment data collection questionnaires or indices,
which are protected by third party copyright laws and
therefore have been excluded.

A subject must have at least one pre-treatment C-SSRS assessment (screening and/or baseline) and at least one on treatment C-SSRS assessment (post-baseline) to be included in any assessment of treatment emergent.

If a "yes" response is given to any suicidal behavior or a "yes" response is given to suicidal ideation questions 3, 4 or 5 on the C-SSRS, the investigator will be prompted to complete the Possible Suicidality Related Questionnaire (PSRQ).

All C-SSRS tables will be presented for subjects whilst on study.

## 8.2.1. C-SSRS Suicidal Ideation or Behaviour on Study [T13.52, T23.45].

The number and percentage of subjects with each category of suicidal ideation or behavior during treatment (starting after Day 1 assessment) will be presented for Year 1, and Year 2. For suicidal ideation, the maximum ideation score (1-5) at any time during the relevant period will be presented. For suicidal behavior, all behaviors (6-10) present at any time during the relevant period will be presented. This will be regardless of whether the subject had pre-treatment history (up to and including baseline). The categories of suicidal ideation and behavior are presented in increasing order of severity from 1 to 5, and 6-10 respectively.

## 8.2.2. C-SSRS Suicidal Ideation or Behavior Relative to Pre-Treatment [T13.53, T23.46].

The number and percentage of subjects with treatment-emergent suicidal ideation or behavior -post-baseline will be presented for Year 1 and Year 2.

A subject must have at least one pre-treatment C-SSRS assessment (screening and/or baseline) and at least one Year 1 or Year 2 (respectively) C-SSRS assessment to be included in this display.

A subject may have treatment emergent suicidal ideation and/or behavior.

The following categories will be presented:

- The number (%) of subjects with any treatment emergent suicidal ideation (1-5)
  - The number (%) of subjects with any treatment emergent more severe suicidal ideation (4-5)
- The number (%) of subjects with any treatment emergent suicidal behavior (6-10)
- The number (%) of subjects with any treatment emergent suicidal ideation (1-5) or suicidal behavior (6-10)

Note: treatment emergent suicidality can only be assessed in subjects with a pre-treatment maximum ideation score of 4 or lower (as subjects with a pre-treatment ideation score of 5 have no potential to worsen on the 1-5 ideation scale)

## 8.2.3. C-SSRS Shift Changes in Categories from Pre-Treatment to On-Study [T13.54, T23.47].

A summary of the shift from maximum pre-treatment C-SSRS category to maximum category during Year 1 and Year 2 separately will be produced by treatment group.

The pre-treatment period for ideation is based on the lifetime, current and baseline history. For behavior, it is based on the lifetime and baseline history. A subject must have at least one pre-treatment assessment and at least one assessment during Year 1 or Year 2 (respectively) in order to be included in these displays.

The table will display the number and percentage of subjects within the specific shift categories: No suicidal ideation or behavior, suicidal ideation, and suicidal behavior.

Each subject will appear in the table only once. For the purposes of this table only, a subject with both suicidal ideation and suicidal behavior in any period (pre-treatment/on treatment/on-study) will appear in the category of suicidal behavior only.

## 8.2.4. C-SSRS Shift Changes in Categories from Year 1 to Year 2 [T23.48].

A summary of the shift from last Year 1 C-SSRS assessment to maximum Year 2 C-SSRS assessment will be produced by treatment group.

The last Year 1 is based on the current assessment. A subject must have at least one Year 1 assessment, and at least one assessment during Year 2 in order to be included in these displays.

The table will display the number and percentage of subjects within the specific shift categories: No suicidal ideation or behavior, suicidal ideation, and suicidal behavior.

Each subject will appear in the table only once. For the purposes of this table only, a subject with both suicidal ideation and suicidal behavior in any period (pre-treatment/on treatment/on-study) will appear in the category of suicidal behavior only.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards.

For laboratory analyses analytes will be analyzed and summaries and analyses will be performed based on the observed data. No imputation will be done for missing data. Baseline is defined as described in Section 5.3. See Protocol Appendix 9 for a list of laboratory parameters. Laboratory toxicity grades will be assigned based on DMID (see Section 15.8 Appendix 8: Laboratory Parameters and Toxicity Grades) by the laboratory,

with the exception of Lymphopenia (as there is no DMID grade). Lymphopenia will be graded as per CTCAE v4.03.

Calcium, will be presented as hypercalcaemia and hypocalcaemia separately (with each subject appearing in both categories) and similarly for sodium (hypernatremia, hyponatremia), potassium (hyperkalemia, hypokalemia), and glucose (hyperglycemia, hypoglycemia).

Listings will be generated for all laboratory results and for Grade 3 or Grade 4 laboratory toxicity results [L13.13 – L13.24, L23.14 - L23.26].

If a numeric laboratory value, has a non-detectable level reported in the database, then typically the numeric value is missing, and a character value starting with '<x' or '>x' is present. A numeric value will be derived using the number of decimal places in the observed character values i.e.

- 2 Decimal Places = '< x 'becomes x -0.01
- 1 Decimal Place = '> x' becomes x + 0.1
- 0 Decimal Places = '< x' becomes x 1

## 8.3.1. Laboratory Descriptive Statistics by Visit

Descriptive statistics for each analyte will be displayed for each visit for both the Year 1 and Year 1&2 reporting separately. The tables will display the mean value, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum. No statistical tests will be performed [T13.55, T13.59, T13.63, T13.67, T13.74, T23.49, T23.53, T23.57, T23.61, T23.68].

A line graph will be produced for each analyte which displays the mean value (±SE) by visit and treatment group for both Year 1 and Year 1&2 separately [F13.01-F13.05, F23.01-F23.05].

## 8.3.2. Laboratory Toxicity ≥ 2 Grade Shift Post-Baseline

Toxicity grade shifts from baseline of  $\geq 2$  grades will be summarized during treatment for each laboratory parameter within each laboratory category (hematology, liver function, electrolytes, other chemistries, urinalysis and immunoglobulins) for Year 1 and Year 1&2 separately. The table will display the number and percentage of subjects with at least one  $\geq 2$  grade shift as well as the specific shift categories: Grade 0 to 2, Grade 0 to 3, Grade 0 to 4, Grade 1 to 3, Grade 1 to 4 and Grade 2 to 4 [T13.57, T13.61, T13.65, T13.69, T13.72, T13.76, T23.51, T23.55, T23.59, T23.63, T23.66, T23.70].

## 8.3.3. Laboratory Reference Range Shifts from Baseline by Visit

For laboratory tests without toxicity grades, shifts relative to the normal range will be summarized for each analyte as shifts 'to low' and shifts 'to normal/high.' For the 'to low' category the percentage of subjects with at least one low post-baseline value relative

to the baseline will be displayed using the categories: remained low and normal/high to low. For the 'to normal/high' category the percentage of subjects with at least one normal/high post-baseline value relative to baseline will be displayed using the categories: remained normal/high and low to normal/high. No statistical tests will be performed. This analysis will be performed for Year 1 and Year 1&2 separately [T13.58, T13.62, T13.66, T13.70, T13.73, T23.52, T23.56, T23.60, T23.64, T23.67].

A laboratory value that is above the testing laboratory's normal range will be considered a high abnormal laboratory value. A laboratory value that is below the testing laboratory's normal range will be considered a low abnormal value.

## 8.3.4. Immunoglobulin Reference Range Shifts from Baseline by Visit

For immunoglobulins (IgA, and IgM) reference range shifts will be summarized across all visits based on the baseline normal range category. For subjects with immunoglobulin values below the LLN, the number and percentage of subjects who 'remained low' or went 'to normal/high' post-baseline will be summarized. Similarly, for subjects with immunoglobulin values within the normal range or above the ULN, the number and percentage of subjects who 'remained normal/high' or went 'to low' post-baseline will be summarized. This analysis will be performed for Year 1 and Year 1&2 separately [T13.77, T23.71].

## 8.3.5. Worst Laboratory Toxicity Grade Post-Baseline

Laboratory toxicity will be graded using grades corresponding to mild, moderate, severe, and life-threatening when possible. The worst laboratory toxicity grade for each laboratory parameter within each laboratory category (hematology, liver function, electrolytes, other chemistries, urinalysis and immunoglobulins) during Year 1 and Year 1&2 separately will be presented. Data for both scheduled and unscheduled visits will be included. For calcium, sodium, potassium and glucose, grades associated with hypo- and hyper- conditions will be included [T13.56, T13.60, T13.64, T13.68, T13.71, T13.75, T23.50, T23.54, T23.58, T23.62, T23.65, T23.69].

## 8.3.6. Immunoglobulin Below LLN by Visit

The number and percentage of subjects with immunoglobulin values (IgG, IgA, and IgM) below the LLN at each visit will also be presented for all subjects and then repeated for subjects ≥ LLN at baseline for Year 1 and Year 1&2 separately. No statistical test will be performed [T13.78, T13.79, T23.72, T23.73].

## 8.3.7. Immunoglobulin Relative to LLN by Visit

The number and percentage of subjects with immunoglobulin values (IgG, IgA, and IgM) greater than or equal to the LLN at each visit will also be presented for all subjects and then repeated for subjects < LLN at baseline for Year 1 and Year 2 separately. No statistical test will be performed [T13.80, T13.81, T23.74, T23.75].

## 8.3.8. Immunogenicity

For the immunogenicity assessment for belimumab, two types of antibody assays will be performed, i.e. a binding assay and neutralizing assay. For the immunogenicity assessment for rituximab only a binding assay will be performed. For the binding assay, there will be 3-testing steps. A screening assessment is performed which produces a result of positive or negative. Confirmed positive samples will be further characterised for a relative level of binding (titre value). Subjects will be viewed as positive for antidrug antibody (ADA) if the confirmation assay is positive. Subjects, who confirm positive in the anti-belimumab ADA assay, will be evaluated for the presence of neutralising antibody (Nab) response with the NAb assay, which again produces a result of positive or negative.

For incidence of subjects with positive binding antibody during the study period, a table will be produced summarizing results for the binding antibody assay by treatment group and visit. The table will include the number and proportion of subjects in each results category for each visit in the study period (including early withdrawal visit). Binding confirmatory assay results will be categorized as negative, persistent positive (defined as a positive immunogenic response at least two consecutive assessments during the study period or a single result at the final assessment in the study period) or transient positive (defined as a single positive immunogenic response that does not occur at the final assessment in the study period).

Results will be summarized by visit and by treatment group for belimumab (Year 1 and Year 2, separately) and for Arms A and B only for rituximab (Year 1) [T13.82 T13.83, T23.76]. A listing of immunogenicity results will also be presented [L13.33, L23.33].

## 8.3.9. Further Research Samples

Blood leukocyte analysis and B cell receptor samples collected at selected sites in the USA will be reported separately and are not considered in this RAP.

B Cell subsets collected at selected sites in the European Union (EU) will be reported separately and are not considered in this RAP.

## 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including vital signs will be based on GSK Core Data Standards, unless otherwise specified.

## 8.4.1. Vital Signs

A summary of vital signs and change from baseline in vital signs will be presented by visit for Year 1 and Year 2 separately. Weight will be included in these summaries [T13.84, T13.85, T23.77, T23.780].

## 8.4.2. Neurological Assessment

Findings consistent with the diagnosis of Progressive Multifocal Leukoencephalopathy (PML) will be recorded as adverse events.

## 9. HEALTH OUTCOMES ANALYSES

Health outcomes reporting will be conducted on the MITT population, following the principles of the Efficacy analysis.

Additional details for the Health Outcome scales are provided in the appendix: Lupus Qol (Section 15.6.10); WPAI (Section 15.6.11); FACIT-Fatigue Scale (Section 15.6.12).. A listing of all health outcomes endpoints will be presented [L24.01-L24.03].

Exit interviews assessing patients experience of the clinical trial will be databased and reported separately.

The Health Outcome scales are completed by the subject and are very subjective, therefore, all data after the COVID-19 environment onset date (Section 15.6.16) is very likely to be either missing due to the pandemic or affected by the pandemic. It is also expected that the Health Outcomes data collected at different stages of the COVID-19 pandemic may be affected in different ways. As per the second additional analysis for the primary Efficacy endpoint, there may be intangible ways that the data may have been affected even if it has been collected, therefore we cannot distinguish between affected and unaffected data after the COVID-19 environment onset date.

For these reasons, additional analyses defined below have been added for Week 52 and Week 64. A hypothetical strategy was already proposed to deal with missing data due to study withdrawal and this has been expanded to also define the COVID-19 environment onset date as an Intercurrent Event for any subject who has their (scheduled) Week 52 (or Week 64) assessment on or after the onset date. The data for these subjects will be treated as missing values and will be assumed to be Missing At Random (MAR). It will be imputed using Multiple Imputation methods, which take into account the subjects baseline characteristics and their existing pre-COVID data.

The analysis for Week 104 has not been modified as all observed Week 104 data will be collected after the COVID-19 environment onset date, so the Multiple Imputation approach will not be possible. This means that the results should be interpreted with caution.

Additional post-SAC analyses may be carried out to assess the impact of the COVID-19 pandemic on the Health Outcomes data.

## 9.1. Statistical Methodology Specification for Continuous Endpoints

#### **Endpoints**

For all reported timepoints upto Week 52 (Year 1 reporting) and upto week 104 (Year 2 reporting):

Patient Global Assessment (PtGA) of Disease Activity

Change from baseline in PtGA by visit [T14.01, T24.01].

#### LupusQoL Domain Scores

• Change from baseline in each of the 8 LupusQoL Domain scores by visit [T14.02, T24.02].

## FACIT-Fatigue Scale Score

Change from baseline in FACIT-Fatigue Scale score by visit [T14.03, T24.03].

Work Productivity and Activity Impairment (WPAI)

- Change from baseline in WPAI percent overall work productivity impairment by visit [T14.05, T24.05].
- Change from baseline in WPAI percent activity impairment score by visit [T14.06, T24.06].

#### **Derivation**

Derivation of the endpoints is provided in Section 15: Lupus Qol (Section 15.6.10); WPAI (Section 15.6.11); FACIT-Fatigue Scale (Section 15.6.12).

## **Strategy for Intercurrent (Post-Randomization) Events**

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subjects not had missing data.

## Imputation of Data for Missed Visits, and Following Study Withdrawal

- A bayesian repeated measures normal model will be fitted to the observed data, using a
  Markov Chain Monte Carlo approach, adjusting for treatment group, baseline SLEDAI-2K
  score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline
  corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day). Non-informative
  priors will be used
- Quasi-independent samples will be drawn from the posterior distributions for the parameters
  of the multivariate normal distribution for each treatment group and each missingness
  pattern.
- Each sample leads to a separate imputed dataset, in which the missing values are replaced by values drawn randomly from their conditional distribution. This distribution is based on the observed data and the covariates for that subject using the imputation model and the sampled parameter values.

•

These steps will be repeated at least 1000 times.

## **Model Specification**

- Each imputed dataset will be analyzed using ANCOVA to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score (≤9 vs. ≥10), baseline immunosuppressant use (use vs. non-use), and baseline corticosteroid dose (prednisone equivalent ≤10 mg/day vs. >10 mg/day) and baseline value.
- The resulting treatment differences and their SEs will be combined across imputations using Rubin's rules.

## Model Checking & Diagnostics

The Kolmogorov-Smirnov D statistic will be used to test the assumption of normality. Residuals will be reviewed to assess the homogeneity of variance assumption.

#### **Model Results Presentation**

The tables will display:

- Baseline: the number subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, maximum for each arm
- At each visit:
  - the number subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum
  - LS Mean, and standard error of the LS Mean for each arm at Weeks 52, 64 and 104.
  - the treatment difference and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
  - the p-value for treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

# 9.1.1. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic (Continuous Endpoints upto Week 52 and Week 64)

The analysis will be repeated, but visits that were conducted on or after the COVID-19 environment onset date (Section 15.6.16) will be considered as impacted and hence removed from the analysis, as if the subjects had withdrawn.

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subjects not had missing data (including the missing data from the removal of impacted COVID-19 visits). Weeks 72 and 104 are anticipated to have too much data post the COVID-19 environment onset date and hence will not be included.

## Patient Global Assessment (PtGA) of Disease Activity

Change from baseline in PtGA by visit [T14.08,T24.08].

#### LupusQoL Domain Scores

• Change from baseline in each of the 8 LupusQoL Domain scores by visit [T14.09,T24.09].

#### FACIT-Fatigue Scale Score

• Change from baseline in FACIT-Fatigue Scale score by visit [T14.10,24.09]

## Work Productivity and Activity Impairment (WPAI)

- Change from baseline in WPAI percent overall work productivity impairment by visit [T14.12, 24 12]
- Change from baseline in WPAI percent activity impairment score by visit [T14.13, 24.13].

For change from baseline endpoints, a plot of LS means +/- SE by visit and treatment group will be provided.[Year 1: F14.01, Year 1 and 2 combined, but only up to Week 64: F24.01-24.06].

## 9.2. Statistical Methodology Specification for Proportion Endpoints

## **Endpoint / Variables**

 The proportion of participants with an improvement in FACIT-fatigue score exceeding the minimal clinically important difference (MCID is >=4) by visit.

#### Derivation

Derivation of the FACIT endpoint is provided in Section 15.6.12. A subject is considered to have an improvement exceeding the minimal clinically important difference if they have  $\geq$ 4 points improvement in their FACIT-Fatigue Scale score from baseline.

Imputation of Data for missed visits, and following study withdrawal...

Missing Data will be imputed as detailed in Section 9.1.1, then categorized as Responder/Non-Responder using the derivation above. For consistency of results, the same seed will be used for the imputation of missing data on the continuous FACIT scale and the imputation on the continuous scale that is then dichotomized into the binary response.

## **Model Specification**

- Each imputed dataset will analyzed using the proposed statistical analyses planned for the primary endpoint. The FACIT-fatigue score at baseline will also be included as a covariate.
- The resulting Odds Ratios and their SEs will be combined across imputations using Rubin's rules.

## **Model Checking & Diagnostics**

 The model and diagnostics checks proposed for the primary endpoint will be repeated for this endpoint.

#### **Model Results Presentation**

- For each endpoint a table [T14.04, T24.04]. will display:
  - the number, percentage, SE of percentage, and the 95% CI for the percentage of subjects achieving a response by treatment group,
  - the observed difference in percentage of responders for the comparison of Arm B vs Arm A; and Arm B vs Arm C,
  - the odds ratio and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C at Weeks 52, 64 and 104.
  - the p-value for the odds ratio the treatment difference for Arm B vs Arm A at Weeks 52, 64 and 104.

## 9.2.1. Additional Analyses to Assess the Impact of the Coronavirus Disease 2019 (COVID-19) Pandemic

The analysis will be repeated however visits that were conducted on or after the COVID-19 environment onset date (Section 15.6.16) will be considered as impacted and hence removed from the analysis, as if the subjects had withdrawn.

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subjects not had missing data (including the missing data from the removal of impacted COVID-19 visits). Weeks 72 and 104 are anticipated to have too much data post the COVID-19 environment onset date and hence will not be included.

The proportion of participants with an improvement in FACIT-fatigue score exceeding the minimal clinically important difference (MCID is >=4) by visit [T14.11, T24.11].

## 9.3. Health Care Resource Utilization

The health care resource utilization (HCRU) data will be used to conduct exploratory economic analyses of:

- Number of outpatient/hospital clinic visits
- Number of emergency room/urgent care facility visits
- Number and duration of in-patient hospitalizations (total nights, including duration by wards [intensive care unit vs. general ward])
- Use of over the counter (non-prescription) medication.

These data will be provided by CRF Health, and planned analyses will be described in a separate document

A listing of data will be provided at Year 2 [L24.04]. Health care resource utilization will be summarised at Week 52 for Year 1 (T14.07), and at Week 104 for Year 1&2 (T24.07).

Duration of hospitalization will be summed for subjects with more than 1 hospitalisation. Subjects with ongoing hospitalization at Week 52 will be truncated for the Week 52 (Year 1) summary. Subjects with ongoing hospitalization at Week 104 will be truncated for the Week 104 (Year 2) summary at the last known date of hospitalization (i.e. including post study hospitalization if the hospitalization is ongoing at Week 104).

If subjects are withdrawing due to hospitalization then an additional exploratory analysis will be performed shortly after the Statistical Analysis Complete milestone.

## 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

Biomarker Endpoints, Autoantibodies, complement, and peripheral B lymphocytes (referred to as B cells) will be collected per the study calendar (Section 15.2 Appendix 2: Schedule of Activities). The peripheral B lymphocytes will be measured (using FACS analysis). The specific biomarkers collected and analyzed are listed in Table 4:

Table 4 Biomarkers for Analysis

| Autoantibodies | Immunoglobulin |
|---|---|
| aCL (IgA, IgG, IgM) | IgG, IgM, and IgA |
| ANA | B cells (present in tables in this order) |
| Beta-2-glycoprotein | CD19+ Total B cells (cells/mL) |
| (IgA, IgG, IgM) | |
| Lupus anticoagulant | B cells CD20+ (cells/mL and % of CD19+ Total B cells) |
| Anti-dsDNA | Naive B cells IgD+ (cells/mL and % of CD19+ Total B cells) |
| | Naive CD20+ CD27- (cells/mL and % of CD19+ Total B cells) |
| Extractable nuclear antigens (ENAs) | Activated Total B cells CD95+ (cells/mL and % of CD19+ Total B cells) |
| Anti-Ribosomal-P; | Memory CD20+ CD27+ (cells/mL and % of CD19+ Total B cells) |
| | Non-switched memory CD27+ IgD+ (cells/mL and % of CD19+ |
| Anti-RNP-70; | Total B cells) |
| | Switched memory CD27+ IgD- (cells/mL and % of CD19+ Total B |
| Anti-SS-A; | cells) |
| | Plasmablasts CD27b CD38b (cells/mL and % of CD19+ Total B |
| Anti-SS-B | cells) |
| | Plasmablasts CD20+ CD27b CD38b (cells/mL and % of CD19+ |
| Anti-Smith | Total B cells) |
| | Plasmablasts CD20- CD27b CD38b (cells/mL and % of CD19+ |
| Complement | Total B cells) |
| | Transitional CD10+ CD24b CD27- CD38b (cells/mL and % of |
| C3 | CD19+ Total B cells) |
| | Transitional CD24b CD27- CD38b (cells/mL and % of CD19+ Total |
| C4 | B cells) |
| T cells | Cytokines |
| CD3+ Total T cells | BLyS (Total and Free) |
| (/uL) | |
| CD8+ T cells (/uL) | |
| CD4+ T cells (/uL) | |

For the duration of the study, biomarker data (serum immunoglobulin isotypes IgA and IgM and B cell results) that have the potential to unblind the study team will not be transferred to the blinded study team. Instead, blinded datasets will only contain data from the baseline visit (hence not impacted by treatment group). These datasets will

display the format for the real datasets which will be received following unblinding. This will ensure that programs written using blinded data will still run on the real treatment codes and real unblinded data following the first database lock.

## 10.1. Biomarker Change and Percent Change from Baseline Analyses

#### **Endpoints**

The change from baseline and percent change (not for % endpoints) from baseline will be evaluated by visit for each of the biomarkers listed in Table 4 [T15.01-15.02, T15.04-T15.07, T15.09-T15.12, T15.14-T15.15, T25.01-25.02, T25.04-T25.07, T25.09-T25.12, T25.14-T25.15,]. Tables of descriptive statistics for changes in Year 2 relative to at the end of Year 1 will be summarised for immunoglobulins, auto-antibodies and B-Cells [T25.21, T25.22,T25.23].

## **Population of Interest**

The Intent-to-Treat population will be used for the analysis.

## Intercurrent Event Strategy

The Year 1 analyses will be performed on the observed data up to IP discontinuation. No imputation will be done for missing data.

The Year 1&2 analyses will be performed on the observed data for subjects who completed Week 52 on treatment (Ongoing and on treatment at Week 52 analysis as defined in Section 7.1.5). No imputation will be performed for missing data (data post re-start Belimumab will not be considered.

## **Model Specification**

Immunoglobulins and Complement

An ANCOVA will be used to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score ( $\leq 9 \text{ vs.} \geq 10$ ), baseline immunosuppressant use (use vs. non-use), baseline corticosteroid dose (prednisone equivalent  $\leq 10 \text{ mg/day vs.} > 10 \text{ mg/day}$ ), and baseline value (continuous).

If the distribution of the observed data is not consistent with conducting ANCOVA then a non-parametric rank ANCOVA will also be conducted.

Auto-Antibody, B-Cells, T-Cells, and BLyS (Total and Free):

A Rank ANCOVA will be used to evaluate the treatment effect controlling for treatment group, baseline SLEDAI-2K score ( $\leq 9$  vs.  $\geq 10$ ), baseline immunosuppressant use (use vs. non-use), baseline corticosteroid dose (prednisone equivalent  $\leq 10$  mg/day vs.  $\geq 10$  mg/day), and rank baseline value (continuous).

#### Model Checking & Diagnostics

For the ANCOVA analysis the Kolmogorov-Smirnov D statistic will be used to test the assumption of normality. Residuals will be reviewed to assess the homogeneity of variance assumption.

#### **Model Results Presentation**

The tables will display:

- Baseline: the number subjects, number of subjects, mean, standard error, standard deviation, median, 25th percentile, 75th percentile, minimum, maximum for each arm
- the number of subjects, mean, standard error, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum, and maximum, for each arm at each visit
- For ANCOVA analysed endpoints the LS Mean, standard error of the LS Mean, treatment difference for each arm, and 95% confidence interval (CI) for the comparison of Arm B vs Arm A; and Arm B vs Arm C will be presented at Weeks 52, 64, and 104
- For all endpoints the p-value for treatment difference for Arm B vs Arm A will be presented at Weeks 52, 64, and 104.

For change from baseline endpoints, a plot of LS means +/- SE or Median +/- Quartiles (dependent on observed data distribution) by visit and treatment group will be provided.

There will also be additional reporting of lab parameters (Haematology, chemistry, urinalysis and other chemistries) to explore the changes in Year 2 relative to at the end of Year 1. Descriptive statistic tables considering the change from Week 52 by visit for Year 2 will be produced [T25.16-25.19].

## 10.2. Shifts in Immunoglobulins, Autoantibodies, and Complement by Visit

## Endpoints [T15.03, T15.08, T15.13, T25.03, T25.08, T25.13].

Shift tables will be used to summarize the changes in immunoglobulins, autoantibodies, and complement by treatment group and visit. Autoantibodies will be evaluated for shifts from positive to negative. Immunoglobulins and complement will be evaluated for shifts from Low to Normal/High.

| Autoantibody | Positive | Negative |
|---|---|---|
| Anti-dsDNA | >=30 IU/mL | <30 IU/mL |
| ANA | >=80 Titer | <80 Titer |
| aCL | If any of the three aCL | If at least 1 is non-missing |
| | parameters, IgG (>=14 | then aCL is negative; |
| | U/mL), IgA (>=11 U/mL) or | otherwise aCL is missing. |
| | IgM (>=12 U/mL), is positive. | |
| Beta-2-glycoprotein isotypes: | ≥21 U/mL | <21 U/mL |
| IgA, IgG, IgM | | |
| Lupus anticoagulant | N/A | |
| ENAs | > Upper limit of normal range | ≤ Upper limit of normal range |
| Cytokines | | |
| BlyS (Total and Free) | <75 <sup>th</sup> percentile | >=75 <sup>th</sup> percentile |
| Ig and Complement | Low | Normal/High |
| IgG | <6.94 g/L | ≥6.94 g/L |
| IgA | <0.81 g/L | ≥0.81 g/L |
| IgM | <0.48 g/L | ≥0.48 g/L |
| C3 | <90 mg/dL | ≥90 mg/dL |
| C4 | <10 mg/dL | ≥10 mg/dL |

#### Statistical Analysis

Fisher's exact test will be performed within each baseline category to evaluate the treatment effect at Week 52 only.

#### **Summary Measure**

The difference in proportions Arm B (Combination)— Arm A (Control) will be used to measure the treatment effect.

#### **Population of Interest**

The Intent-to-Treat population will be used for the analysis.

## Intercurrent Event Strategy

These analyses will be performed on the observed data up to IP discontinuation. No imputation will be done for missing data.

## **Variables**

• Immunoglobulins, autoantibodies, and complement endpoints evaluated one at a time.

Treatment (belimumab plus rituximab=1, belimumab plus placebo=0)

#### **Results Presentation**

For IgG, IgA, IgM, C3,C4, and C3 and C4 combined baseline data will be summarized as the number and percent of subjects who are low or normal/high at baseline. For post-baseline visits the data will be summarized by baseline status defined as low or normal/high. Among subjects low at baseline the shifts presented will be low to normal/high and low to low. Among subjects normal/high at baseline, the shifts presented will be normal/high to normal/high and normal/high to low.

For anti-dsDNA, ANA, aCL, Beta-2-glycoprotein, Lupus anticoagulant, ENAs and BlyS, baseline data will be summarized as the number and percent of subjects who are positive and negative at baseline. For post-baseline visits the data will be summarized by baseline status defined as positive or negative. Among subjects positive at baseline, the shifts presented will be positive to negative and positive to positive (no change). Among subjects negative at baseline, the shifts presented will be negative to negative (no change) and negative to positive.

## **Subgroup Analyses**

Subgroup analyses will not be conducted

## 11. PHARMACOKINETIC ANALYSES

## 11.1. Primary Pharmacokinetic Analyses

Descriptive statistics for serum belimumab (from all three treatment arms combined) and rituximab concentrations will be displayed for each visit for Year 1 and for Years 1&2 Combined. The tables will display the mean value, standard deviation, 95% confidence interval, geometric mean, geometric standard deviation, geometric 95% confidence interval, coefficient of variation (%), median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, and maximum. No statistical tests will be performed [T16.01, T16.02, T26.01].

A line graph will be produced which displays the median belimumab or rituximab concentration values along with 25<sup>th</sup> and 75<sup>th</sup> percentiles by visit Year 1 and for Years 1&2 Combined [F16.01, F16.02, F26.01].

A listing of serum belimumab and rituximab PK concentration-time data will be presented [L16.01, L16.02, LL26.01].

## 11.1.1. Endpoint / Variables

## 11.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Reporting Standards for Pharmacokinetic).

## 11.1.2. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic PK population, unless otherwise specified.

## 11.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical Principals.

Unless otherwise specified, endpoints / variables defined in Section 11.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

## 12. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

## 12.1. Statistical Analyses / Methods

There will not be a formal requirement to carry out a population pharmacokinetic (PopPK) analysis for this study. However, depending on the study results a PopPK analysis may be performed on a post-hoc basis to quantity the combined effects of belimumab and rituximab in an adult SLE population with respect to belimumab PK, the pharmacological response, and efficacy and safety end-points.

- To develop a PopPK model that characterizes the PK disposition of belimumab following sub-cutaneous administration in adult subjects with SLE.
- Evaluate the potential effect of rituximab administration on belimumab PK parameters.
- Estimate the individual PK parameters for each subject in the study receiving belimumab and summarise across the study.
- Evaluate the effect of belimumab exposure on the response of selected biomarkers, efficacy and safety end-points when dosed alone and in combination with rituximab.

Belimumab serum concentration-time data will be analyzed using a non-linear mixed-effects modelling approach. Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively. All pharmacokinetic data will be stored in the Archives, GlaxoSmithKline Pharmaceuticals, R&D.

## 13. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

Pharmacokinetic/Pharmacodynamic (PD) analyses are not prospectively planned for this study. Based on the results obtained, exploratory analyses may be performed on an ad hoc basis.

## 14. REFERENCES

Buyon JP, Petri MA, Kim MY, et al. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: A randomized trial. Ann Intern Med 2005;142(12 Pt 1):953-62.

Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Tables, May 2001.http://www.niaid.nih.gov/LabsAndResources/resources/DMIDClinRsrch/Document s/dmidadulttox.doc

Franklyn K, Chak Sing Lau, Sandra V Navarra, Worawit Louthrenoo, Aisha Lateef, Laniyati Hamijoyo, C Singgih Wahono, Shun Le Chen, Ou Jin, Susan Morton, Alberta Hoi, Molla Huq, Mandana Nikpour, Eric F Morand, for the Asia-Pacific Lupus Collaboration. Definition and initial validation of a Lupus Low Disease Activity State (LLDAS). Ann Rheum Dis 2016;75:1615–1621

Gladman DD, Ibanez D, Urowitz MB. Systemic lupus Erythematosus disease activity index 2000. J Rheumatol 2002;29(2):288-91.

Mehrotra D V, Fang Liu, Thomas Permutt. Missing data in clinical trials: control-based mean imputation and sensitivity analysis. Pharmaceutical Statistics 2017; 16: 378-392

Neergard. Reducing the risk of blood thinners. Associated press, September 2006.

Oon S, Molla Huq, Vera Golder, Pei Xuan Ong, Eric F Morand, Mandana Nikpour. Lupus Low Disease Activity State (LLDAS) discriminates responders in the BLISS-52 and BLISS-76 phase III trials of belimumab in systemic lupus erythematosus. Ann Rheum Dis 2019; 78: 629-633

Petri M, Buyon J, Kim M. Classification and definition of major flares in SLE clinical trials. Lupus. 1999;8:685-91.

Petri M, Kim MY, Kalunian KC, et al. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med 2005;353(24):2550-8.
# 15. APPENDICES

# 15.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 15.1.1. Exclusions from Per Protocol Population

The per protocol population will be based on the review of the important protocol deviations as detailed in PDMP review document

Important protocol deviations in these categories of the PDMP will be assessed as detailed for exclusion from the per protocol population

### ELIGIBILITY CRITERIA NOT MET

Subjects who do not meet the following criteria

Did not have a clinical diagnosis of SLE according to the ACR criteria (Inclusion Criterion 2).

Did not have clinically active SLE disease defined as a SLEDAI-2K score  $\geq 6$  at screening (Inclusion Criterion 3)

Did not have unequivocally positive ANA test results from 2 independent time points (Inclusion Criterion 4)

Was not on a stable SLE treatment regimen at baseline as defined in the protocol (Inclusion Criteria 5)

Received an excluded medication prior to Day 0 (Exclusion Criteria 23-26) and adjudicated to have had a reasonable probability of impacting on the assessment of efficacy post Day 1.

# ASSESSMENT OR TIME POINT COMPLETION and VISIT COMPLETION

Missed assessment

Missed SLEDAI-2K assessment at Week 52 will be excuded

Out Of Window Assessment

More than 28 days late for Week 52 visit or Week 52 SLEDAI-2K assessment

WRONG STUDY TREATMENT/ADMINISTRATION/DOSE Study treatment not administered per protocol

Subjects randomised to Arms A or B who did not receive all of both scheduled rituximab / rituximab-placebo infusions

Subjects with 4 or more missed consecutive Belimumab doses.

Subjects with 4 or more missed consecutive Belimumab doses irrespective of subject reinitiating Belimuab injections in the presence of the investigator

Wrong study treatment or assignment administered

Subjects who did not receive their assigned treatment will be assessed on a case by case basis.

### STUDY PROCEDURES

Study blinding/unblinding procedures

Subjects from whom their Investigator/site staff/GSK Clinical team did not remain blinded to treatment assignment through Week 52/Exit visit efficacy evaluation

# OTHER REASONS

As determined during

protocol population review meeting prior to unblinding that are determined to have the potential to impact the efficacy evaluation.

# 15.2. Appendix 2: Protocol Defined Schedule of Activities

Table 5 Double-blind Treatment Phase Procedures: Year 1, Arms A and B

| Double-Blind Treatment Phase Procedures | Screening<br>(35 to | | | | Tre | | | – Arms A | | | | | | Unsched-<br>uled Visit | Early<br>Withdrawal | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | 1 day(s)<br>before<br>D1) | D1<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | (1) | Visit (b) | (8<br>weeks<br>post<br>last<br>dose) |
| Informed consent | Χ | | | | | | | | | | | | | | | • |
| Inclusion and exclusion criteria | Χ | X (m) | | | | | | | | | | | | | | |
| Genetics Informed consent | X (r) | | | | | | | | | | | | | | | |
| Randomization | | Χ | | | | | | | | | | | | | | |
| Assessments: Clinic | | | | | | | | | | | | | | | | |
| Full physical exam including height and weight | X | | | | | | | | | | | | | | | |
| 12-lead ECG | Χ | | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | | |
| Medical history (includes substance usage) | Х | | | | | | | | | | | | | | | |
| Past and current medical conditions including cardiovascular medical history | Х | | | | | | | | | | | | | | | |
| Vital signs | Х | | | | | | | | | | | | | | | |
| Symptom-driven physical exam, vital signs | | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х |
| Weight | | Χ | | | | | | | Χ | | | | Х | | Х | |
| Assessments: Independent Asse | essor | | | | | | | | | | | | | | | |
| SLEDAI-2K: Blinded Assessor (t) | | Χ | | | | Χ | | | Χ | | Χ | | Χ | Χ | Χ | |
| Assessments: Principal Investig | ator | | | | | | | | | | | | | | | |
| SLEDAI-2K: Investigator | Χ | Χ | Χ | | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Χ | |
| C-SSRS Baseline/Screening | Х | | | | | | | | | | | | | | | |
| C-SSRS Since Last Visit | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |

| Double-Blind Treatment Phase Procedures | Screening<br>(35 to | | | | | | | - Arms A | | , | | | | Unsched-<br>uled Visit | Early<br>Withdrawal | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | 1 day(s)<br>before<br>D1) | D1<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | (1) | Visit (b) | (8<br>weeks<br>post<br>last<br>dose) |
| Neurological Assessment | Χ | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х |
| SLE Flare Index (n) | | Χ | Х | | Χ | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | X | |
| SLICC-ACR Damage Index | | Х | | | | | | | | | | | Х | | Х | |
| Physician Global Assessment (PGA) | | Х | Х | | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | |
| Survival Assessment (d) | | | | | | | | | | | | | Х | | | |
| Assessments: Patient Reported | Outcomes (F | ROs) | | | | | | | | | | | | | | |
| Patient Global Assessment (c) | | Χ | | | Χ | Х | | | Χ | | Х | | Х | | Х | |
| FACIT-Fatigue (c) | | Χ | | | Χ | Х | | | Χ | | Χ | | Χ | | X | |
| Lupus QoL (c) | | Χ | | | Χ | Χ | | | Χ | | Χ | | Χ | | X | |
| WPAI: Lupus (c) | | Χ | | | Χ | Х | | | Χ | | Х | | Х | | Х | |
| Post-treatment interview (o) | | | | | | | | | | | | | Χ | | X | |
| Central Laboratory Tests | | | | | | | | | | | | | | | | |
| Drug and alcohol screen | Χ | | | | | | | | | | | | | | | |
| HIV, Hep B and Hep C screen | Χ | | | | | | | | | | | | | | | |
| Pregnancy test (WCBP) (e) | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ |
| Laboratory assessments (include liver chemistries) | Х | Х | Χ | Х | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Х |
| Serum immunoglobulin<br>(IgA, IgM, IgG) | Х | Х | Х | Х | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Х |
| Urinalysis | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Χ | Х | Χ | Χ | Χ | Х |
| Anti-dsDNA/ANA,<br>Complement C3/C4 | Х | Х | Х | | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Extractable nuclear antigens (ENAs) | | Х | | | Χ | | | | Х | | | | Х | | Х | |
| PT/PTT | Χ | Χ | | | Χ | | | | Χ | | | | Χ | Χ | X | |

| Double-Blind Treatment Phase Procedures | Screening<br>(35 to | | | | | | | - Arms A | | ` , | | | | Unsched-<br>uled Visit | Early<br>Withdrawal | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | 1 day(s)<br>before<br>D1) | D1<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | (1) | Visit (b) | (8<br>weeks<br>post<br>last<br>dose) |
| Antiphospholipid antibodies (aCL, lupus anticoagulant, ± beta-2-glycoprotein-1) | | Х | | | X | | | | X | | | | Х | Х | Х | |
| Labs and Biomarkers | | | | l | | | | | | | l | | | l | | |
| B cells subsets | | Χ | Х | | | | Χ | | Х | | Χ | | Х | | Х | Х |
| BLyS Protein | | Χ | | | | | | | | | | | Χ | | Х | |
| Immunogenicity: Belimumab | | Х | X(f) | X(f) | Χ | | | | Х | | | | Х | Х | Х | Х |
| Immunogenicity: Rituximab | | Χ | X(f) | X(f) | Χ | | | | Χ | | | | Х | Х | Х | |
| Pharmacokinetics: Belimumab | | | X(f) | | Χ | | | | Х | | | | Х | Х | Х | Х |
| Pharmacokinetics: Rituximab | | | X(g) | X(g) | Χ | | | | Χ | X(h) | | | | Х | Х | Х |
| Genetic sample | | Х | | | | | | | | | | | | | | |
| Exploratory Further Research | | | | | | | | | | | | | | | | |
| Blood Leukocyte Analysis (PBMC) (p) | | Χ | | | | | | | | | | | Х | | Х | |
| RNA for Interferon Signature | | Χ | | | | | | | | | | | | | | |
| B cell receptor (q) | | Χ | | | | | | | | | | | | Χ | X | |
| B cells subsets – (u) | | Χ | Х | | | | | | | | | | Х | | Х | |
| Study Treatment | | | | • | | | | | , | | • | | , | | | |
| Training on use of Autoinjector | Χ | Χ | | | | | | | | | | | | | | |
| Dispense/Train or Collect<br>Electronic Diary | | Χ | | | | | | | | | | | | | Х | |
| Dispense Belimumab for weekly dosing (SC) | | X (i) | X (s) | | X | Χ | Χ | Χ | | Χ | Х | Х | | | | |
| Rituximab or Rituximab-Placebo (IV) | | | X<br>(j) | X<br>(j) | | | | | | | | | | X<br>(j) | | |
| Discontinue immunosuppressants | | | X | • | | | | | | | | | | | | |
| Initiate corticosteroid taper | | | | | | X (k) | | | | | | | | | | |

| Double-Blind Treatment Phase Procedures | Screening<br>(35 to | | | | Tre | atment | Period - | - Arms A | and B | (a) | | | | Unsched-<br>uled Visit | Early<br>Withdrawal | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | 1 day(s)<br>before<br>D1) | D1<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | (1) | Visit (b) | (8<br>weeks<br>post<br>last<br>dose) |
| Target for steroid corticosteroid dose to reach prednisone equivalent ≤5 mg/day | | | | | | | | | Х | | | | | | | |
| Study Visit Review Procedures | 1 | | 1 | 1 | | | 1 | 1 | 1 | | 1 | 1 | | | | |
| AE/SAE review | | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | X | X | Χ | Χ | X | X | Χ |
| Concomitant medication review (including SLE medications) | Х | Х | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х |
| Review HCRU and Patient Diary | | | Χ | Χ | Χ | X | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | |

- a. Starting at Week 4 and throughout the study period including follow-up, a study visit time window ± 7 days is acceptable. Note: Every effort should be made to schedule the visit in this window, however if the COVID-19 pandemic situation affects the ability to achieve this then, for those COVID-19 specific instances, the visit window can be expanded to ±28 days.
- b. Early Withdrawal Visit 1-4 weeks after last dose for participants that withdraw from the study.
- c. To be conducted prior to clinical assessments.
- d. Survival assessment at Week 52 for participants who withdraw before Week 52.
- e. Serum pregnancy test at Screening; Urine pregnancy test at all other visits, including pregnancy test 16 weeks after last dose of belimumab. The pregnancy test 16 weeks after the last dose of belimumab may be done at home, with the results reported by telephone call to the clinic. See Protocol Section 9 for pregnancy test requirements a.
- f. At Week 4 and Week 6 pre-rituximab/ rituximab-placebo dose.
- g. At Week 4 post-rituximab/rituximab-placebo dose and at Week 6 pre- and post- rituximab/rituximab-placebo dose.
- h. At Week 32 only.
- i. The first dose of belimumab will be administered at the clinic and the subject needs to stay for 3 hours post dose for observation.
- j. Premedication administration will be given 30 minutes prior to each rituximab / rituximab-placebo dose and the subject needs to stay in clinic for 1 hour post dose for observation (i.e., Clinical monitoring including vital signs). If the subject misses the Week 4 dosing visit and dosing will take place during an unscheduled visit, the first dose of rituximab should be scheduled no later than 7 days after Week 4. The second dose of rituximab must be administered at least 2 weeks but not more than 3 weeks after the first rituximab dose. NOTE: Contact Medical Monitor if the date of a) first dose is more than 1 week past week 4, and b) if the date of the second dose of rituximab would exceed 3 weeks after the first dose. During unscheduled visits, procedures for Immunogenicity and PK will follow the schedule for Week 4 and Week 6.
- k. It is recommended that the steroid taper be initiated on Week 12 to reach the target prednisone equivalent of ≤5 mg/day at Week 26, but the taper schedule is at the discretion of the investigator.

- I. Procedures to be performed at Unscheduled Visits are based on reason for Unscheduled Visit, including adverse event or discontinuation of study agent. Guidance is provided in the Study Reference Manual.
- m. The interim medical history, including SLE medications, should be reviewed prior to randomization to assure that the participant's eligibility has not changed.
- n. Blood samples for a B cell receptor analysis should be obtained in the event of a suspected SLE Flare (refer to footnote q).
- o. To be conducted at US sites only.
- p. To be conducted only at US study sites.
- q. To be conducted only at US study sites. B-cell receptor samples are also collected when subjects experience a suspected SLE Flare.
- r. Separate Genetics informed consent as needed per country specific requirements. Genetics informed consent and sample can be obtained any time after baseline.
- s. If a subject happens to be scheduled for an infusion (week 4 and/or 6) on the same day of the week as their normally scheduled belimumab injection, whenever possible, the day of the belimumab injection should be altered within the dosing window to separate the day of the injection from the day of the infusion to allow for appropriate safety monitoring of the infusion. If subject has already self-administered the belimumab dose on the day of IV infusion, contact study Medical Monitor for guidance prior to administering the rituximab/rituximab-placebo dose.
- t. Independent assessor will perform symptom-driven physical examination to include, at a minimum, assessments of eyes, mouth, skin, lungs, cardiovascular system, abdomen, and extremities (including joints). Independent assessors must have a source document (paper record in the study file) where the findings in the clinical exam and laboratory analyses supporting the scoring of S2K are described.
- u. To be conducted only at selected European sites

Table 6 Double-blind Observational Phase Procedures: Year 2, Arms A and B

| | | Obser | vational Perio | d – Arms A | and B (a) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arms A and B Double-blind Observational Phase Procedures (W=Week) | W60 | W64 | W72 | W80 | W88,<br>W96 | W104 | Unscheduled<br>Visit (e) | Early<br>Withdrawal<br>Visit (f) | Follow-up visit<br>(8 weeks post<br>last dose) (j) |
| Assessments: Clinic | | | • | | | | | | |
| Symptom-driven physical exam, vital signs | Х | Χ | Х | Х | Х | Х | X | Χ | Х |
| Weight | | | | | | Х | | Χ | |
| Assessments: Independent Assessor | | | | | | | | | |
| SLEDAI-2K: Blinded Assessor (m) | | Х | | Х | | Х | X | Χ | |
| Assessments: Principal Investigator | | | | | | | | | |
| SLEDAI-2K: Investigator | Х | Χ | Х | Х | Х | Х | X | Χ | |
| C-SSRS Since Last Visit | Х | Х | Х | Х | Χ | X | X | Χ | Х |
| Neurological assessment | Х | Х | Х | Х | Х | Х | X | Χ | Х |
| SLE Flare Index (g) | Х | Х | Х | Х | Х | Х | X | Χ | |
| SLICC-ACR Damage Index | | | | | | Х | | Χ | |
| Physician's Global Assessment (PGA) | Х | Х | Х | Х | Х | Х | Х | Х | |
| Survival assessment (c) | | | | | | Х | | | |
| <b>Assessments: Patient Reported Outcomes</b> | (PROs) | | | | | | | | |
| Patient Global Assessment (b) | | Х | Х | | | Х | | Χ | |
| FACIT-Fatigue (b) | | Х | Х | | | Х | | Χ | |
| Lupus QoL (b) | | Х | Х | | | Х | | Χ | |
| WPAI: Lupus (b) | | Х | Х | | | Х | | Χ | |
| Exit Interview (h) | | | | | | Х | | Χ | |
| Central Laboratory Tests | | | | | | | | | |
| Urine pregnancy test (WCBP) (d) | Х | Х | Х | Х | Х | Х | X | Χ | Х |
| Laboratory assessments (include liver chemistries) | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Serum immunoglobulin (IgA, IgM, IgG) | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Urinalysis | Х | Х | Х | Х | Χ | Х | Х | X | Х |
| Anti-dsDNA/ANA, Complement C3/C4 | Х | Х | Х | Х | Χ | Х | Х | X | Х |
| Extractable nuclear antigens (ENAs) | Х | | | Х | | Х | | Χ | |
| PT/PTT | | | | Х | | Х | Х | Х | |

| | | Obser | vational Perio | d – Arms A | and B (a) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arms A and B Double-blind Observational Phase Procedures (W=Week) | W60 | W64 | W72 | W80 | W88,<br>W96 | W104 | Unscheduled<br>Visit (e) | Early<br>Withdrawal<br>Visit (f) | Follow-up visit<br>(8 weeks post<br>last dose) (j) |
| Antiphospholipid antibodies (aCL, lupus anticoagulant, ± beta-2-glycoprotein-1) | Х | | | Х | | Х | Х | Х | |
| Labs and Biomarkers | | | | | | | | | |
| B cells subsets | Х | | | Χ | | Χ | | Χ | X |
| BLyS Protein | Х | Χ | Χ | Χ | Χ | Χ | | Χ | |
| Immunogenicity: Belimumab | | | | Χ | | X | X | Χ | X |
| Immunogenicity: Rituximab | | | | | | | X | Χ | |
| Pharmacokinetics: Belimumab | Х | Χ | Χ | Χ | | | X | Χ | X |
| Pharmacokinetics: Rituximab | | | | | | | X | Χ | X |
| Exploratory Research | | | | | | | | | |
| Blood Leukocyte Analysis (PBMC) (k) | | | | Χ | | X | | Χ | |
| B cell receptor (I) | | | | | | X | X | Χ | |
| B cell subsets (n) | Х | | | Χ | | Χ | | Χ | |
| Study Treatment | | | | | | | | | |
| Collect Electronic Diary | | | | | | Х | | Χ | |
| Study Visit Review Procedures | | | | | | | | | |
| AE/SAE review | Х | Χ | Χ | Х | Χ | Χ | Х | Χ | X |
| Concomitant medication review (including SLE medications) | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Review HCRU and Patient Diary (i) | Х | Х | Х | Х | Х | Х | Х | Х | |

- a. During this study period including follow-up, a study visit time window ± 7 days is acceptable. Note: Every effort should be made to schedule the visit in this window, however if the COVID-19 pandemic situation affects the ability to achieve this then, for those COVID-19 specific instances, the visit window can be expanded to ±28 days.
- b. To be conducted prior to clinical assessments.
- c. Survival assessment at Week 104 for participants who withdraw before Week 104.
- d. The pregnancy tests 12 months after the last dose of rituximab / rituximab-placebo (Week 58) and 16 weeks after the last dose of belimumab (Week 68) may be done at home, with the results reported by telephone call to the clinic. See Protocol Section 9 for pregnancy test requirements for participants that withdraw.(Argentina only: In addition to pregnancy testing at the specified clinic visits, a urine pregnancy test is to be performed at home at Week 56, Week 68, Week 76, Week 84, Week 92, and Week 100, with the results reported by telephone call to the clinic.)

- e. Procedures to be performed at Unscheduled Visits are based on reason for Unscheduled Visit, including adverse event or discontinuation of study agent. Guidance is provided in the Study Reference Manual.
- f. Participants who withdraw from the study are required to complete an Early Withdrawal Visit 1-4 weeks after withdrawal from the study.
- g. Blood samples for a B cell receptor analysis should be obtained in the event of a SLE Flare (refer to footnote I).
- h. To be conducted at US sites only.
- i. Diary review is only necessary if the patient receive Belimumab re-start therapy.
- j. Follow up visit is required only for subjects who receive belimumab re-start therapy at any time between Week 52 and Week 104.
- k. To be conducted only at US study sites.
- I. To be conducted only at US study sites. B-cell receptor samples are also collected when subjects experience a SLE Flare.
- m. Independent assessor will perform symptom-driven physical examination to include, at a minimum, assessments of eyes, mouth, skin, lungs, cardiovascular system, abdomen, and extremities (including joints). Independent assessors must have a source document (paper record in the study file) where the findings in the clinical exam and laboratory analyses supporting the scoring of S2K are described.
- n. To be conducted at select European centers.

Table 7 Open-Label Treatment Phase Procedures: Year 1, Arm C

| Treatment Phase Procedures | Screening | | | | | Trea | itment F | eriod – | Arm C ( | a) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | (35 to<br>1 day(s)<br>before D1) | D1,<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | Unsched-<br>uled Visit<br>(h) | Early<br>Withdrawal<br>Visit (b) | Follow-<br>up Visit<br>(8 weeks<br>post last<br>dose) |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | Χ | X (i) | | | | | | | | | | | | | | |
| Genetics Informed consent | X (m) | | | | | | | | | | | | | | | |
| Randomization | | Χ | | | | | | | | | | | | | | |
| Assessments: Clinic | | | | | | | | | | | | | | | | |
| Full physical exam including height and weight | X | | | | | | | | | | | | | | | |
| 12-lead ECG | X | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | |
| Medical history (includes substance usage) | Х | | | | | | | | | | | | | | | |
| Past and current medical conditions including cardiovascular medical history | Х | | | | | | | | | | | | | | | |
| Vital signs | Х | | | | | | | | | | | | | | | |
| Symptom-driven physical exam, vital signs | | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Weight | | Х | | | | | | | Χ | | | | Х | | Х | |
| Assessments: Independent As | sessor | | | | | | | | | | | | | | | |
| SLEDAI-2K: Blinded Assessor (n) | | Х | | | | Χ | | | Х | | Х | | Х | Х | Х | |
| Assessments: Principal Inves | | | | | | | | | | | | | | | | |
| SLEDAI-2K: Investigator | Х | Х | Χ | | Χ | Χ | Χ | Х | Χ | Х | Х | Χ | Χ | Χ | Χ | |
| C-SSRS Baseline/Screening | Χ | | | | | | | | | | | | | | | |
| C-SSRS Since Last Visit | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Х | Χ | Х | Χ |
| Neurological Assessment | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Χ | Χ | Χ | Х |
| SLE Flare Index (j) | | Х | Х | | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | - |

| Treatment Phase Procedures | Screening | | | | | Trea | tment F | eriod – | Arm C ( | a) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D=Day, W=Week) | (35 to<br>1 day(s)<br>before D1) | D1,<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | Unsched-<br>uled Visit<br>(h) | Early<br>Withdrawal<br>Visit (b) | Follow-<br>up Visit<br>(8 weeks<br>post last<br>dose) |
| SLICC-ACR Damage Index | | Χ | | | | | | | | | | | Χ | | Χ | |
| Physician Global Assessment (PGA) | | Х | Х | | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | |
| Survival Assessment (d) | | | | | | | | | | | | | Х | | | |
| Assessments: Patient Reporte | ed Outcomes | (PROs) | | | | | | | | | | | | | | |
| Patient Global Assessment (c) | | Х | | | Χ | Χ | | | Χ | | Х | | Х | | Х | |
| FACIT-Fatigue (c) | | Х | | | Χ | Χ | | | Х | | Χ | | Х | | Х | |
| Lupus QoL (c) | | Х | | | Χ | Χ | | | Х | | Χ | | Х | | Х | |
| WPAI: Lupus (c) | | Χ | | | Χ | Χ | | | Х | | Х | | Х | | Х | |
| Treatment Interview (k) | | | | | | | | | | | | | Х | | Х | |
| Central Laboratory Tests | | | | | | | | | | | | | | | | |
| Drug and alcohol screen | X | | | | | | | | | | | | | | | |
| HIV, Hep B and Hep C screen | Х | | | | | | | | | | | | | | | |
| Pregnancy test (WCBP) (e) | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | Χ |
| Laboratory assessments (include liver chemistries) | Х | Х | Х | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Х |
| Serum immunoglobulin<br>(IgA, IgM, IgG) | Х | Х | Х | Х | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х |
| Urinalysis | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | Χ |
| Anti-dsDNA/ANA,<br>Complement C3/C4 | Х | Х | Х | | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х |
| Extractable nuclear antigens (ENAs) | | Х | | | Х | | | | Х | | | | Х | | Х | |
| PT/PTT | Χ | Χ | | | Χ | | | | Χ | | | | Х | Χ | Х | |
| Antiphospholipid antibodies | | | | | | | | | | | | | | | | |
| (aCL, lupus anticoagulant, ± | | Х | | | Χ | | | | Χ | | | | Х | Χ | Х | |
| beta-2-glycoprotein-1) | | | | | | | | | | | | | | | | |
| Labs and Biomarkers | | | | | | | | | | | | | | | | |
| B cells subsets | | Χ | Χ | | | | Χ | | Χ | | Χ | | Х | | X | Χ |

| Treatment Phase Procedures (D=Day, W=Week) | Screening<br>(35 to | | | | | Trea | tment P | eriod – | Arm C ( | a) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (D-Day, W-Week) | 1 day(s)<br>before D1) | D1,<br>(Base-<br>line) | W4 | W6 | W8 | W12 | W16 | W20,<br>W24 | W26 | W28,<br>W32,<br>W36 | W40 | W44,<br>W48 | W52 | Unsched-<br>uled Visit<br>(h) | Early<br>Withdrawal<br>Visit (b) | Follow-<br>up Visit<br>(8 weeks<br>post last<br>dose) |
| BLyS Protein | | Χ | | | | | | | | | | | X | | X | |
| RNA for interferon signature | | X | | | | | | | | | | | | | | |
| Immunogenicity: Belimumab | | X | Х | Х | Χ | | | | Χ | | | | Х | Χ | Χ | Χ |
| Pharmacokinetics: Belimumab | | | Χ | | Χ | | | | Χ | | | | Х | Х | Х | Χ |
| Genetic sample | | Х | | | | | | | | | | | | | | |
| Exploratory Research | | | | | L | L | | | · | | • | l . | • | | • | |
| B cells subsets (o) | | Χ | Χ | | | | | | | | | | | | Х | |
| B-cell Receptor (I) | | Х | | | | | | | | | | | | Х | Х | |
| Study Treatment | | | | | 1 | T | | | | 1 | ı | 1 | | | • | |
| Training on use of Autoinjector | Х | Χ | | | | | | | | | | | | | | |
| Dispense/Train or Collect<br>Electronic patient diary | | Χ | | | | | | | | | | | | | Х | |
| Dispense Belimumab for weekly dosing (SC) | | X<br>(f) | Х | | Х | Х | Χ | Χ | | Χ | Х | Х | Х | | | |
| Initiate corticosteroid taper | | | | | | (g) | | | | | | | | | | |
| Target for corticosteroid dose to reach prednisone equivalent ≤5 mg/day | | | | | | | | | Х | | | | | | | |
| Study Visit Review Procedure | S | | • | | | | | | | | | | | | | |
| AE/SAE review | | Χ | Х | Х | Х | Х | Χ | Χ | Х | Χ | Χ | Х | Х | Χ | Х | Χ |
| Concomitant medication review (including SLE medications) | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Review HCRU and Patient<br>Diary | | | Х | Х | Х | Χ | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | |

- a. Starting at Week 4and throughout the study period including follow-up, a study visit time window ± 7 days is acceptable. Note: Every effort should be made to schedule the visit in this window, however if the COVID-19 pandemic situation affects the ability to achieve this then, for those COVID-19 specific instances, the visit window can be expanded to ±28 days.
- b. Early Withdrawal Visit 1-4 weeks after last dose for participants that discontinue study and withdraw from the study.
- c. To be conducted prior to clinical assessments.
- d. Survival assessment at Week 52 for participants who withdraw before Week 52.
- e. For WCBP Serum pregnancy test at Screening; Urine pregnancy test at all other visits, including pregnancy test 16 weeks after last dose of belimumab. The pregnancy test 16 weeks after the last dose of belimumab may be done at home, with the results reported by telephone call to the clinic. See Protocol Section 9 for pregnancy test requirements for participants that withdraw.
- f. The first dose of belimumab will be administered at the clinic and the subject needs to stay for 3 hours post dose for observation.
- g. It is recommended that the steroid taper be initiated on Week 12 to reach the target prednisone equivalent of ≤5 mg/day at Week 26, but the taper schedule is at the discretion of the investigator.
- h. Procedures to be performed at Unscheduled Visits are based on reason for Unscheduled Visit, including adverse event or discontinuation of study agent. Guidance is provided in the Study Reference Manual.
- i. The interim medical history, including SLE medications, should be reviewed prior to randomization to assure that the participant's eligibility has not changed.
- j. Blood samples for a B cell receptor analysis should be obtained in the event of a SLE Flare (refer to footnote I).
- To be conducted at US sites only.
- I. To be conducted only at US study sites. B-cell receptor samples are also collected when subjects experience a SLE Flare.
- m. Separate Genetics informed consent as needed per country specific requirements. Genetics informed consent and sample can be obtained any time after baseline.
- n. Independent assessor will perform symptom-driven physical examination to include, at a minimum, assessments of eyes, mouth, skin, lungs, cardiovascular system, abdomen, and extremities (including joints). Independent assessors must have a source document (paper record in the study file) where the findings in the clinical exam and laboratory analyses supporting the scoring of S2K are described.
- o. To be conducted at select European centers.

Table 8 Open-Label Treatment Phase Procedures: Year 2, Arm C

| | | | Treatment F | Period – Arm | C (a) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm C<br>Treatment Phase Procedures<br>(W=Week) | W60 | W64 | W72 | W80 | W88,<br>W96 | W104 | Unscheduled<br>Visit (e) | Early<br>Withdrawal<br>Visit | Follow-up<br>Visit (8<br>weeks post<br>last dose) |
| Assessments: Clinic | | | | | | | | | |
| Symptom-driven physical exam, vital signs | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Weight | | | | | | Х | | Х | |
| Assessments: Independent Assessor | | | | | | | | | |
| SLEDAI-2K: Blinded Assessor (i) | | Х | | Χ | | Х | Х | Х | |
| Assessments: Principal Investigator | | | | | | | | | |
| SLEDAI-2K: Investigator | Х | Х | Х | Χ | Х | Х | Х | Х | |
| C-SSRS Since Last Visit | Х | Х | Х | Χ | X | Х | Х | Х | Х |
| Neurological assessment | Х | Х | Х | Χ | X | Х | Х | Х | Х |
| SLE Flare Index (f) | Х | Χ | X | Χ | X | Х | X | Χ | |
| SLICC-ACR Damage Index | | | | | | X | | Х | |
| Physician Global Assessment (PGA) | Х | X | X | X | X | Х | X | Х | |
| Survival assessment (c) | | | | | | X | | | |
| <b>Assessments: Patient Reported Outcor</b> | mes (PROs) | | | | | | | | |
| Patient Global Assessment (b) | | X | X | | | X | | Χ | |
| FACIT-Fatigue (b) | | X | X | | | X | | Χ | |
| Lupus QoL (b) | | X | X | | | X | | Χ | |
| WPAI: Lupus (b) | | Χ | Χ | | | Х | | Χ | |
| Exit Interview (g) | | | | | | Х | | Χ | |
| Central Laboratory Tests | | | | | | | | | |
| Urine pregnancy test (WCBP) (d) | Х | Х | Х | Х | X | Х | X | X | X |
| Laboratory assessments (include liver chemistries) | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Serum immunoglobulin (IgA, IgM, IgG) | Χ | Х | Χ | Χ | Х | Х | Х | Х | Х |
| Urinalysis | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Anti-dsDNA/ANA, Complement C3/C4 | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Extractable nuclear antigens (ENAs) | Х | | | Х | | Х | | Х | |

| | | | Treatment I | Period – Arm | C (a) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm C<br>Treatment Phase Procedures<br>(W=Week) | W60 | W64 | W72 | W80 | W88,<br>W96 | W104 | Unscheduled<br>Visit (e) | Early<br>Withdrawal<br>Visit | Follow-up<br>Visit (8<br>weeks post<br>last dose) |
| PT/PTT | | | | Х | | Х | Х | Χ | |
| Antiphospholipid antibodies (aCL, lupus anticoagulant, ± beta-2-glycoprotein-1) | Х | | | Х | | Х | Х | Х | |
| Labs and Biomarkers | | | | | | | | | |
| B cells subsets | Χ | | | X | | X | | Χ | Х |
| Immunogenicity: Belimumab | | | | Х | | Х | Х | Χ | Х |
| Pharmacokinetics: Belimumab | | | | X | | X | X | Χ | Х |
| Exploratory Research | | | | | | | | | |
| B cell receptor (h) | | | | | | X | X | Х | |
| Study Treatment | | | | | | | | | |
| Collect Electronic Diary | | | | | | Х | | Χ | |
| Dispense Belimumab for weekly dosing (SC) | Χ | Х | Х | Х | Х | | | | |
| Study Visit Review Procedures | | | | | | | | | |
| AE/SAE review | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medication review (including SLE medications) | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Review HCRU and Patient Diary | Χ | Х | Х | Χ | Х | Х | Х | Х | |

| | | | Treatment F | Period – Arm | C (a) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm C<br>Treatment Phase Procedures<br>(W=Week) | W60 | W64 | W72 | W80 | W88,<br>W96 | W104 | Unscheduled<br>Visit (e) | Early<br>Withdrawal<br>Visit | Follow-up<br>Visit (8<br>weeks post<br>last dose) |

- a. During this study period including follow-up, a study visit time window ± 7 days is acceptable. Note: Every effort should be made to schedule the visit in this window, however if the COVID-19 pandemic situation affects the ability to achieve this then, for those COVID-19 specific instances, the visit window can be expanded to ±28 days.
- b. To be conducted prior to clinical assessments.
- c. Survival assessment at Week 104 for participants who withdraw before Week 104.
- d. The pregnancy test 16 weeks after the last dose of belimumab may be done at home, with the results reported by telephone call to the clinic.
- e. Procedures to be performed at Unscheduled Visits are based on reason for Unscheduled Visit, including adverse event or discontinuation of study agent. Guidance is provided in the Study Reference Manual.
- f. Blood samples for a B cell receptor analysis should be obtained in the event of a SLE Flare (refer to footnote h).
- g. To be conducted at US sites only.
- h. To be conducted only at US study sites. B-cell receptor samples are also collected when subjects experience a SLE Flare.
- i. Independent assessor will perform symptom-driven physical examination to include, at a minimum, assessments of eyes, mouth, skin, lungs, cardiovascular system, abdomen, and extremities (including joints). Independent assessors must have a source document (paper record in the study file) where the findings in the clinical exam and laboratory analyses supporting the scoring of S2K are described.

J.

# 15.3. Appendix 3: Assessment Windows

# 15.3.1. Definitions of Assessment Windows for Analyses

The data is analyzed as per the planned visit assignment.

Exit/withdrawal and unscheduled visits will be slotted to the appropriate planned visit. The assigned visit is based on the interval in which the Study Day for the exit/withdrawal or unscheduled visit falls according to intervals (inclusive) provided below. For completeness, the table also includes visits which are not slotted; these visits will have 'na' for 'not available' listed for the Interval Start and End Day.

| Analysis Set / | Parameter | Target <sup>1</sup> | Analysis | Window | Analysis | Analysis |
|---|---|---|---|---|---|---|
| Domain | (if applicable) | | Timepoint Timepoint | | Timepoint<br>Number⁴ | Timepoint |
| All | All | NA | NA | NA | 10 | Screening |
| Year 1 Treatme | nt Phase visits: | | _ | | | _ |
| All | All | 1 | NA | NA | 20 | Baseline |
| | | 29 | 2 | 35 | 30 | Week 4 |
| | | 43 | 36 | 49 | 40 | Week 6 |
| | | 57 | 50 | 70 | 50 | Week 8 |
| | | 85 | 71 | 98 | 60 | Week 12 |
| | | 113 | 99 | 126 | 70 | Week 16 |
| | | 141 | 127 | 154 | 80 | Week 20 |
| | | 169 | 155 | 175 | 90 | Week 24 |
| | | 183 | 176 | 189 | 100 | Week 26 |
| | | 197 | 190 | 210 | 110 | Week 28 |
| | | 225 | 211 | 238 | 120 | Week 32 |
| | | 253 | 239 | 266 | 130 | Week 36 |
| | | 281 | 267 | 294 | 140 | Week 40 |
| | | 309 | 295 | 322 | 150 | Week 44 |
| | | 337 | 323 | 350 | 160 | Week 48 |
| | | 365 | 351 | 392 | 170 | Week 52 |
| | | 365 | na | Na | 175 | Survival-<br>W52 <sup>2</sup> |
| Year 2 Phase V | isits: | | | | | |
| All | All | 421 | 393 | 434 | 180 | Week 60 |
| | | 449 | 435 | 476 | 190 | Week 64 |
| | | 505 | 477 | 532 | 200 | Week 72 |
| | | 561 | 533 | 588 | 210 | Week 80 |
| | | 617 | 589 | 644 | 220 | Week 88 |
| | | 673 | 645 | 700 | 230 | Week 96 |
| | | 729 | 701 | 742 | 240 | Week 104 |

| Analysis Set / | Parameter | Target <sup>1</sup> | Target <sup>1</sup> Analysis Window | | Analysis | Analysis |
|---|---|---|---|---|---|---|
| Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint<br>Number⁴ | Timepoint |
| | | 729 | na | na | 245 | Survival-<br>W104 <sup>2</sup> |
| | | Na | na | na | 250 | Follow-Up <sup>3</sup> |

# NOTES:

<sup>&</sup>lt;sup>1</sup> Study Day with Baseline/Treatment Start Date as Day 1. Baseline record will be derived in each analysis dataset, analysis visit number will be 15.

<sup>&</sup>lt;sup>2</sup> Survival visit for subjects who withdraw from the double-blind treatment phase but consent to the Week 52 and Week 104 survival assessments.

<sup>&</sup>lt;sup>3</sup> The follow-up visit occurs 8 weeks after last dose of belimumab for subjects who discontinue study treatment and withdraw from the study up to (i) Week 52 in Arms A and B or (ii) Week 104 in Arm C.

<sup>&</sup>lt;sup>4</sup> If there are multiple visits within a visit window, the visit closest to the target date will be used. If there are two visits equidistant from the target date, then the scheduled visit will be given preference, if both are unscheduled then the first assessment will be used.

# 15.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 15.4.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before the first exposure date to study treatment |
| Concomitant | Any medication that is not a prior. Note that medications with partial or missing start and/or stop dates will be assumed to be concomitant unless there is evidence through comparison of partial dates to suggest otherwise |

# 15.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date, having been absent pre- |
| Emergent | treatment, or that worsens relative to the pre-treatment state. |

# 15.5. Appendix 5: Data Display Standards & Handling Conventions

# 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | : us1salx00259 |
| HARP Compound | : gsk1550188 |
| Study location | : gsk1550188\mid205646 |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for all reporting efforts. | |

# 15.5.2. Reporting Standards

### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

# **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DPs.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study treatment dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations)
     will be included in listings but omitted from figures, summaries and statistical analyses.

# **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables with the exception of certain summaries by year interval in which unscheduled visits may appear in the "anytime post baseline" category where specified e.g. worst laboratory toxicity grades.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Sta | Refer to IDSL Statistical Principals 7.01 to 7.13. |

# 15.6. Appendix 6: Derived and Transformed Data

### 15.6.1. General

# **Multiple Measurements at One Analysis Time Point**

- For continuous data, the mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- For continuous data, if there are two values within a time window (as per Section 15.3.1) the value
  closest to the target day for that window will be used. If values are the same distance from the target,
  then the scheduled assessment will be used, if both assessments are also unscheduled then the 1st
  assessment will be taken.
- For categorical data, if there are two values within a time window (as per Section 15.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the value prior to the target day will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables.

# Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

# **Study Completion**

- A participant is considered to have completed the study if he/she has completed all phases
  of the study, including the Week 104 Visit, as defined in the Schedule of Activities(SoA) (see
  Section 2 of the protocol)
- A participant is considered to have completed the double-blind treatment phase (Year 1) of the study if he/she has completed all 52 weeks of the double-blind treatment phase, including the Week 52 Visit, as defined in the SoA (see Section 2 of the protocol)
- Participants who discontinue study treatment and withdraw from the study up to Week 52
  are required to complete an Early Withdrawal Visit and a Follow-up Visit; the Early
  Withdrawal Visit is scheduled 1 to 4 weeks after the last dose of belimumab and the Followup Visit is scheduled 8 weeks after the last dose of belimumab
- Participants in Arms A or B who withdraw from the study after Week 52 are required to complete an Early Withdrawal Visit 1-4 weeks after withdrawal from the study.
- Participants in Arm C who discontinue study treatment and withdraw from the study after Week 52 are required to complete an Early Withdrawal Visit and a Follow-up Visit; the Early Withdrawal Visit is scheduled 1 to 4 weeks after the last dose of belimumab and the Followup Visit is scheduled 8 weeks after the last dose of belimumab

# Visit assessments completed late

In the event that a PGA, or SLE flare assessment, which may be only completed once labs have been returned to the site, is recorded later than the visit date, then an imputed date will be used. The imputed PGA / SLE flare assessment date will be the earliest date for a completed SLEDAl-2K (IBA or PI) assessment. This may be different than the earliest visit within that window. If there are no SLEDAl-2K assessment dates available then the visit date is used.

# 15.6.2. Study Population

# **Age Derivation**

Age on any specified day (e.g. screening, 1st dose etc.) will be derived as:

If the specified day is on or after the 30th June then:

Year of specific timepoint – DOB year

If the specified day is before the 30th June then:

(Year of specific timepoint – DOB year) -1

(Note this assumes day and month of birth is 30 June - as this information is not collected) Age at baseline will be defined as the latest of randomization date and baseline visit date, and derived as above.

# **Treatment Compliance – Belimumab**

• Percent compliance will be calculated based on the formula:

Percent Compliance = 100\* (Number of injections prescribed - Number of injections missed) / Number of injections prescribed

# **Extent of Exposure – Belimumab**

• Number of days of exposure to belimumab will be calculated based on the formula:

# Duration of Exposure in Days = Last injection date - First injection date + 7

- Only complete dates will be used when calculating duration of exposure. First and last injection dates will be used, regardless of any missed doses.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

# Extent of Exposure – Rituximab

- Dose intensity in mg will be calculated as the cumulative actual dose divided by 2.
- If the total volume of an infusion is not administered, the actual dose infused for that visit will be calculated as:

Actual Dose infused (mg) = Planned Dose (mg) \* Percentage of volume infused

# On Treatment Exposure (Year 1)

Number of days of On-Treatment exposure will be calculated based on the formula:

# **Duration of On-Treatment Exposure in Days**

- = Year 1 on-treatment end date (see Section 5.12) First Belimumab injection date + 1
- Only complete dates will be used when calculating duration of study exposure.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

# On-Study Exposure (Years 1&2 Combined)

• Number of days of On-Study exposure will be calculated based on the formula:

# On-Study Exposure (Years 1&2 Combined)

# Duration of On-Study Exposure in Days = Date of study completion or withdrawal – First Belimumab injection date + 1

- Only complete dates will be used when calculating duration of study exposure.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

# **Disease Duration**

When the start day is missing, impute with 01. When the start day and month is missing, impute with 01 January. This will impute the longest possible duration.

# 15.6.3. SLEDAI-2K Total and Organ System Domain

# SLEDAI-2K Total and Organ System Domain Scores

SLEDAI-2K assessments consist of 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each of 9 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease (marked 'No').

Organ system domain scores are the sum of the weights of items within the organ domain as defined in Table 9.

In this study, proteinuria is evaluated using spot-urine protein [represented as protein-creatinine ratio or PC Ratio in the laboratory dataset]. in lieu of the 24-hour urine collection, as evaluated by the investigator.

Table 9 SLEDAI-2K

| Organ System | Descriptor | Weight | |
|---|---|---|---|
| CNSa | | | nical Outcome Assessment data collection questionnaires or |
| | indices, which are p | protected by | third party copyright laws and therefore have been excluded. |



a. In the summaries and analyses of SLEDAI-2K organ systems, CVA will be moved from the CNS to the Vascular organ system and the Constitutional organ system will be eliminated and its one component, fever, will be moved to the hematologic organ system.

Adapted from the original source: [Gladman, 2002]. Used with permission from author (Murray Urowitz).

- Blinded independent assessors will conduct the SLEDAI-2K at key time points. The primary and major secondary efficacy endpoints will be conducted using the blinded independent assessors' SLEDAI-2K data
- For SLEDAI-2K after the Day 1 visit, the window is -10 days to + 7 days from the date of assessment post Day 1 visit, excluding the sample that was used in the previous visit assessment.

The SLEDAI-2K score is the sum of <u>all 24</u> individual items from the SLEDAI-2K.

# SLEDAI-2K missing values

SLEDAI-2K missing scores for laboratory parameters i.e.

Renal CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



Will be imputed from the previous assessment if the previous assessment is no more than 35days prior.

When it is not possible to calculate SLEDAI-2K score but it is still possible to ascertain that the SLEDAI-2K score is >0, >2, or >4, then this information will be used in the derivation of disease control, clinical remission, complete remission, and LLDAS.

Similarly, when it is possible to determine that the maximum possible value for the SLEDAI-2K, assuming the highest score for missing values is <=2 or <=4 then this will be used in the derivation of disease control nd LLDAS.

# **SLEDAI-2K Organ System Improvement and Worsening**

In the analysis of SLEDAI-2K organ system improvements and worsening, CVA will be moved from the CNS to the Vascular organ system and the Constitutional organ system will be eliminated and its one component, fever, will be moved to the hematologic organ system

# Clinical SLEDAI-2K Score (Excluding Serological Activity)

The clinical SLEDAI-2K score (Excluding Serological Activity assessments) is the sum of <u>22 of the 24</u> individual items from the SLEDAI-2K, excluding the following 2 items:



The scoring of the 22 questions is weighted in the same manner as the SLEDAI-2K, however the maximum theoretical score is now 101.

Note that the wording in the Protocol was "Serological activity score, i.e., anti-dsDNA positivity and/or hypocomplementemia, is excluded from the Clinical SLEDAI-2K endpoint". The endpoint has been clarified here by using the names of the two SLEDAI-2K item scores, however, this does not represent a change to the planned endpoint, just a clarification.

### Partial but informative SLEDAI-2K score

If after imputation for missing questions the SLEDAI-2K total score is still not derivable due to missing individual questions, then the minimum possible score will be considered (sum of the answered questions).

Similarly a maximum possible score (observed questions + maximum response for missing questions) will be considered.

### 15.6.4. Disease Control

# **Endpoint Definition**

The disease control endpoint is defined as:

• SLEDAI-2K score ≤2 (IBA\*),

- Not a Treatment failure
- Not a Study withdrawal

The same derivation will be applied to the secondary endpoint "Disease control (PI)" using the principal investigators assessment of the SLEDAI-2K.

# Imputation of Missing values - IBA assessment

Missing IBA assessments based on laboratory assessments i.e.:

Urinary Casts, Hematuria, Proteinuria, Pyuria, Low Complement, Increased DNA Binding, Thrombocytopenia, and Leukopenia

will be imputed from the PI assessment if the laboratory sample (for the PI assessment) was drawn no more than 35 days prior. An imputed assessment can not be used to impute another assessment.

There will be no imputation of missing IBA assessments based on physical examination

# Imputation of Missing values - PI assessment

If an individual question of the SLEDAI-2K assessment or the full assessment is missed the previous assessment may be used as a substitute if it was no more than 35 days prior. An imputed assessment cannot be used to impute another assessment.

### Partial but informative SLEDAI-2K score

If after imputation for missing questions the SLEDAI-2K total score is still not derivable due to missing individual questions, then the minimum possible score will be considered. If the minimum possible score is >2 then the subject will be considered as a non-responder. Similarly a maximum possible score will be considered to determine if the maximum possible score is <2.

### Time to Disease Control Sustained to Week 104

A subject has a sustained disease control at a visit if all of the following criteria are met:

- 1 In disease control at the visit
- 2 In disease control at the first visit that is at least 24 study weeks prior, or if disease control cannot be assessed at that visit, then in disease control at the visit prior.
- 3 In disease control for all assessed visits between (1) and (2). Note assessments can be missing.

Note: 24 weeks refers to the difference in visit 'labels' not calendar weeks between visits.

The first visit of sustained disease control is defined as the 1<sup>st</sup> visit that the subject is a disease control responder and all subsequent visits up to and including Week 104 the subjects is also a disease control responder. Missing assessments are not considered.

Time to disease control sustained to Week 104 =

1st visit of sustained disease control - treatment start date (Day 1) +1

# **Duration of Disease Control**

The duration of disease control is defined as the longest period between 2 visits that the subject is a disease control responder at all visits. Missing assessments are not considered.

Duration of disease control = longest period where

1st visit of disease control – last visit of disease control + 1

| Example<br>Subject | SLEDAI-2K score at Week<br>52 | Study Withdrawal<br>(including Lost to<br>Follow-up, or Death)<br>prior to Week 52 | Treatment<br>Failure prior to<br>Week 52 | IP Discontinuation prior to Week 52 | Main Estimand<br>(Hybrid) | Supportive<br>Estimand<br>(Composite) | (Hybrid On<br>Treatment) | Treatment<br>Policy |
|---|---|---|---|---|---|---|---|---|
| 1 | >2 | N | N | N | NR | NR | NR | NR |
| 2 | >2 | N | N | Υ | NR | NR | Excluded | NR |
| 3 | >2 | N | Υ | N | NR | NR | NR | NR |
| 4 | >2 | N | Y and prior to IP<br>discontinuation<br>Y but post IP | Υ | NR | NR | NR | NR |
| 5 | >2 | N | discontinuation | Υ | NR | NR | Excluded | NR |
| 6 | <=2 | N | N | N | R | R | R | R |
| 7 | <=2 | N | N | Υ | R | NR | Excluded | R |
| 8 | <=2 | N | Y<br>Y and prior to IP | N | NR | NR | NR | R |
| 9 | <=2 | N | discontinuation | Υ | NR | NR | NR | R |
| 10<br>11 | <=2 Incomplete* or entirely missing | N<br>N | Y but post IP discontinuation | Y | NR<br>NR | NR<br>NR | Excluded<br>NR | R<br>NR |
| | Incomplete* or entirely missing but not due to | | | | | | | |
| 12 | study withdrawal<br>Incomplete* or entirely<br>missing but not due to | N | N | Υ | NR | NR | Excluded | NR |
| 13 | study withdrawal Incomplete* or entirely | N | Y | N | NR | NR | NR | NR |
| 14 | missing but not<br>meaningful<br>Incomplete* or entirely | N | Y and prior to IP discontinuation | Υ | NR | NR | NR | NR |
| 15 | missing but not due to study withdrawal | N | Y but post IP discontinuation | Υ | NR | NR | Excluded | NR |
| 16 | Missing - does not exist due to study withdrawal | Y and at the same time as IP discontinuation | N | Υ | NR | NR | NR | NR |

| Example<br>Subject | SLEDAI-2K score at Week<br>52 | Study Withdrawal<br>(including Lost to<br>Follow-up, or Death)<br>prior to Week 52 | Treatment<br>Failure prior to<br>Week 52 | IP Discontinuation prior to Week 52 | Main Estimand<br>(Hybrid) | Supportive<br>Estimand<br>(Composite) | (Hybrid On<br>Treatment) | Treatment<br>Policy |
|---|---|---|---|---|---|---|---|---|
| 17 | Missing - does not exist due to study withdrawal | Y but post IP discontinuation | N | Υ | NR | NR | Excluded | NR |
| 18 | Missing - does not exist due to study withdrawal | Y and at the same time as IP discontinuation | Y and prior to IP discontinuation | Υ | NR | NR | NR | NR |
| 19 | Missing - does not exist due to study withdrawal | Y but post IP discontinuation | Y and prior to IP discontinuation | Υ | NR | NR | NR | NR |
| 20 | Missing - does not exist due to study withdrawal | Y but post IP discontinuation | Y but post IP discontinuation | Υ | NR | NR | Excluded | NR |

# R = Responder; NR = Non-Responder

<sup>\*</sup>Incomplete: does not include partial scores where it is possible to determine that the total score must be >2, or that the maximum possible score (assuming worst case for missing data) is <=2

### 15.6.5. Clinical Remission

# **Endpoint Definition**

Clinical remission for Arms A & B (secondary endpoint) is defined as:

- Clinical SLEDAI-2K score<sup>#</sup> = 0 (IBA\*),
- Not a Treatment Failure
- Did not withdraw from the study
- 7-day average corticosteroids at a prednisone equivalent dose of 0mg/day for the assessment (7 day average is the average of current and 6 previous days)

The same derivation will be applied to the secondary endpoint "clinical remission (PI)" using the principal investigators assessment of the SLEDAI-2K.

# Imputation of Missing values - IBA assessment

Missing IBA assessments based on laboratory assessments i.e.:

Urinary Casts, Hematuria, Proteinuria, Pyuria, Thrombocytopenia, and Leukopenia will be imputed from the PI assessment if the laboratory sample (for the PI assessment) was drawn no more than 35 days prior. An imputed assessment can not be used to impute another assessment.

There will be no imputation of missing IBA assessments based on physical examination

# Imputation of Missing values - PI assessment

If an individual question of the SLEDAI-2K assessment or the full assessment is missed the previous assessment may be used as a substitute if it was no more than 35 days prior. An imputed assessment cannot be used to impute another assessment.

# Partial but informative Clinical SLEDAI-2K score

If after imputation for missing questions the Clinical SLEDAI-2K score is still not derivable due to missing individual questions, then the minimum possible score will be considered (sum of the answered questions). If the minimum possible score is >0 then the subject will be considered as an observed non-responder (rather than non-responder due to missing data).

# Clinical Remission Sustained For At Least 24 Weeks

Sustained response will be reported for all weeks post Week 52 (Year 2), and at any timepoint (i.e. any subjects who had a sustained response at any time during Year 2). Statistical analysis will only be conducted at Week 104 and at 'any timepoint'.

A subject has a sustained remission at a visit if all of the following criteria are met:

- 1 In clinical remission at the visit
- 2 In clinical remission at the first visit at least 24 study weeks prior, or if clinical remission cannot be assessed at that visit, then in clinical remission at the visit prior.
- 3 In clinical remission for all assessed visits between (1) and (2). Note assessments can be missing.

Note: 24 weeks refers to the difference in visit 'labels' not calendar weeks between visits.

<sup>\*</sup>See Section 15.6.3

<sup>\*</sup>at baseline the principal investigators assessment will be used

### Time to Clinical Remission Sustained to Week 104

The first visit of sustained clinical remission is defined as the 1<sup>st</sup> visit that the subject is a clinical remission responder and all subsequent visits up to and including Week 104 the subjects is also a clinical remission responder. Missing assessments are not considered (the rules for sustained response for at least 24 weeks as defined above are also applied here).

Time to clinical remission sustained to Week 104 =

1st visit of sustained clinical remission - treatment start date (Day 1) +1

# **Duration of Clinical Remission**

The duration of clinical remission is defined as the longest period between 2 visits that the subject is a clinical remission responder at all visits. Missing assessments are not considered Duration of clinical remission = longest period where

1st visit of clinical remission – last visit of clinical remission + 1

# 15.6.6. Complete Remission

# **Endpoint Definition**

Complete remission for Arms A & B (secondary endpoint) is defined as:

- SLEDAI-2K score = 0 (IBA\*),
- Not a Treatment Failure (specific to Arms A&B)
- Did not withdraw from the study
- 7-day average corticosteroids at a prednisone equivalent dose of 0mg/day for the assessment (7 day average is the average of current and 6 previous days)

Complete remission for Arm C (the exploratory endpoint) is defined as:

- SLEDAI-2K score = 0 (IBA\*),
- Not a Treatment Failure (specific to Arm C)
- Did not withdraw from the study
- 7-day average corticosteroids at a prednisone equivalent dose of 0mg/day for the assessment (7 day average is the average of current and 6 previous days)

\*at baseline the principal investigators assessment will be used

Note some tables will contain the endpoint using these 2 different definitions in the same table.

# Imputation of Missing values - IBA assessment

Missing IBA assessments based on laboratory assessments i.e.:

Urinary Casts, Hematuria, Proteinuria, Pyuria, Low Complement, Increased DNA Binding, Thrombocytopenia, and Leukopenia

will be imputed from the PI assessment if the laboratory sample (for the PI assessment) was drawn no more than 35 days prior. An imputed assessment can not be used to impute another assessment.

There will be no imputation of missing IBA assessments based on physical examination

# Imputation of Missing values - PI assessment

If an individual question of the SLEDAI-2K assessment or the full assessment is missed the previous assessment may be used as a substitute if it was no more that 35 days prior. An imputed assessment cannot be used to impute another assessment.

# Partial but informative SLEDAI-2K score

If after imputation for missing questions the SLEDAI-2K total score is still not derivable due to missing individual questions, then the minimum possible score will be considered (sum of the answered questions). If the minimum possible score is >0 then the subject will be considered as an observed non-responder (rather than non-responder due to missing data).

# Complete Remission Sustained For At Least 24 Weeks

Sustained response will be reported for all weeks post Week 52 (Year 2), and at any timepoint (i.e. any subjects who had a sustained response at any time during Year 2). Statistical analysis will only be conducted at Week 104 and at 'any timepoint'.

A subject has a sustained remission at a visit if all of the following criteria are met:

- 1 In complete remission at the visit
- 2 In complete remission at the first visit at least 24 study weeks prior, or if complete remission cannot be assessed at that visit, then in clinical remission the visit prior.
- 3 In complete remission for all assessed visits between (1) and (2). Note assessment can be missing.

Note: 24 weeks refers to the difference in visit 'labels' not calendar weeks between visits.

# 15.6.7. SFI FLARE INDEX

# SLEDAI-2K Flare Index (Adapted from Buyon, 2005; Petri, 2005; Neergard, 2006. Petri, 1999) Mild-moderate flare Severe flare FCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



 The modified SLE Flare index excludes severe flares that are triggered only by an increase is SLEDAI-2K Score to greater than 12.

The following scoring rules are based on the SLEDAI-2K flare index:

- SFI reports the first mild /moderate or severe flare occurrence since the last non-missing assessment.
- The SLEDAI-2K criteria will be assessed programmatically (based on the PI assessment at the visit that the flare was reported) to determine if the SLEDAI-2K criteria for a flare has been met and used for the assessment of flare, irrespective of what was recorded on the SFI form.
- Although there are boxes on the form for the investigator to classify the most recent flare to mild/moderate or severe, the classification will be re-derived from the subcategory scores. Flares originally marked severe will be downgraded to "Not Severe" if the only reason marked is a change in SLEDAI-2K score to >12.
  - In this case, if any of the mild/moderate reasons are checked or if the SLEDAI-2K score has a change from the last non-missing assessment of at least 3, then the flare will be considered mild/moderate. Otherwise this not a flare

The last non-missing assessment is the last previous visit were SLE flare was assessed (and is not entirely missing).

# Partial but informative SLEDAI-2K score

If after imputation for missing questions the SLEDAI-2K total score is still not derivable due to missing individual questions, then the minimum possible score will be considered (sum of the answered questions). Similarly a maximum possible score (sum of observed questions + maximum response for missing questions) will be considered. If from these scores it is possible to determine that there has be an increase in score from the previous visit of at least 3 then this will be used as indication of a mild/moderate flare. However if it is not possible to determine whether there has been a change of at least 3 from the previous assessment then no assumption will be made about the presence of a mild/moderate flare.

# 15.6.8. Physicians Global Assessment (PGA) Scoring

# Physicians Global Assessment (PGA) Scoring

PGA is collected on a 10cm visual analogue scale (VAS). However, the standard scoring range for the PGA is 0 to 3, therefore the score will be rescaled for reporting by multiplying the collected score by 3/10.

# 15.6.9. Lupus Low Disease Activity State (LLDAS)

| Endpoint Definition | | |
|---|---|---|
| Criteria | Source data and derivation | Rationale |
| SLEDAI-2K ≤4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity; | SLEDAI – 2K score as assessed by the principal investigator Individual stated organ systems must have a score of 0, Note: Cardiopulmonary = Cardiovascular & respiratory organ system Vasculitis = Vascular organ system Fever = Constitutional organ system Data on hemolytic anemia and | |
| no new features of lupus disease activity compared with the previous assessment; | gastrointestinal activity are not available and is not considered in evaluating this criterion but assumed to be captured in the PGA item. No worsening of any of the item scores of the SLEDAI–2K (principal investigator assessment) score compared to the previous assessment | Compared to previous visit to reflect a stable disease state. |
| PGA (scale 0-3) ≤1; | PGA as reported (closest assessment to the target date that is within the visit window) | |
| current prednisolone<br>(or equivalent) dose<br>≤7.5 mg daily; | 7 day average prednisone dose (day of visit and 6 prior days) assessed on the day of the SLEDAI-2k assessment | 7 Day average due<br>to the planned<br>tapering, as subjects<br>may be on a dosing<br>regimen that varies<br>by day (e.g. 1mg<br>every other day) |
| well tolerated standard<br>maintenance doses of | The dose on the <u>day of</u> the SLEDAI-<br>2K assessment must not exceed: | The protocol stated 'equivalent' |

# **Endpoint Definition** medications to those immunosuppressive azathioprine: 300mg/day drugs and approved stated in . [Oon. methotrexate 25mg/week • biological agents. 2019] supplement leflunomide 40mg/day excluding Mycophenolate On the day of investigational drugs sodium < 2.88 g/day assessment as Mycophenolate mofetil≤4g/day identified in the publications cyclophosphamide < 2.5 mg/kg/day 6-mercaptopurine <= 300mg/day Cyclosporine<=4mg/kg/day Tacrolimus <= 0.2 mg/kg/day Sirolimus<=2mg/day Thalidomide <= 200 mg/day mizoribine<=150mg/day Not to be taken within 28 days prior to the assessment: Intravenous Cyclophosphamide Other investigation agent Anti-TNF therapy (adalimumab, etanercept, infliximab) Other biologics (abatacept, anakinra) **IVIG** Plasmapheresis Topical treatments will not be considered Not Study withdrawal Did not withdraw or (including death and discontinue for any lost to follow-up reason

# SLEDAI-2K Component: Imputation of Missing values - PI assessment

If an individual question of the SLEDAI-2K assessment or the full assessment is missed the previous assessment may be used as a substitute if it was no more than 35 days prior. An imputed assessment can not be used to impute another assessment.

# SLEDAI-2K Component: Partial but informative SLEDAI-2K score

If after imputation for missing questions the SLEDAI-2K total score is still not derivable due to missing individual questions, then the minimum possible score will be considered (sum of the answered questions). If the minimum possible score is >4 then the subject will be considered as a non-responder.
#### SLEDAI-2K Component: Imputation of Missing values – PI assessment

Similarly a maximum possible score (observed questions + maximum response for missing questions) will be considered to determine if the maximum possible score is  $\leq 4$ .

### 15.6.10. Lupus QOL Scale

The LupusQoL consists of 34 items in eight domains. The number of items in each domain and the item numbers that refer to that domain are tabulated below:



The LupusQoL has a five-point Likert response scale for each item and are scored as:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Each domain of the LupusQoL is scored separately as:

Calculate the mean raw domain score by adding up the item response scores for the domain and then divide by the number of items answered in that domain. Mean raw domain scores can only be obtained when at least 50% of the items for the domain are answered. A non-applicable response is treated as unanswered.

Transform the mean raw domain score by dividing by four (the number of Likert responses [five] minus one) and then multiplying by 100, as below:

#### Mean raw domain score x 25 = Transformed score for domain

Transformed scores range from  $0^{\circ}$  or  $0^{\circ}$  to  $100^{\circ}$ 

#### 15.6.11. Work Productivity and Activity Impairment (WPAI)

The WPAI consists of 6 questions

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



The following summary measures will be derived:



If a question is missing all summary measures that use that question will not be derived.

Only the 'Percent overall work impairment due to Lupus' and 'Percent activity impairment due to Lupus' are summarised in the tables.

### 15.6.12. Functional Assessment of Chronic Illness Therapy (FACIT)

The FACIT – Fatigue scale consists of 13 questions:



Each Question is answered on a Likert response scale and scored as numbered:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

The total score is the sum of the responses (inverted for reversed items) multiplied by 13, then divided by the number of questions answered i.e.

$$\frac{\{(4-HI7)+(4-HI12)+(4-An1)+(4-An2)+(4-An3)+(4-An4)+An5+An7+(4-An8)+(4-An12)+(4-An14)+(4-An15)+(4-An16)\}*13}{Number\ of\ questions\ answered}$$

The total score will only be derived if at least 11 questions (80%) of the scale is completed.

# 15.6.13. Disease Control Without Current Immunosuppressant and with Current Corticosteroids ≤ 5mg/day

#### **Disease Control**

Disease control for Arms A & B (the primary endpoint) is defined as:

- SLEDAI-2K score ≤2 (IBA\*),
- Without immunosuppressants on the day of the assessment and 55 days prior to the assessment.
- 7-day average corticosteroids at a prednisone equivalent dose of ≤5mg/day for the assessment (7 day average is the average of current and 6 previous days)
- Without study withdrawal

Disease control for Arms C (the exploratory endpoint) is defined as:

- SLEDAI-2K score ≤2 (IBA\*),
- Without any new immunosuppressants, and not greater than the maximum of baseline (Day 1) day and Week 12 visit dose on the day of the assessment and 55 days prior to the assessment,
- 7-day average corticosteroids at a prednisone equivalent dose of ≤5mg/day for the assessment (7 day average is the average of current and 6 previous days)
- Without study withdrawal

Note some tables will contain the endpoint using these 2 different definitions in the same table.

The same derivation will be applied to the secondary endpoint "disease control (PI)" using the principal investigators assessment of the SLEDAI-2K.

#### 15.6.14. Prednisone Equivalent Conversion

- A concomitant medication is identified as a steroid if at least one associated ATC code (ATCCD1 ATCCD6) begins with 'H02.' Mineralocorticords are included in the group of ATC codes beginning with 'H02' but do not have sufficient anti-inflammatory properties to be considered as a prednisone equivalent. For this reason, the conversion factor has been set to 0.
- The following routes are considered to provide systemic exposure: oral, buccal, parenteral subcutaneous, intramuscular, intradermal, and intravenous. Although not systemic, intra-articular steroids are also identified for treatment failure rules. Topical routes of administration are excluded (e.g., topical, conjunctival, intranasal).
- At data base release, all preferred terms identified with an ATC code beginning with 'H02' will be reviewed to ensure a conversion factor exists for all terms with a systemic route of administration.
- Similarly, all routes of administration for preferred terms with an ATC code beginning with 'H02' will be reviewed to ensure all systemic routes have been identified in the list below.

<sup>\*</sup>at baseline the principal investigators assessment will be used

- In order to be converted the frequency and dose of the steroid must be present with the unit dose in milligrams (mg) or grams (g). Doses recorded in grams will be converted to milligrams by multiplying the dose in grams by 1000 prior to applying the conversion factor.
- Reported dose for systemic steroid is converted to prednisone equivalent dose using conversion factor for each particular medication (refer to online calculator http://www.globalrph.com/corticocalc.htm).

Prednisone Equivalent = Collected X Conversion x Frequency
Daily Dose (mg) Dose (mg) Factor Factor

| Prednisone Conversion Factors (mg) | |
|-------------------------------------|---------------------------------------|
| Treamsone conversion ractors (mg) | Conversion factor for converting to a |
| Preferred term | prednisone-equivalent dose |
| BETAMETHASONE | 8.3333` |
| BETAMETHASONE DIPROPIONATE | 8.3333` |
| BETAMETHASONE SODIUM PHOSPHATE | 8.3333` |
| BETROSPAM | 8.3333` |
| BUDESONIDE | 0.3333` |
| CORTISONE | 0.2 |
| CORTISONE ACETATE | 0.2 |
| CRONOLEVEL | 8.3333` |
| DEFLAZACORT | 0.8333` |
| DEXAMETHASONE | 6.6666` |
| DEXAMETHASONE ACETATE | 6.6666` |
| DEXAMETHASONE SODIUM PHOSPHATE | 6.6666` |
| FLUDROCORTISONE | 0 |
| FLUOCORTOLONE | 3 |
| HYDROCORTISONE | 0.25 |
| HYDROCORTISONE ACETATE | 0.25 |
| HYDROCORTISONE SODIUM SUCCINATE | 0.25 |
| MEPREDNISONE | 1.25 |
| METHYLPREDNISOLONE | 1.25 |
| METHYLPREDNISOLONE ACETATE | 1.25 |
| METHYLPREDNISOLONE SODIUM SUCCINATE | 1.25 |
| PARAMETHASONE | 2.5 |
| PREDNISOLONE | 1 |
| PREDNISOLONE ACETATE | 1 |
| PREDNISOLONE SODIUM PHOSPHATE | 1 |
| PREDNISOLONE SODIUM SUCCINATE | 1 |
| PREDNISONE | 1 |
| PREDNISONE ACETATE | 1 |
| TRIAMCINOLONE | 1.25 |
| TRIAMCINOLONE ACETATE | 1.25 |

| Prednisone Conversion Factors (mg) | |
|---|---|
| Preferred term | Conversion factor for converting to a prednisone-equivalent dose |
| TRIAMCINOLONE ACETONIDE | 1.25 |

| Combination Products: Prednisone Conversion Factors (mg) | | |
|---|---|---|
| Preferred term | Ingredients | Conversion factor for converting to a prednisone-equivalent dose |
| CELESTONA BIFAS | Betamethasone acetate + | 8.3333` |
| | Betamethasone sodium phosphate | |
| DEPO-MEDROL MED<br>LIDOKAIN | Methylprednisolone + Lidocaine | 1.25 |
| CELESTAMINE | Betamethasone + | 8.3333` |
| | Dexchlorpheniramine maleate | |
| SYNBETAMINE | Betamethasone + | 8.3333` |
| | Dexchlorpheniramine maleate | |

| Frequency Factors | |
|-------------------|--------|
| Frequency | Factor |
| BID | 2 |
| BIW | 2/7 |
| HS | 1 |
| OAM | 1/30 |
| Once | 1 |
| PRN | Null |
| Q2H | 12 |
| Q2W | 1/14 |
| Q3H | 8 |
| Q3MO | 1/84 |
| Q3w | 1/21 |
| Q4H | 6 |
| Q4W | 1/28 |
| Q6H | 4 |
| Q8H | 3 |
| QAM | 1 |
| QD | 1 |
| QH | 24 |
| QHS | 1 |
| QID | 4 |
| QOD | 1/2 |
| QPM | 1 |

| Frequency Factors | | |
|-------------------|--------|---|
| Frequency | Factor | |
| QW | 1/7 | |
| QWK | 1/7 | |
| TID | 3 | |
| TIW | 3/7 | |
| UNK | Null | |
| 2 TIMES PER WEEK | 2/7 | |
| 3 TIMES PER WEEK | 3/7 | |
| EVERY 2 WEEKS | 1/14 | |
| EVERY 3 WEEKS | 1/21 | |
| EVERY 4 Weeks | 1/28 | |
| EVERY WEEK | 1/7 | · |

### 15.6.15. Treatment Failure Rules During Study Conduct

A treatment failure is defined as any subject who receives a protocol-prohibited medication or a dose of allowable (but protocol restricted) medication that results in treatment failure designation prior to the analysis visit of interest (e.g. Week 52, Week 64, Week 104).

The treatment failure rules are detailed in the protocol Section 7.7.

15.6.15.1. Summary

| Occurrence | Post Study Start Treatments | TX<br>Failure:<br>Arms A/B | TX<br>Failure:<br>Arm C |
|---|---|---|---|
| After Day 1 | <ul> <li>NEW anti-malarial medication for<br/>SLE (other than for anti-malarial<br/>prophylaxis)</li> <li>NEW immunosuppressant<br/>medication</li> <li>Prohibited Medications and Non-<br/>Drug therapies</li> </ul> | Yes | Yes |
| After Week 4 | Immunosuppressant medication | Yes | No |
| After Week 12 | Immunosuppressant medication dose<br>increased over baseline (Day 1) or<br>Week 12 visit dose, whichever is<br>higher | Not<br>Applicable | Yes |
| Week 27<br>onwards | • Corticosteroid (Prednisone equivalent) dose >5mg/day (Average day of assessment and 6 prior days) | Yes | Yes |

| Occurrence | Post Study Start Treatments | TX<br>Failure:<br>Arms A/B | TX<br>Failure:<br>Arm C |
|---|---|---|---|
| After Week 26 | • High Dose CS for Non-SLE use (Maximum use 7 days, taper [≤5 mg/day]. 21 days) | Yes | Yes |
| After Week 44 | Aspirin doses >1000 mg days if<br>never received such doses between<br>Day 1 and Week 44<br>(Note: It does Not apply if given <7<br>days) | Yes | Yes |
| Weeks 44 to 52* | <ul> <li>NSAIDs (dose above Day 1 or the visit day starting the 8 weeks interval for ≥7 days)</li> <li>Intraarticular CS injections</li> <li>High Dose CS for Non-SLE use</li> </ul> | Yes | Yes |
| After Week 52 | IP – Belimumab SC | Yes | No |
| Weeks 56 to 64* | <ul> <li>NSAIDs (dose above Day 1 or the visit day starting the 8 weeks interval for ≥7 days)</li> <li>Intraarticular CS injection</li> <li>High Dose CS for Non-SLE use</li> </ul> | Yes | Yes |
| Weeks 96 to 104* | <ul> <li>NSAIDs (dose above Day 1 or the visit day starting the 8 weeks interval for ≥7 days)</li> <li>Intraarticular CS injections</li> <li>High Dose CS for Non-SLE use</li> </ul> | Yes | Yes |

<sup>\*8</sup> weeks prior to major efficacy assessments (Primary endpoint [Week 52] and major secondary endpoints [Weeks 64, 104]).

### 15.6.15.2. SLE Medication Categories

| Medication Category | Rule |
|---|---|
| Anti-malarials | Set to "ANTIMALARIALS" if the preferred term begins with "QUINACRINE", |
| | "QUININE", "HYDROXYCHLOROQUINE", |
| | "MEPACRINE", or "CHLOROQUINE" |
| | AND |
| | the route of administration is not 'TOPICAL', 'VAGINAL', 'CONJUNCTIVAL', |
| | 'INTRANASAL', 'INHALATION', 'INTRA-OCULAR', 'INTRATRACHEAL', |
| | 'EPIDURAL', 'INTRA-ARTICULAR', or 'OTHER'. |
| Steroids | Set to 'STEROIDS' if at least one associated ATC code (ATCCD1 – |
| | ATCCD6) begins with 'H02' |
| | AND |
| | Route of administration is |
| | "INTRADERMAL", "INTRAMUSCULAR", "BUCCAL", "PARENTERAL" |
| | "INTRAVENOUS", "ORAL", "SUBCUTANEOUS", or "INTRA-ARTICULAR". |

| Medication Category | Rule |
|---|---|
| Immunosuppressants | Set to 'IMMUNOSUPPRESSANTS' if at least one associated ATC code (ATCCD1 – ATCCD6) begins with 'L04A' or the preferred term begins with "CYCLOPHOSPHAMIDE" (oral and parenteral routes) or "MERCAPTOPURINE" (oral route) AND route of administration is not "TOPICAL" or "OPHTHAMLIC" AND not classified above as "ANTIMALARIALS". |
| NSAIDs | Set to NSAIDs if at least one associated ATC code (ATCCD1 – ATCCD6) begins with 'M01A'.Glucosamine and Chondroitin not considered NSAIDs |
| Aspirin | Set to "ASPIRIN" if CMDECOD contains "ACETYLSALICYLIC ACID" or "ACETYLSALICYLATE LYSINE". |
| Prohibited | Set to "PROHIBITED" if at least one associated ATC code (ATCCD1 – ATCCD6) begins with 'L04AB' or 'V98' or if any of the following conditions are met, if CMDECOD equals ," BELIMUMAB", "ADALIMUMAB", "ETANERCEPT", "INFLIXIMAB", "CERTOLIZUMAB", "TOCILIZUMAB", "GOLIMUMAB", "RITUXIMAB", "ABATACEPT", "ANAKINRA", "CANAKINUMAB", "USTEKINUMAB", "BRODALUMAB", "SECUKINUMAB", "IXEKIZUMAB", "EPRATUZUMAB", "TABALUMAB", "ATACICEPT", "IMMUNOGLOBULIN" (IV route), "CYCLOPHOSPHAMIDE" (IV route), or "PLASMAPHERESIS" |

#### 15.6.15.3. General Conventions

- Assessment of dose is based on analysis dose. Analysis dose is daily dose adjusted
  for dosing frequency, and in the case of steroid is converted to prednisone
  equivalents. Exception is intra-articular dose where analysis dose is not populated.
- In the event there are multiple visit dates within a visit window, the date for determining treatment failure, will be the earliest date at which efficacy data (from SLEDAI-2K (IBA), SLEDAI-2K (PI), PGA, and SLE Flare) is recorded. This may be different than the earliest visit within that window.
- If a critical visit (Week 52, 64, and 104], is missing from efficacy data (from SLEDAI-2K (IBA and PI), PGA, SLE Flare, LLDAS) then the date is imputed as the target day for that visit.
- Actual visit date, not target visit date, is used to assess treatment failures.
  - If the subject's Day 169 (Week 24) study visit occurs on Day 171, the date for Day 171 is used when applying the treatment failure rules.
- Prohibited medications/dosages started on the date of early withdrawal are considered a TF (see clarification below for steroids). If the prohibited medication/dose starts after the date of withdrawal it will not be part of the TF assessment.

- All potential TF rule violation are output programmatically and all adjudicated.
- Clinical may amend the date of TF during adjudication if, for instance, a subject did not meet the criterion on the date identified by the program but did meet it later.

#### 15.6.15.4. Steroids

- SLE-related steroids are steroids where medication type is marked as 'Systemic Lupus Erythematosus (SLE)' (CMTYPCD=156), regardless of reason for medication (CMREAS).
- Total steroids include steroids for SLE and non-SLE reasons.
- Baseline dose is the 7-day average based on the 7 days **prior** to, but not including, treatment start date.
- The average steroid dose on any post baseline day is the sum of the steroids on that day and the prior 6 days divided by 7, so long as all days are post the baseline visit.
- The first day that the TF rule
  - Received a prednisone equivalent corticosteroid 7-day average dose of >5 mg/day after Week 26 visit

is applied will be when all values used in the average steroid dose are after Week 26 visit (not including the week 26 visit day) i.e. 7 days after Week 26 visit

- The final week interval for subjects who complete Week 104 will be 7 days prior to the exit visit date; [exit visit -7 days]. to [exit visit -1 day]. The day of Week 104 visit will not be included.
- The final interval for subjects who withdraw early will be the 7 days up to and including the exit visit date; [exit visit/early withdrawal date -6]. to [exit visit/early withdrawal date]. The day of withdrawal will be included.
- The above rules may miss a subject who starts/increases a steroid close to the day of withdrawal. In this situation it is possible that the subject may have withdrawn prior to the end of the interval for computing their 7-day average exceeding the TF threshold. Hence all subjects whose dose of steroid increased within 7 days (including day of withdrawal) of withdrawal, and have not already crossed the dose threshold for TF based on the 7-day average rule, will be output for clinical adjudication. If clinical adjudication determines these to be treatment failures the date of treatment failure will be set to the date of withdrawal.
- A subject who is receiving 0mg of steroid at baseline will be allowed to take ≤5mg of steroid post baseline without being considered a treatment failure.
- Intra-articular steroids are not included in average steroid dose calculations.
- Subjects with more than one dosing regimen that involves alternate day dosing will be reviewed to ensure the daily dose is calculated correctly.
- The 7 day average steroid >5mg/day rule will include SLE and non-SLE steroids in the identification of potential treatment failures. Treatment failure review will

exclude cases where the 7 day average steroids is >5mg/day due non-SLE steroids on a by subject review basis.

#### Intra-articular (IA) injections

• Participants may receive intraarticular injections during the study with the exception of within 8 weeks prior to the key efficacy endpoints (i.e. Week 52, 64, and 104). A participant who receives any intraarticular injection(s) within 8 weeks before to the Weeks 52, 64, and/or 104 visits will be defined as a treatment failure.

### Corticosteroids for Reasons Other Than SLE Disease Activity

Corticosteroids for non-SLE reasons (e.g., asthma, contact dermatitis, etc) may be given short-term at higher doses than <=5 mg/day according to the following guidelines:

- Up to 750 mg (prednisone) for 1 day, and/or
- Up to 60 mg/day (prednisone) for 2-3 days, and/or
- Up to 40 mg/day (prednisone) for 4-7 days.

After Week 26, the duration of high dose corticosteroids use for reasons other than SLE must not exceed 7 days, after which time, tapering should begin. The total corticosteroid dose must be tapered to <=5 mg/day within 21 days of the 1st dose of a course of high dose corticosteroids given for non-SLE reasons. In addition, no new high dose corticosteroids for reasons other than SLE are allowed that result in an average corticosteroid dose of >5 mg/day during the intervals starting 8 weeks before the key efficacy visits at Weeks 52, 64, and 104. During the intervals of 8 weeks before these efficacy endpoints, any new high dose corticosteroid use will declare the participant as a treatment failure. The day of the Week 44, 56, and 96 visits will count as the start of these 3 intervals (imputed visit date will be used for Week 56).

**NOTE:** Inhaled and topical corticosteroids are allowed throughout the course of the study

#### 15.6.15.5. Anti-malarials

Dose of anti-malarial at baseline is the dose the subject received on the treatment start date (Day 1). If a patient is receiving an anti-malarial at baseline it will be assumed that the dose is stable and not a loading dose.

Anti-malarial therapies may be continued, or dose adjusted during the study.

For non-SLE reasons (e.g., for the experimental treatment of COVID-19) an anti-malarial may be initiated for a subject not previously on an anti-malarial, or dose increased above

the common allowable maximum doses (defined below) according to the following guidelines, for short-term treatment:

- < 21 days treatment duration
- Not during the intervals within 8 weeks before the key efficacy visits (actual visit date) at Weeks 52, 64, and 104.

An anti-malarial may be replaced by another anti-malarial due to documented toxicity or lack of availability at any time during the study.

Clinical loading dose is permitted for initiation or replacement. Whether or not the dose was a loading dose will be assessed by clinical adjudication.

The common allowable maximum doses of anti-malarial drugs are:

- Hydroxychloroquine 400 mg/day
- Chloroquine 500 mg/day
- Quinacrine 100 mg/day

For compounded anti-malarials, no individual component may exceed the maximum dose above.

NOTE: The use of anti-malarials for anti-malarial prophylaxis is permitted.

#### 15.6.15.6. Other Immunosuppressant Agents

#### Arms A, B, and C

- Starting any new immunosuppressant agent after Day 1 for increased lupus
  disease activity will cause the participant to be declared a treatment failure. An
  immunosuppressant agent may however be replaced with one of the agents listed
  below due to documented toxicity or lack of availability. Replacement to be
  determined by clinical review
- New topical immunosuppressive agents (e.g., eye drops, topical creams) are allowed after Day 1.

#### Arms A and B

- Participants can maintain their baseline stable immunosuppressant regimen or adjust their dose as clinically required, up to the Week 4.
- At or prior to the Week 4 visit, immunosuppressants will be discontinued.
- All immunosuppressant medications post Week 4 (day after the visit 4 visit date) will be clinically reviewed to determine if they are a treatment failure.

#### Arms C

- Participants may continue their baseline immunosuppressant agents throughout the study.
- Dosage of existing immunosuppressant agents may be increased as clinically necessary until Week 12. From the day after the Week 12 visit, any increase in dose over the baseline (Day 1) or Week 12 visit dose, whichever is higher, will cause the participant to be declared a treatment failure.

The common allowable maximum doses for immunosuppressant agents at baseline (Day 1) and during the study (pre Week 4 for Arms and B) are listed below:

- Azathioprine 300 mg/day
- 6-mercaptopurine 300 mg/day
- Mycophenolate mofetil (PO)/ mycophenolate mofetil hydrochloride (IV) 4 g/day
- Mycophenolate sodium (PO) 2.88 g/day
- Methotrexate 25 mg/week
- Oral cyclophosphamide 2.5 mg/kg/day
- Cyclosporine 4 mg/kg/day\*
- Tacrolimus 0.2 mg/kg/day\*
- Sirolimus 2 mg/day\*
- Thalidomide 200 mg/day
- Leflunomide 40 mg/day\*
- Mizoribine 150 mg/day
- Other immunosuppressant agents not listed above, the investigator must contact the Medical Monitor for approval

# 15.6.15.7. Nonsteroidal Anti-inflammatory Drugs (NSAIDs), Aspirin, and Acetominophen

NSAIDs and aspirin should be initiated and stabilized prior to entry into the trial.

Baseline is defined as the NSAID/Aspirin received on the treatment start date (Day 1)

NSAIDs may be continued and dose adjusted as clinically indicated until 8 weeks before efficacy visits, i.e., Weeks 52, 64, and 104. During the intervals of 8 weeks before these efficacy endpoints, any increase in the NSAID dose above the dose at Day 1 or the visit day starting the interval of 8 weeks prior to these key efficacy visits, whichever is higher, will declare the participant as a treatment failure unless the NSAID is given for <7 days. The day of the Week 44, 56, and 96 visits will count as the start of these 3 intervals.

An NSAID may be replaced with another NSAID due to documented toxicity or lack of availability. Replacement due to toxicity/ lack of availability will be assessed during clinical adjudication.

New NSAIDs may not be added after Day 1 unless given for <7 days. Initiation of an NSAID after Day 1 that is given >=7 days will declare the participant as a treatment failure.

NSAIDS with an administration route of 'TOPICAL' or 'CONJUNCTIVAL'' will not be considered as TF's.

Aspirin will not be considered in the NSAID TF rules.

<sup>\*</sup>Clinical loading dose is permitted when replacing immunosuppressant agents.

Daily doses of aspirin up to 1000 mg/day are allowed at any time during the study. Daily doses of aspirin above 1000 mg/day may be initiated at any time up to the Week 44 visit and may continue through the end of the study. For participants who never received an aspirin regimen at a dose >1000 mg/day between the Day 1 and Week 44 visit, starting a new aspirin regimen at a dose >1000 mg/day after the Week 44 visit will declare the participant a treatment failure unless the aspirin is given for <7 days.

Daily doses of aspirin above 1000 mg/day may not be initiated in the 8 weeks before Week 64 and 104. The same rules as at Week 44 will be applied at Weeks 56 and 96

ACETYLSALICYLATE LYSINE (in mg) will be converted to standardised dose by multiplying by 0.556.

Acetaminophen (paracetamol) is primarily an analgesic and lacks the anti-inflammatory properties of other NSAIDs. The use of acetaminophen is recommended when possible to treat non-SLE related conditions, in the absence of a pre-existing hepatic function deficiency.

PRN use of NSAIDs or Aspirin will be identified as a potential TF and reviewed on a by subject review basis.

#### 15.6.15.8. Prohibited Medications

Medications prohibited by the protocol specified rule of:

- Other investigational agents (biologic or non-biologic). Investigational applies to any drug not approved for sale in the country in which it is being used.
- Co-enrollment into another study of a different investigational agent or that may interfere with the conduct of this protocol.

cannot be assessed by the data recorded on the CRF, but would be identified through CRA monitoring. Should such events occur they will be addressed through the TF review process.

Receiving a live vaccine is prohibited due to safety reasons but is not a treatment failure criterion.

#### 15.6.15.9. Belimumab in Year 2

This use of PI prescribed belimumab in Year 2 is a treatment failure for subjects in Arms A and B. Incorrectly taking Year 1 belimumab in Year 2 is not a treatment failure. For subjects in Arms A and B all belimumab taken in Year 2 will be adjudicated to determine if it is an incorrect late dose or a prescribed re-start medication.

Receiving belimumab is not a treatment failure for Arm C subjects.

### 15.6.16. Coronavirus Disease 2019 (COVID-19) Environment Onset Date

A COVID-19 environment onset date has been defined by GlaxoSmithKline for each Country as:

| Country | COVID-19) Environment Onset Date |
|-------------------|----------------------------------|
| Argentina | 10/FEB/2020 |
| Brazil | 10/FEB/2020 |
| Canada | 10/MAR/2020 |
| France | 25/FEB/2020 |
| Germany | 10 FEB/2020 |
| Korea, Repubic of | 10/FEB/2020 |
| Mexico | 10/FEB/2020 |
| Netherlands | 10/FEB/2020 |
| Russia Federation | 13/MAR/2020 |
| Spain | 10/FEB/2020 |
| United States | 10/FEB/2020 |

This represents the best estimate of the outbreak of COVID-19 within each Country at this time.

### 15.7. Appendix 7: Reporting Standards for Missing Data

### 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) is defined as completing all phases of the study, including the Week 104 visit.</li> <li>Withdrawn subjects will not be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | <ul> <li>Withdrawal visits will be slotted as per Appendix 3 or will be summarized as withdrawal visits.</li> </ul> |

### 15.7.2. Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should not be displayed as missing.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 15.7.2.1. Missing and Partial Dates

| Partial dates will be displayed as captured in subject listing displays. The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and |
|---|
| recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: o Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and |
| hence the event is considered On treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events. o Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used. Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Missing concomitant medication start date (CMSTDT) is imputed as treatment start date TRTSDT) unless: |
| <ul> <li>concomitant medication end date (CMENDT) is prior to treatment start date (TRTSDT), whether CMENDT is complete (DD/MM/YY) or partial (some combination of CMENDT day, month or year imputed) OR</li> <li>The month or month and year of the partial CMSTDT are different from the</li> </ul> |
| Λi |


| Element | Reporting Detail |
|---|---|
| | <ul><li>"Taken prior to study?" is checked.</li></ul> |
| | If any of the above conditions are met then CMSTDT is imputed with JAN for missing month and 01 for missing day, whatever is applicable. The recorded partial date will be displayed in listings. |

# 15.8. Appendix 8: Laboratory Parameters and Toxicity Grades

| Laboratory<br>Assessments | Parameters | | | | | |
|---|---|---|---|---|---|---|
| Hematology | Platelet Count RBC Count RDW Hemoglobin Hematocrit Activated partial thromoplastin time | | MCV MCH MPV L MCHC %Reticulocytes | | Differ<br>Neutr<br>Lymp<br>Mono<br>Eosin | WBC count with Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils |
| Clinical<br>Chemistry <sup>1</sup> | BUN | Aminotransferase (AST)/ Serum Glutamic- Oxaloacetic Transaminase (SGOT) Creatinine Sodium Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase (SGPT) Glucose – Calcium Alkaline | | n | Total and direct bilirubin | |
| | Creatinine | | | m<br>ruvic | Total Protein | |
| | Glucose –<br>Nonfasting | | | | | eGRF |
| Routine<br>Urinalysis | <ul> <li>Standard Urinalysis Macro and Urinalysis Micro (microscopic examination if blood or protein is abnormal)</li> <li>Specific gravity</li> <li>pH, Glucose, Protein, Blood, Ketones, Occult Blood, Bilirubin, Nitrite, Leukocyte Esterase by dipstick</li> <li>Spot Urine (protein:creatinine ratio)</li> </ul> | | | | | · |
| Immunoglobulins | | | | | | |
| Autoantibodies | <ul> <li>ANA titer</li> <li>Anti-dsDNA</li> <li>aCL</li> <li>Beta-2-glycoprotein</li> <li>Lupus anticoagulant</li> <li>Extractable nuclear antigens (ENAs)</li> </ul> | | | | | |

| Laboratory<br>Assessments | Parameters |
|---|---|
| Serum<br>Complement | <ul><li>Complement C3</li><li>Complement C4</li></ul> |
| Urine Drug<br>Screen | Amphetamines, Barbiturates, Benzodiazepines, Cocaine Metabolites,<br>Marijuana Metabolites, Methadone, Opiates, Phencyclidine,<br>Propoxyphene, Ethanol |
| Genetics | Blood sample collection |
| Belimumab PK | Blood sample collection |
| Rituximab PK | Blood sample collection |
| RNA Interferon<br>Signature | Blood sample collection |
| PBMC | Blood sample collection |
| Immunogenicity | Blood sample collection |
| B Cell Subset | Blood sample collection |
| B-Cell Receptor | Blood sample collection |
| BLyS Protein | Blood sample collection |
| Other Screening<br>Tests | Follicle-stimulating hormone and estradiol (as needed in women of non-childbearing potential only) |
| | <ul> <li>Serum human chorionic gonadotropin (hCG) pregnancy test (as needed<br/>for women of childbearing potential)</li> </ul> |
| | Serology (HIV antibody, hepatitis B surface antigen [HBsAg], and hepatitis C virus antibody) |
| | • |

#### NOTES:

Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are stated in the protocol. All events of ALT ≥3 × upper limit of normal (ULN) and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).

Laboratory parameters may need to have units converted for reporting. Equivalent units are:

 $1x10^9/L = 1,000,000,000 cells/L = 1,000 cells/\mu L = 1,000 cells/mm^3$  1g/L = 100 mg/dL = 100 mg/100 mL = 1 mg/mL

#### 15.8.1. **Adverse Event and Laboratory Value Severity Grade Tables**

| <u>HEMATOLOGY</u> | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| | MILD | <u>MODERATE</u> | <u>SEVERE</u> | POTENTIALLY LIFE-<br>THREATENING |
| Hemoglobin<br>Leukocytes<br>Absolute Neutrophil Count<br>Platelets | | > 8.0 – 9.5 g/dL<br>2000-2999/mm3<br>1000-1499/mm3<br>50,000 –<br>74,999/mm3 | 6.5 - 8.0 g/dL<br>1000-1999/mm3<br>500-999/mm3<br>25,000 -<br>49,999/mm3 | < 6.5 g/dL<br>< 1000/mm3<br>< 500/mm3<br>< 25,000/mm3 |
| Prothrombin Time (PT) | > 1.0-1.25 x<br>ULN* | > 1.25-1.5 x ULN | > 1.5-3.0 x ULN | > 3.0 x ULN |
| Partial Thromboplastin Time (PTT) | > 1.0-1.66 x<br>ULN | > 1.66-2.33 x<br>ULN | > 2.33-3.0 x ULN | > 3.0 x ULN |
| Methemoglobin | 5.0-10.0 % | 10.1-15.0 % | 15.1-20.0 % | > 20% |
| | | | | (continued) |

\*ULN = Upper Limit of Normal.

Modified from DMID Adult Toxicity Tables, 2001

| CARDIOVASCULAR Cardiac Arrhythmia | GRADE 1<br>MILD | GRADE 2 MODERATE Asymptomatic/transient; dysrhythmia; no treatment req | GRADE 3 <u>SEVERE</u> Recurrent/persistent dysrhythmia. Symptomatic; treatment req | GRADE 4 POTENTIALLY LIFE- THREATENING Unstable dysrhythmia hospitalization and treatment required |
|---|---|---|---|---|
| Hypotension | Transient orthostatic hypotension, no treatment | Symptoms correctable with oral fluid treatment | IV fluid req,<br>no hospitalization<br>req | Hospitalization req |
| Hypertension | Transient,<br>increase<br>> 20 mm/Hg; no<br>treatment | Recurrent; chronic<br>increase<br>> 20 mm/Hg, treatment<br>req | Acute treatment<br>req; out patient<br>hospitalization<br>possible | Hospitalization req |
| Pericarditis | Minimal effusion | Mild/moderate<br>asymptomatic effusion,<br>no treatment | Symptomatic<br>effusion,<br>pain, ECG changes | Tamponade OR pericardiocentesis OR surgery req |
| Hemorrhage, Blood<br>Loss | - | Mildly symptomatic;<br>no treatment required | Gross blood loss<br>OR<br>1-2 units transfused | Massive blood loss OR > 2 units transfused |
| | | | | (continued) |

<sup>1.</sup> Modified from (DMID) Adult Toxicity Tables, 2001

| CHEMISTRIES | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Sodium | | | | |
| Hyponatremia | 130-135 meg/L | 123-129 meg/L | 116-122 meg/L | < 116 meg/L |
| Hypernatremia | 146-150 meq/L | 151-157 meq/L | 158-165 meg/L | > 165 meg/L |
| Potassium | · | · | · | · |
| Hypokalemia | 3.0-3.4 meq/L | 2.5-2.9 meq/L | 2.0-2.4 meq/L | < 2.0 meq/L |
| Hyperkalemia | 5.6-6.0 meg/L | 6.1-6.5 meg/L | 6.6-7.0 meg/L | > 7.0 meg/L |
| Phosphate | · | · | · | • |
| Hypophosphatemia | 2.0-2.4 mg/dL | 1.5-1.9 mg/dL | 1.0-1.4 mg/dL | < 1.0 mg/dL |
| Calcium- (Corrected For Albu | | · · | · · | · · |
| Hypocalcemia | 7.8-8.4 mg/dL | 7.0-7.7 mg/dL | 6.1-6.9 mg/dL | < 6.1 mg/dL |
| Hypercalcemia | 10.6-11.5 mg/dL | 11.6-12.5 mg/dL | 12.6-13.5 mg/dL | >13.5 mg/dL |
| Magnesium | · · | · · | · · | · · |
| Hypomagnesemia | 1.2-1.4 meg/L | 0.9-1.1 meg/L | 0.6-0.8 meg/L | < 0.6 meg/L |
| Albumin | · | · | · | ' |
| Hypoalbuminemia | 3.00-3.49 g/dL | 2.50-2.99 g/dL | 2.00-2.49 g/dL | < 2.00 g/dL |
| Bilirubin (Total) | · · | · · | · · | · · |
| Hyperbilirubinemia (Total) | > 1.0-1.5 x ULN | > 1.5-2.5 x ULN | > 2.5-5 x ULN | > 5 x ULN |
| Glucose | | | | |
| Hypoglycemia | 55-64 mg/dL | 40-54 mg/dL | 30-39 mg/dL | < 30 mg/dL |
| Hyperglycemia | 116-160 mg/dL | 161-250 mg/dL | 251-500 mg/dL | > 500 mg/dL |
| (nonfasting & no prior | · · | · · | · · | · · |
| diabetes) | | | | |
| Triglycerides | 151-399 mg/dL | 400-750 mg/dL | 751-1200 mg/dL | > 1200 mg/dL |
| Creatinine | > 1.0-1.5 x ULN | > 1.5-3.0 x ULN | > 3.0-6.0 x ULN | > 6.0 x ULN |
| Uric Acid | | | | |
| Hyperuricemia | 7.5-10.0 mg/dL | 10.1-12.0 mg/dL | 12.1-15.0 mg/dL | > 15.0 mg/dL |
| Liver Transferases (AST, | 1.25-2.5 x ULN | > 2.5-5.0 x ULN | > 5.0-10.0 x ULN | > 10.0 x ULN |
| ALT, and GGT) | | | | |
| Alkaline Phosphatase | 1.25-2.5 x ULN | > 2.5-5.0 x ULN | > 5.0-10.0 x ULN | > 10.0 x ULN |
| Pancreatic Enzymes | | | | |
| Amylase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Pancreatic amylase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Lipase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Hypoglobulinemia (IgG)* | 550-700 mg/dL | 400-549 mg/dL | 250-399 mg/dL | < 250 mg/dL |
| | | | | (continued) |

Modified from (DMID) Adult Toxicity Tables, 2001

| GASTROINTESTINAL | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4<br>POTENTIALLY LIFE-<br>THREATENING |
|---|---|---|---|---|
| Nausea | Mild OR<br>transient;<br>reasonable intake<br>maintained | Mod discomfort<br>OR intake<br>decreased<br>for < 3 days | Severe discomfort<br>OR<br>minimal intake<br>for ≥ 3 days | Hospitalization required |
| Vomiting | Mild OR<br>transient;<br>2-3 episodes/day<br>OR<br>mild vomiting<br>lasting<br>< 1 week | Mod OR persistent; 4-5 episodes per day; OR vomiting lasting > 1 week | Severe vomiting of<br>all foods/fluids in 24<br>hours<br>OR orthostatic<br>hypotension<br>OR IV treatment<br>req | Hypotensive shock OR hospitalization required for IV treatment req |
| Diarrhea | Mild or transient;<br>3-4 loose stools<br>per day<br>OR mild diarrhea<br>lasting<br>< 1 week | Mod OR persistent; 5-7 loose stools per day or diarrhea lasting ≥ 1 week | Bloody diarrhea;<br>OR orthostatic<br>hypotension<br>OR > 7 loose<br>stools/day<br>OR IV treatment req | Hypotensive shock OR hospitalization req |
| Oral<br>Discomfort/Dysphagia | Mild discomfort,<br>no difficulty<br>swallowing | Difficulty swallowing but able to eat and drink | Unable to swallow solids | Unable to drink fluids;<br>IV fluids req |
| Constipation | Mild | Moderate | Severe | Distention with vomiting |

Modified from (DMID) Adult Toxicity Tables, 2001

| RESPIRATORY | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br><u>SEVERE</u> | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Cough<br>(for aerosol<br>studies) | Transient; no treatment | Treatment associated cough; inhaled bronchodilator | Uncontrolled cough; systemic treatment req | |
| Bronchospasm<br>Acute | Transient; no<br>treatment;<br>FEV1 70% to<br>< 80%<br>(or peak flow) | treatment req;<br>normalizes with<br>bronchodilator;<br>FEV1 50% to < 70%<br>(or peak flow) | No Normalization<br>with bronchodilator;<br>FEV 25% to < 50%<br>(or peak flow),<br>retractions | Cyanosis; FEV1 < 25%<br>(or peak flow) OR intubated |
| Dyspnea | Dyspnea on exertion | Dyspnea with normal activity | Dyspnea at rest | Dyspnea requiring O2 therapy |

| URINALYSIS Proteinuria | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| <i>Dispstick</i><br>Protein | 1+ | 2-3 + | 4 + | Nephrotic syndrome |
| Spot Urine: Protein:Creatinine Ratio mg/mg | 0.2-1.0 | > 1.0-2.0 | > 2.0-3.5 | > 3.5 |
| 24 Hour Urine:<br>Protein | 200 mg - 1g<br>loss/day | > 1-2 g loss/day | > 2-3.5 g loss/day | Nephrotic syndrome<br>OR > 3.5 g loss/day |
| Hematuria | Microscopic only<br>> 3 to < 10<br>RBC/hpf | Gross, No clots ≥ 10 RBC/hpf | Gross plus clots OR<br>RBC casts | Obstructive OR transfusion required |

RBC = red blood cell; hpf = high power field.
Modified from (DMID) Adult Toxicity Tables, 2001

| MISCELLANEOUS | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Fever (oral > 12 hours) | 37.7-38.5°C or<br>100.0-101.5°F | 38.6-39.5°C OR<br>101.6-102.9°F | 39.6-40.5°C OR<br>103-105°F | > 40.5°C OR > 105°F |
| Headache | Mild; No<br>treatment req | Mod; or non-<br>narcotic analgesia<br>treatment | Severe; OR responds to initial narcotic treatment | Intractable; OR requiring repeated narcotic treatment |
| Allergic Reaction | Pruritus without rash | Localized urticaria | Generalized<br>urticaria<br>angioedema | Anaphylaxis |
| Cutaneous/Rash/<br>Dermatitis | Erythema,<br>pruritus rash<br>OR dry<br>desquamation | Diffuse<br>maculopapular<br>OR dry<br>desquamation | Vesiculation OR<br>moist<br>desquamation<br>ulceration | ANY ONE: mucous<br>membrane involvement,<br>suspected<br>Stevens-Johnson (TEN),<br>erythema multiforme, necrosis<br>req surgery, exfoliative<br>dermatitis |
| Local Reaction<br>(secondary<br>to parenteral<br>treatment- not<br>vaccination or skin<br>test) | Erythema | Induration < 10 mm<br>OR inflammation<br>OR phlebitis | Induration > 10 mm<br>OR ulceration | Necrosis of skin |
| Fatigue | Normal activity<br>Reduced < 25% | Normal activity<br>Reduced 25-50% | Normal activity reduced > 50%; cannot work | Unable to care for self |

Modified from (DMID) Adult Toxicity Tables, 2001

### **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| NEUROLOGIC | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Neuro-<br>cerebellar | Slight<br>incoordination OR<br>dysdiadochokinesia | Intention tremor OR<br>dysmetria OR slurred<br>speech<br>OR nystagmus | Ataxia requiring<br>assistance to walk or<br>arm incoordination<br>interfering with ADLs | Unable to stand |
| Neuro-psych/<br>mood | | None | Severe mood changes requires medical intervention | Acute psychosis requiring Hospitalization |
| Paresthesia<br>(burning,<br>tingling, etc) | Mild discomfort;<br>no treatment<br>needed | Mod discomfort<br>non-narcotic analgesia<br>req | Severe discomfort;<br>OR narcotic<br>analgesia req with<br>symptomatic<br>improvement | Incapacitating; OR not responsive to narcotic analgesia |

| Neuro-motor | Mild weakness in<br>muscle of feet but<br>able to walk and/or<br>mild increase or<br>decrease in<br>reflexes | Mod weakness in feet<br>(unable to walk on heels<br>and/or toes), mild<br>weakness in hands, still<br>able to do most hand<br>tasks and/or loss of<br>previously present reflex<br>or development of<br>hyperreflexia<br>and/or unable to do<br>deep knee<br>bends due to weakness | Marked distal<br>weakness (unable to<br>dorsiflex toes or foot<br>drop), and mod<br>proximal weakness<br>ie, in hands<br>interfering with ADLs<br>and/or requiring<br>assistance to walk<br>and/or unable to rise<br>from chair<br>unassisted | |
|---|---|---|---|---|
| Neuro-sensory | Mild impairment<br>sensations,<br>(ie, vibratory,<br>pinprick, hot/cold in<br>great toes) in focal<br>area or<br>symmetrical<br>distribution | Mod impairment mod<br>de-sensation,<br>(ie, of vibratory, pinprick,<br>hot/cold to ankles)<br>and/or joint position or<br>mild impairment that is<br>not symmetrical. | Severe impairment<br>(dec or loss of<br>sensation to knees<br>or wrists) or loss of<br>sensation of at least<br>mod degree in<br>multiple different<br>body areas (ie,<br>upper and lower<br>extremities) | Sensory loss involves limbs and trunk |

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-<br>THREATENING |
| Lymphopenia | >0.8 (GI/L) | <=0.8 - >.5(GI/L) | <=0.5->0.2(GI/L) | <=0.2(GI/L) |
| Source: CTCAE | 4.03 | | | |

# 15.9. Appendix 9: Biomarkers

| | SI BIOMARKER DATASET | | | SDTM LB DATASET | | |
|---|---|---|---|---|---|---|
| Name | BICATCD | BICAT | BITESTCD | BIORRESU | LBTESTCD | LBSTRESU |
| | GSK_TestCode | GSK_TestName | | GSK_Unit | SDTM<br>TESTCD | SDTM UNIT |
| Anti-dsDNA | ANDSAB | Anti-dsDNA antibody | CONC | IU/ML | ADSDNAAB | IU/mL |
| C3 | C3 | Complement component 3 | CONC | G/L | C3 | g/L |
| C4 | C4 | Complement component 4 | CONC | G/L | C4 | g/L |
| CD19+ Total B cells | CD19 | CD19+ | CONC | CELLS/ML | CD19 | 10^3/L |
| B cells CD20+ | CDX111 | CD19+ CD20+ | CONC | CELLS/ML | CDX111_C | 10^3/L |
| B cells CD20+ | CDX111 | CD19+ CD20+ | PCTBCELL | % | CDX111_P | % |
| Naive B cells<br>IgD+ | CDX203 | CD19+ CD27-<br>IgD+ | CONC | CELLS/ML | CDX203 | 10^3/L |
| Naive B cells<br>IgD+ | CDX203 | CD19+ CD27-<br>IgD+ | PCTBCELL | % | CDX203 | % |
| Naive CD20+<br>CD27- | CDX731 | CD19+CD20+C<br>D27- | CONC | CELLS/ML | CDX731_C | 10^3/L |
| Naive CD20+<br>CD27- | CDX731 | CD19+CD20+C<br>D27- | PCTBCELL | % | CDX731_P | % |
| Activated<br>Total B cells<br>CD95+ | CDX742 | CD19+CD95b+ | CONC | CELLS/ML | CDX742_C | 10^3/L |
| Activated<br>Total B cells<br>CD95+ | CDX742 | CD19+CD95b+ | PCTBCELL | % | CDX742_P | % |
| Memory<br>CD20+ CD27+ | CDX732 | CD19+CD20+C<br>D27+ | CONC | CELLS/ML | CDX732_C | 10^3/L |
| Memory<br>CD20+ CD27+ | CDX732 | CD19+CD20+C<br>D27+ | PCTBCELL | % | CDX732_P | % |
| Non-switched<br>memory<br>CD27+ IgD+ | CDX84 | CD19+ CD27+<br>lgD+ | CONC | CELLS/ML | CDX84 | 10^3/L |

| | SI BIOMARKER DATASET | | | SDTM LB DATASET | | |
|---|---|---|---|---|---|---|
| Name | BICATCD | BICAT | BITESTCD | BIORRESU | LBTESTCD | LBSTRESU |
| | GSK_TestCode | GSK_TestName | | GSK_Unit | SDTM<br>TESTCD | SDTM UNIT |
| Non-switched<br>memory<br>CD27+ IgD+ | CDX84 | CD19+ CD27+<br>IgD+ | PCTBCELL | % | CDX84_PC | % |
| Switched<br>memory<br>CD27+ IgD- | CDX86 | CD19+ CD27+<br>IgD- | CONC | CELLS/ML | CDX86 | 10^3/L |
| Switched<br>memory<br>CD27+ IgD- | CDX86 | CD19+ CD27+<br>IgD- | PCTBCELL | % | CDX86_PC | % |
| Plasmablasts<br>CD27b CD38b | CDX734 | CD19+CD27b+<br>CD38b+ | CONC | CELLS/ML | CDX734_C | 10^3/L |
| Plasmablasts<br>CD27b CD38b | CDX734 | CD19+CD27b+<br>CD38b+ | PCTBCELL | % | CDX734_P | % |
| Plasmablasts<br>CD20+ CD27b<br>CD38b | CDX735 | CD19+CD20+C<br>D27b+CD38b+ | CONC | CELLS/ML | CDX735_C | 10^3/L |
| Plasmablasts<br>CD20+ CD27b<br>CD38b | CDX735 | CD19+CD20+C<br>D27b+CD38b+ | PCTBCELL | % | CDX735_P | % |
| Plasmablasts<br>CD20- CD27b<br>CD38b | CDX736 | CD19+CD20-<br>CD27b+CD38b+ | CONC | CELLS/ML | CDX736_C | 10^3/L |
| Plasmablasts<br>CD20- CD27b<br>CD38b | CDX736 | CD19+CD20-<br>CD27b+CD38b+ | PCTBCELL | % | CDX736_P | % |
| Transitional<br>CD24b CD27-<br>CD38b | CDX199 | CD19+ CD24b+<br>CD38b+ CD27- | CONC | CELLS/ML | CDX199 | 10^3/L |
| Transitional<br>CD24b CD27-<br>CD38b | CDX199 | CD19+ CD24b+<br>CD38b+ CD27- | PCTBCELL | % | CDX199_P | % |
| Transitional<br>CD10+ CD24b<br>CD27- CD38b | CDX738 | CD19+CD10+C<br>D24b+CD27-<br>CD38b+ | CONC | CELLS/ML | CDX738_C | 10^3/L |
| Transitional<br>CD10+ CD24b<br>CD27- CD38b | CDX738 | CD19+CD10+C<br>D24b+CD27-<br>CD38b+ | PCTBCELL | % | CDX738_P | % |
| CD3+ Total T cells | CD3 | CD3+ | CONC | GI/L | CD3 | 10^9/L |
| CD4+ T cells | CDX03 | CD3+ CD4+ | CONC | GI/L | CDX03 | 10^9/L |
| CD8+ T cells | CDX02 | CD3+ CD8+ | CONC | GI/L | CDX02 | 10^9/L |

## 15.10. Appendix 10: Abbreviations & Trade Marks

### 15.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| aCL | Anti-cardiolipin |
| ACR | American College of Rheumatology |
| ADA | Anti-Drug Antibody |
| ADA | Analysis Data Model |
| - | |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANA | Anti-nuclear Antibody |
| ANCOVA | Analysis of Covariance |
| anti-dsDNA | Anti-double-stranded DNA |
| BLyS | B-Lymphocyte Stimulator |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CMQ | Customized MedDRA Query |
| CNS | Central Nervous System |
| CSR | Clinical Study Report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| EU | European Union |
| FACIT-Fatigue | Functional Assessment of Chronic Illness Therapy - Fatigue Scale |
| FACS | Florescence Activated Cell Sorting |
| FDA | Food and Drug Administration |
| GSK | GlaxoSmithKline |
| HZ | Herpes Zoster |
| IBA | Independent Blinded Assessor |
| ICH | International Conference on Harmonisation |
| ICF | Informed Consent Form |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| lg | Immunoglobulin |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| IV | Intravenous |
| LLDAS | Lupus Low Disease Activity State |
| LLN | Lower Limit of Normal |
| LOQ | Limit of Quantification |
| MAR | Missing At Random |
| MCID | Minimal Clinically Important Difference |

| Abbreviation | Description |
|--------------|----------------------------------------------------------|
| MedDRA | Medical Dictionary for Regulatory Activities |
| MITT | Modified Intent-To-Treat |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| OI | Opportunistic Infections |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PGA | Physician Global Assessment |
| PI | Principal Investigator |
| PISR | Post-Injection Systemic Reactions |
| PK | Pharmacokinetic |
| PopPK | Population Pharmacokinetic |
| PP | Per Protocol |
| PROs | Patient Reported Outcomes |
| PSAP | Program Safety Analysis Plan |
| PT | Preferred Term |
| PtGA | Patient Global Assessment |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SDTM | Study Data Tabulation Model |
| SLE | Systemic Lupus Erythematosus |
| SLEDAI | Systemic Lupus Erythematosus Disease Activity Index |
| SLEDAI-2K | Systemic Lupus Erythematosus Disease Activity Index 2000 |
| SLICC | Systemic Lupus International Collaborating Clinics |
| SOC | System Organ Class |
| TB | Tuberculosis |
| ULN | Upper Limit of Normal |
| WPAI | Work Productivity and Activity Impairment Questionnaire |

### 15.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| BENLYSTA (belimumab) |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Rituxan |
| SAS |

### 15.11. Appendix 11: List of Data Displays

### 15.11.1. Data Display Numbering

RAP generated displays follow the Format A XY.ZZ, where:

A refers to the reporting effort i.e.

- T = Table
- L = Listing
- F = Figure

X refers to the reporting effort i.e.

- 1 = After all subjects have completed Week 52 i.e. Year 1 data
- 2 = After all subjects have completed Week 104 i.e. Year 2 & Year 1&2

Y refers to the Section i.e.

- 1 = Study population
- 2 = Efficacy
- 3 = Safety
- 4 = Health outcomes
- 5 = Biomarkers
- 6 = Pharmacokinetic

ZZ is an incremental count with a new number for every output.

### 15.11.2. Mock Example Shell Referencing

Example mock-up displays are provided in documents

205646 Study Pop Shells

205646 Efficacy Shells

205646 Safety Shells

205646 Health Outcomes Shells

205646 Biomarker Shells

205646 PK Shells

#### 15.11.3. Deliverables

| Delivery | Description |
|---|---|
| DB SAC | Double Blind Statistical Analysis Complete – Primary SAC for Year 1 |
| EOS SAC | End of Study Statistical Analysis Complete – EoS SAC for Year 2 and Years 1&2 Combined |

### 16. ATTACHMENTS

### 16.1. Attachment 1: AESI Preferred Term Definitions

The AESI definitions under the current version of MedDRA at the time of reporting will be found via the following IMMS pathname:

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/